

# Strong Families Start at Home/ Familias Fuertes Comienza en Casa

Full Protocol for Intervention Delivery

A Home-based Video and Motivational Interviewing Intervention to Improve Preschoolers Diet Quality and Parent

Protocol Revision History Version Number: 1

Version Date: 02/19/2020

| Full Proto | col for Intervention Delivery | 0 |
|---|---|---|
| | Study Team Roster | 2 |
| | Participating WIC Sites | 3 |
| | Study Abstract | 4 |
| | Study Objectives | 4 |
| | Overview of Study Timeline and Data Collection Timepoints | 5 |
| | Role of Support Coach | 5 |
| | Scheduling and Communication | 6 |
| | Study Intervention | 6 |
| | Home Visits | 6 |
| | First Home Visit | 8 |
| | Potential Questions/Scenarios & Responses for Home Visit 1 | 12 |
| | Second Home Visit | 12 |
| | Potential Questions/Scenarios & Responses for Home Visit 2 | 13 |
| | Third Home Visit | 13 |
| | Potential Questions/Scenarios & Responses for Home Visit 3 | 15 |
| | Phone Calls | 14 |
| | Fidelity and Quality Control Measures | 15 |
| | Communication | 15 |
| Intervention | on Materials in English | 16 |
| | Visit 1 Script | 17 |
| | Visit 2 Script | 30 |
| | Visit 3 Script | 37 |
| | Phone Call Script | 45 |
| | Intervention Text Messages | 51 |
| Material | es para la Intervención | 57 |
| en Españo | ol . | 57 |
| | Visit 1 Script | 58 |
| | Visit 2 Script | 70 |
| | Visit 3 Script | 78 |
| | Phone Call Script | 87 |
| | Text Messages | 93 |



| Control Materials English | 98 |
|------------------------------------|-----|
| Visit 1 Script | 99 |
| Visit 2 Script | 106 |
| Activities | 112 |
| Visit 3 Script | 115 |
| Phone Call Script | 120 |
| Control Text Messages | 126 |
| Materiales para control en español | 129 |
| VIsit 1 Script | 130 |
| Visit 2 Script | 136 |
| Actividades | 143 |
| Visit 3 Script | 146 |
| Phone Call Script | 152 |
| Text Messages | 159 |

### Study Team Roster

| Alison Tovar | PI | alison_tovar@uri.edu<br>4018749855 |
|--------------|----|------------------------------------|



| Patricia Risica | Co-I | patricia_risica@brown.edu |
|---|---|---|
| Kim Gans | Co-I | Kim.Gans@chip.uconn.edu |
| Karen McCurdy | Co-I | kmccurdy@uri.edu |
| Ernestine Jenning | CHW supervision, MI training, and adherence | ernestine_jennings@brown.e<br>du |
| Katelyn Fox | RA/ Project manager | katelyn fox@uri.edu<br>401-787-0821- personal<br>401-545-9105 - study |
| Andrea Ramirez | RA | andrea_ramirez@uri.edu<br>401-441-4812 |
| Amy Moore | PRN | amy_moore@uri.edu |
| Maggi | RA<br>Video coding | margaret_samson@my.uri.ed<br>u |
| Adam | UGRA | adam_brice@my.uri.edu |
| Ivonne | UGRA | ivone_sical@my.uri.edu<br>401-500-9449 |
| Haley Blanchette | JWU Intern | hblanchette01@jwu.edu |
| Rachel | UGRA | rachel_oliva@my.uri.edu |
| Patricia Castillo | CHW | 401- 654-9187 |
| Yesicca Cranshaw | CHW | 401-300-2258 |
| Heidi Samaoya | CHW | 401-248-5008 |

### Participating WIC Sites

| Meeting Street/St Josephs | Megan Sheehy | msheehy@meetingstreet.org, |
|---------------------------|--------------|----------------------------|
|---------------------------|--------------|----------------------------|



| Sankofa/West Elmwood | Isabella Fiore | isabellefiore8@gmail.com<br>ifiore@westelmwood.org |
|---|---|---|

#### Study Abstract

There is an urgent need to create effective interventions to help parents establish a healthy diet among their children early in life, especially among low-income and ethnically diverse families. U.S. children eat too little fruits and vegetables and whole grains, and too many energy dense foods, dietary behaviors associated with increased morbidity from cardiovascular diseases. Contributing to this poor diet is consuming foods outside the home, having unhealthy foods available in the home and lack of home-prepared meals. Parents play a key role in shaping their child's diet and best practices suggest that parents should involve children in food preparation, offer, model and encourage a variety of healthy foods. In addition, while parents help to shape food preferences, not all children respond in the same way and certain appetitive traits, such as satiety responsiveness (sensitivity to internal satiety signals), food responsiveness (sensitivity to external food cues), and enjoyment of food may help explain some of these differences. Prior interventions among preschool aged children to improve their diet have not used a holistic approach that fully targets the home food environment, by focusing on food quality, food preparation, and positive feeding practices while acknowledging a child's appetitive traits. This proposal will build upon pre-pilot work to develop and pilot-test the feasibility, acceptability and preliminary efficacy of a novel home-based intervention with low-income ethnically diverse families of preschool children to inform a future fully powered randomized controlled trial. The proposed 6-month intervention will include 3 monthly home visits by a community health worker (CHW) trained in motivational interviewing, that include in-home cooking demos. In between visits, parents will receive tailored text-messages 2x/wk. and monthly mailed tailored materials. During the last 3 months CHW phone calls will replace the home visits. The intervention will be tailored for individual families based on the child's appetitive traits. The aims are as follows: Aim 1. To conduct focus groups with 40 ethnically diverse parents of preschoolers to inform the development of and adaptation of the intervention components; Aim 2. To conduct a pilot RCT with 60 parent-child pairs (30 intervention/30 control) to determine the feasibility and acceptability of the enhanced intervention and determine the preliminary efficacy on child diet quality, feeding practices and availability of healthy foods in the home. The proposed research will lay the groundwork for a larger RCT to educate, support, motivate, and empower lowincome parents to prepare healthy meals and use healthy feeding practices, which will improve children's diets and ultimately their health.

#### Study Objectives

Aim 1: To conduct a pilot randomized controlled trial with 60 parent-child pairs (30 intervention/30 control) from ethnically diverse, low-income families with preschoolers to:



#### Aim 1.1: Determine the feasibility and acceptability of the enhanced intervention.

Aim 1.2 Determine the preliminary efficacy of the enhanced intervention on changes in children's diet quality (primary outcome) and parental feeding practices and availability of healthy foods in the home (secondary outcomes) and calculate effect sizes for a future randomized controlled trial (RCT).

We hypothesize that the intervention will be feasible and acceptable to parents and that parentchild pairs randomized to the intervention condition will demonstrate greater improvements in the outcomes after six months compared to the comparison condition (attention control of a school readiness intervention).

Exploratory aim: Explore how parents' skills, perceived competence and intrinsic motivation are related to changes in children's diet quality and parental feeding practices.

#### Overview of Study Timeline and Data Collection Timepoints



#### Role of Support Coach

Support coaches will be involved with home visit 1, home visit 2, home visit 3, phone visit 4, phone visit 5, and phone visit 6.

The role of the support coach is to



- 1. Schedule visits and phone calls.
- 2. Deliver scripted MI sessions using provided materials.
- 3. Review meal recording clip and recommendations sent by research staff.
- 4. Collaborate with culinary intern during in home cooking demonstration.
- 5. Record "process data". All visits will have data collection forms (to be completed after each session by the support coach) & a satisfaction questionnaire (to be completed by the participant at the end of the home sessions) that will be entered via RedCap Software. Each support coach will have their own username and password to enter data into RedCap. Each coach will have access to two projects titled "Home Visiting R34 Intervention" and "Spanish Home Visiting R34 Intervention".
- 6. Communicate regularly with research staff. See study roster for contact information.
  - a. Primary contacts Katelyn Fox (redcap/ nutrition/ feeding) & Ernestine Jennings (MI/Coaching)

#### Scheduling and Communication

The first home visit with the participants will be scheduled by study staff during the baseline data collection visit based on the support coach's availability in the google calendar. Coaches should ensure that their availability is entered into the google calendar by the 15th of the month for the following month. Project manager will alert coaches when new participants have been scheduled and to which group they have been assigned via email and text.

After the first visit, coaches will be responsible for scheduling subsequent visits based on their availability (and for feeding your child group visit 2 the JWU intern's availability). Dates for visits will be entered in google calendar by study ID number and also must be entered into Redcap form titled "Home Visit and Phone Call Schedule". It is important that the visit date also be entered into redcap because this is the form that will automatically prompt the reminder call/texts.

Each participant will receive a reminder of their visit 3 days & 1 day prior. If a participant indicates that they need to reschedule the visit, the project manager will alert the coach and the coach will reach out to the family to reschedule the visit based on their availability. If a coach needs to reschedule a visit they should also update the visit date in Redcap so that reminder text messages reflect the correct date.

#### Study Intervention

#### Home Visits

Prior to each home visit, the support coach will login to Redcap; Redcap Application and download the participants record and obtain contact information & address by following the commands below. Note you will need access to wifi for this function.



My Projects> choose project based on language of participant >Refresh Set Up & Data> Get a Partial Set of Data> Participant ID> download checked records/events> Collect Data>Recruitment> Eligibility









#### First Home Visit

Prior to the visit access Strong Families Start at Home Google Drive for content you will be using for home visit 1. It is important that you access google drive while connected to wifi and select "make available offline" in the document settings so that you are able to access it if the internet connection is poor in the home.

Select Support Coach Name Drive folder and choose study id number, where you will find the following items:

1. Video clip

A video clip will be in the folder. Play first clip, this will be the positive practice. Pause the clip when "clip 2" appears on the screen. Provide feedback then press play to review the negative clip and provide feedback"

If a participant does not submit a video prior to the visit you will be provided "test clips"

\*If I-Pad freezes and you are not able to review the video with the participant would explain to family, thank them for sending in the video, and ask if it's ok that you would like to offer feedback on what they sent. Then review feedback from.

2. Feedback form: The URI team will summarize the context of the meal or the reading activity, depending on the intervention or control group and will provide some language both for the positive practice and the practice that can be improved upon.

If participant does not submit a video prior to the visit you will be provided "sample feedback form"



3.

Eating behavior tailored information. During the baseline data collection session, parents completed a survey answering questions about their child's eating behaviors. Depending on their responses and their child's eating behaviors, we will be providing them with some tailored information (if applicable)

If participant has been identified to have one of the traits based on their responses, read the corresponding section of script and provide additional corresponding handout. If no trait is identified skip that section of the script. The following icons will be used to identify each trait



**Food Fussiness** 



Low Satiety Responsiveness



High Food Responsiveness

You will also need the following materials

- 1. Study Timeline
- 2. Handouts 1 and 2 "Raising a Healthy Eater Doesn't Need to be Stressful" and Healthy Eating Starts at Home
- 3. Goal sheet
- 4. Recipes to select from for the second home visit "Lentil Soup or Black Bean Salad"
- 5. Coloring sheets for child

Please record all sessions using the provided recording device. You will be uploading therecordings to your Google Drive folders after the home visits.



At the end of the home visit open I-Pad & Redcap Application select Collect Data> Participant Record>Home Visit 1 and complete all forms





- 1. Home Visit and Phone Call Schedule
  - a. Use both google calendar and redcap for scheduling the next visit.
  - b. Remember that the culinary intern will be attending this visit if the participant is in the intervention group, so schedule based on your availability and hers. If there is no overlapping availability in the google calendar schedule based on your availability and contact the culinary intern directly to find a time where both are available.
- 2. Home Visit and Phone Call Checklist



- a. Here you can enter photo of goal sheet.
- b. If you prefer to take handwritten notes & enter into redcap after the visit that is OK
- c. After home visit, upload audio file to your google drive folder.
- 3. Home Food Prep Form.
  - a. Please add information on which recipe the participant selected
  - b. Ask them if they prefer to purchase or for us to purchase ingredients
  - c. Any notes for home cooking session
- 4. Satisfaction questionnaire Visit 1 & 3
  - a. Hand IPAD to participant to complete.

When all data forms have been completed and you are connected to wifi send the record to the online project by clicking "send data to server".



Once data are backed reset the app by clicking "refresh set up & data". This will ensure you have the most updated version of the app and will remove data from the I-Pad to ensure there is enough space to save the next participant.





#### Second Home Visit

You will need the following materials

- 1. Handouts 3 "Tips for organizing grocery shopping" and 4"Involve Children at the Grocery Store and Improve Eating at Home"
- 2. Goal sheet
- 3. Recipe book

Culinary Intern will purchase and provide food for visit and connect with coach prior to visit to coordinate.

Deliver intervention per script. Community health worker will deliver all intervention materials and culinary student will guide the food prep activity and provide all materials.

At the end of the home visit open I-Pad & Redcap Application. Collect Data>
Participant Record>
Home Visit 2

Complete the following forms

- 1. Home Visit and Phone Call Schedule
  - a. Enter date in google calendar & redcap



- 2. Home Visit and Phone Call Checklist
  - a. Here you can enter photo of goal sheet.
  - b. If you prefer to take handwritten notes & enter into redcap after the visit that is OK
  - c. Upload audio file to your google drive folder.
- 3. Satisfaction questionnaire Food Prep Visit
  - a. Hand to participant to complete.
    - i. \*note there is an additional satisfaction form for this visit for the activity. Please choose the form that corresponds with the activity "food prep" or "reading".

When all data forms have been completed and you are connected to wifi send the record to the online project by clicking "send data to server". Once data are backed up reset the app by clicking "refresh set up & data". This will ensure you have the most updated version of the app and will remove data from the I-Pad to ensure there is enough space to save the next participant.

#### Third Home Visit

This visit is very similar to visit 1, where you review feedback from the video with the parent.

Access Strong Families Start at Home Google Drive for content you will be using for visit 3. Access google drive while connected to WIFI and select "make available offline" in the document settings so that you are able to access it if the internet connection is poor in the home.

Select Support Coach Name Drive folder and choose study id number, where you will find the following items:

- 1. Video clip
  - a. Video clip will state clip 1 & clip 2one showing a positive practice and one showing a practice they can improve upon
- 2. Feedback form: The URI team will summarize the context of the meal or the reading activity, depending on the intervention or control group and will provide some language both for the positive practice and the practice that can be improved upon.



- 3. Only for Intervention group: Feeding trait tailored information. During the baseline data collection session, parents completed a survey answering questions about their child's eating behaviors. Depending on their responses and their child's eating behaviors, we will be providing them with some tailored information (if applicable)
  - a. If participant has been identified to have one of the traits based on their responses, read the corresponding section of script and provide additional corresponding handout

You will also need the following materials

- 1. Handouts 5 "Structure for Strong Families" and 6 "Family Mealtime Rules"
- 2. Goal sheets

Deliver intervention per script.

At the end of the home visit open I-Pad & Redcap Application Collect Data>
Participant Record>
Home Visit 3
Complete the following forms

- 1. Home Visit and Phone Call Schedule
  - b. Use both google calendar and redcap for scheduling the next visit.
  - c. This next visit will be a phone call
- 5. Home Visit and Phone Call Checklist
  - a. Here you can enter photo of goal sheet.
  - b. If you prefer to take handwritten notes & enter into redcap after the visit that is OK
  - c. Upload audio to google drive folder.
- 6. Satisfaction questionnaire Visit 1 & 3
  - a. Hand to participant to complete on the IPAD.

When all data forms have been completed and you are connected to WIFI send the record to the online project by clicking "send data to server". Once data are backed, reset the app by clicking "refresh set up & data". This will ensure you have the most updated version of the app and will remove data from the I-Pad to ensure there is enough space to save the next participant.

Phone Calls

Deliver intervention per script.

At the end of the home visit open I-Pad & Redcap Application



Collect Data>
Participant Record>
Phone Call Visit 4-6
Complete the following forms

- 1. Home Visit and Phone Call Schedule
  - a. Use both google calendar and redcap for scheduling the next visit.
  - b. This next visit will be a phone call to visit 5 & 6.
  - c. After visit 6 will need to schedule follow up data collection visit. Please contact Katelyn Fox for data collection team availability prior to this visit.
- 2. Home Visit and Phone Call Checklist
  - a. Here you can enter photo of goal sheet if you choose to write it or enter in the goal section.

Following the visit goal sheets will be mailed to participants.

#### Fidelity and Quality Control Measures

Study staff will review 10% of all home visits to assess fidelity and MI adherence using the MITI coding tool. If discrepancies more reviews may be conducted. In addition, the support coaches will meet to discuss visits with Ernestine.

#### Communication

Weekly meetings will be held between support coaches, Ernestine and Katelyn Fox during the first month of the project to discuss any issues that come up.

Bi-weekly meetings with study team.



### Intervention Materials in English

\*Note: For all study scripts, Bolding is used to signify what the support coach should be saying, and non-bolding is meant to provide instructions.



#### Recorder Script

(Prior to turning on recorder)

Thank you for meeting with me today. I wanted to remind you that I will be recording the session. The recording will be used to make sure each session is delivered the same way to each family. As stated in the consent form, all of the recordings will be kept in a secure place and destroyed once we complete the study. The information from the recordings will only be shared with study staff. If you are ready I will turn on the recorder now.

#### Introduction

Hi Mr./Ms. \_\_\_\_\_ my name is \_\_\_\_ and I am your support coach from the Strong Families Start at Home study at The University of Rhode Island. Today we will meet for about 1 hour. We will look at clips from your meal video that you sent us and discuss any thoughts or concerns you have about feeding your child. We will also talk about some information on healthy eating and strategies to help children eat better.

Refer to Study Timeline:

After this first meeting today, we will meet once a month for the next two months to discuss preparing meals, grocery shopping and strategies to help you feed your child. You will also receive text messages with information for you and your child. Later you will be mailed additional materials and I will call you once a month to check in on goals, problem solve and cheer you on. Once the study ends you will have one final visit with the research staff to do the same measurements you did before today's visit.

What questions do you have about the study?

•5 Minutes



Study timeline handout



#### Typical Day

First, I would like to get to know a little about your family meals.

How would you describe a typical meal with (child's name)?

If participant is unsure how to answer,

Tell me about yesterday's dinner? or

Share with me anything you think is important about meals with (child's name)

Ask the participant to tell their story. Interrupt as little as possible. Use open ended questions to keep them talking (e.g. "What happens next?", "Tell me more.")

When thinking about a typical meal with (child's name), what parts of the meal work well?

Interrupt as little as possible. Use open ended questions to keep them talking (e.g. "What happens next?", "Tell me more.")

When thinking about a typical meal with (child's name) what parts of the meal do not work so well?

Interrupt as little as possible. Use open ended questions to keep them talking (e.g. "What happens next?", "Tell me more.")

Thank you for sharing your experiences. I feel like I have a much better understanding of your approach to meals. It sounds like... Summarize the meal overview highlighting perceived strengths and barriers

#### 5 minutes



Key points: Do not try to solve problems -- our goal is to:
Gather information
Let families know you are listening
Hear their challenges and concerns
Convey a non-judgmental tone.



#### Review Video:

Now let's take a minute to watch two clips that were chosen from your family meal video. We will stop between each clip and discuss what you think. Remember, only you know what's best for your family. I'm here to talk about your thoughts and experiences when feeding your child.

Play clip 1 (Positive Practices). Pause when the screen says clip 2, explore and provide feedback.

#### What sticks out from the video?

Elicit thoughts about the videos process (filming a family meal and sending it in to the researchers).

Prompts to explore \* if parent has already offered the information you do not need to ask the question.

What surprises you, if anything? Why?

What, if anything, did you do to get your child to eat?

What, if anything worked?

What, if anything, might you want to do differently in the future?

If it's okay with you, I would like to share some thoughts on the meal.

Wait for affirmation then share feedback on positive meal practices.

What are your thoughts about these ideas?

Now let's take a look at the second clip.

What sticks out from the video?

Elicit thoughts about the videos process (filming a family meal and sending it in to the researchers).

#### 15 minutes



Feedback Sheet



Mealtime Video Clips on I-PAD



Key Points:

Identify and elicit change talk.

<u>DESIRE</u>: Want, wish, like ABILITY: Can, could, able

REASON: Specific reason for change

NEED: Need to, have to, must, important, etc.

(without stating specific reason)

COMMITMENT: Will, intend to, going to, etc.

ACTIVATION: Ready to, willing to (without

specific commitment)

TAKING STEPS: Reporting recent specific action (step) toward change

Responding to Change Talk:

Explore. Ask for elaboration: how, in what ways, why? Ask for examples: when was the last time this happened (e.g., for an adverse consequence).

<u>Affirm</u>. Express agreement, appreciation, encouragement, etc. for the desire/need/etc. to change.

Reflect. This is the most common response to change talk – to offer a simple or complex reflection (. "I hear you saying that xxx" or "You feel it is difficult to xx")

Summary. Think about the conversation like a field of flowers – pick the sentences you would like to highlight, those that focus on change, and present them back to the family in a Change talk is also collected in "bouquet" summaries. You can select what to focus on in this process.



Prompts to explore \* if parent has already offered the information you do not need to ask the question.

What surprises you, if anything? Why?

What, if anything, did you do to get your child to eat?

What, if anything worked?

What, if anything, might you want to do differently in the future?

If it's okay with you, I would like to share some thoughts on the meal.

Wait for affirmation then share feedback on negative meal practices.

What are your thoughts about these ideas?

Summarize Feedback session

It appears there are several things that you are doing well and ...

We also discussed some areas with room for improvement and you feel this information is ...

Thank you for sending this video in. This was a great discussion. I also have some printed materials that you might be interested in.



#### Review Printed Materials

During this portion of the visit, you will provide information and share some materials.

We hear from other parents that mealtimes can sometimes be stressful. Some research suggests that understanding what the roles of parents and children are during meals can make mealtimes less stressful.

#### Can I share a little bit more about this?

Provide "Raising a Healthy Eater doesn't Need to be Stressful Handout."

This first page says that the role of parents is to decide on what, where, and when children eat. You are in charge of the food that comes into your home and what your child can have at meals and snacks.

If you worry that your child won't eat what you pick there are some things you can do to help them.

You can offer them healthy choices, serve new foods with foods your child already likes, and role modeling healthy eating-kids always want to copy their parents.

It also says that your child is responsible for deciding how much they eat and learning how to behave at meals. It can be hard to let your child decide how much they will eat, because many parents worry if their child will eat enough. Remember that if you provide them 3 meals and 2-3 snacks a day they will get enough food to grow and stay healthy.

The handout also offers some tips on how to make mealtimes more enjoyable. For example; eating with your child as often as you can, having specific meal and snack times, having a set location for meals like the table or the kitchen, limiting distractions like the TV, tablet or computer, and giving small portions on your child's plate and let them ask for more if they are still hungry. You can see an example

#### 15 minutes

Raising a Healthy Eater doesn't Need to be Stressful



Identify and elicit change talk. It may be helpful to check off changes the family is interested in making on the handout for the goal setting activity.



| on the back about how offering guided choices can help |
|---|
| kids make healthy decisions. |
| Show parents the cartoon on the back of the handout. |
| Explore thoughts on handout. |
| What are your thoughts on this? |
| What concerns do you have about the recommendations? |
| What strategies, if any, on here has your family tried? |
| What suggestions on here are you interested in trying or have thought about? |



Provide "Healthy Eating Starts at Home My Plate" handout.

We also know that many parents want to know what foods are healthy for your child. This second handout talks a little more about healthy eating and how to keep your family healthy. It is based off of "My Plate" which tells us that what we eat should be mostly whole grains, fruits, vegetables, lean protein, and low-fat or fat free dairy. It also has tips on how to get more of these healthy foods in your family's diet.

On the other side of the handout it talks about how to limit foods that aren't as healthy for us such as foods with added sugars and fats like desserts, chips, soda, juice drinks, and fried foods. It encourages you to make it easier for your children to limit these foods by keeping them out of the home. By not having them around you can avoid arguments from kids always asking for sweets or chips. There are also some tips on how you can model healthy eating, which is one way to help children eat healthy!

Show Healthy Eating Starts at Home (with watermelon).

Explore thoughts on this handout

What do you think about this?

What are your thoughts on this?

What concerns do you have about the recommendations?

What strategies, if any, on here has your family tried?

What suggestions on here are you interested in trying or have thought about?



"Healthy Eating Starts at Home"



Time Management Tip
Reflections and exploration of parents'
thoughts on the content are written into the
script -- if time is limited would be OK just to
provide the handout with brief explanation.



#### Child Specific Handout

If the child has been assigned an appetitive trait in their Google Drive folder read the corresponding script and provide additional handout. This will not be for all children.

Would it be ok to share some additional information specific to your child?



Handout for each trait



Food Fussiness

At our first visit, we asked you to answer some questions on your child's eating. Based on those answers, we can see that your child may be fussy eater.

Food fussiness or "picky eating" is a normal stage for many children. It's usually worst at age 2 and decreases by age 5. But, your survey tells us that your child may be fussier than other children. This means that they may only like certain foods or are afraid of trying new foods. Your child might refuse foods or even stop eating foods they used to love!

Parents worry about their fussy eater getting enough nutrition. Sometimes parents try to get their child to eat- by forcing them to eat what is on the plate. But, that usually makes fussy eating worse in the long run.

Provide and review "Helpful Tips for Picky Eaters" handout



Helpful Tips for Picky Eaters



Satiety Responsiveness

At our first visit, we asked you to answer some questions on your child's eating. Based on those answers, we can see that your child may have a hard time knowing when they are full. Parents of children who have trouble knowing when they are full can be tempting to restrict their eating to help them, but this can backfire.

Provide and review "Tips for helping your child with mindful eating" handout







#### Food Responsiveness

At our first visit, we asked you to answer some questions on your child's eating. Based on those answers, we can see that your child may react more strongly than other children to foods that they see or smell. Many parents of children who react this way around food worry that these children will eat too much of foods that taste good but aren't healthy (such as candy or chips). Parents may try to restrict these foods, but this can backfire. As children feel more restricted, they feel like they want those foods even more!

Provide and review "How to Make your Environment Work for You and Your Family"





#### Problem Solving/ Goal Setting

We would like to help you work on something that could help you and your child eat healthier. To do this, we would like to like to talk to you about setting a goal to address the topic you mentioned wanting to change when we went over the handouts

> (If parent identified many changes they were interested in 1. Specific: Make sure goals are detailed. making have them rank which are most important to them, choose 1-2)

Can choose from strategies on handout or participants own goal that aligns with performance objectives.

They should focus on one 1 goal, but if they choose to work on two, please write down both and ask the same questions for each.

Why do you want to make this change? (Desire) (Reflection)

How might you be able to do it? (Ability) (Reflection)

What is one good reason for making the change? (Reasons) (Reflection)

**How important is it, and why?** (0-10) (Need) (Record number) (Reflection)

> Record specific goal from the bottom of the goal setting sheet on the data sheet. The goal of this section is to develop a specific goal and identify barriers. Leave the goal setting sheet with the parent and take a photo to upload later.

#### 15 minutes



**Goal Sheet** 



Keys for Goal Setting: Goals should

- (Who, What, When, Where)
- 2. Measurable: Make sure the participant can identify what will happen when they achieve their goal.
- 3. Achievable: Goals should be realistic, not ideal
- 4. Relevant: Goals should relate to best practices for feeding and nutrition
- 5. Time Bound: Goal should have a timeline of when it will be met within the next time you meet

\*If parent chooses a behavior (ie modeling healthy behaviors) and a food goal (ie decreasing soda) Ideally combine to one goal "Model healthy eating by not having soda at dinner time this week"

Performance Objectives: As part of the study we want participants to achieve the followina

- Increase fruits and vegetables, whole grains, lean proteins served
- Increase accessibility of fruits and vegetables
- Decrease accessibility of treat foods
- Offer choices of healthy options
- Increase family meals/ role modeling
- Have a set location where the family eats, like a table or counter.
- Limit distractions like the TV, tablet, or computer



| Serve small portions and practice letting the child decide when he/she's full. Record Goal and Importance in Redcap Upload picture of goal sheet (if more than one goal record both) |
|---|



#### Assess Readiness to Make Change

Now that you have set a goal about \_[insert topic]\_\_\_\_ for your family, I would like to know how are you feeling right now about \_[insert name of goal]

On a scale of 1 to 10 where 1 means you do not want to do this at all and 10 means you really want to do this. How would you rate yourself? (Readiness)

What made you pick that number and not a lower number (like 1 or 2)? (Motivation)

On a scale of 1-10, rate your confidence or ability to [insert name of goal] \_\_\_\_\_\_, where 1 means you are not at all confident and 10 means you are very confident you can make that change. How would you rate yourself?

What made you pick that number and not a lower number (like 1 or 2)? (Facilitators )

What would it take to get to a higher number (like 8 or 9)? If a 10 What would it take to keep you at a 10?

#### Sample Summary

You feel that you are very motivated to make this change because you (first part of rating). You could (insert comments from parent).

In terms of being able to make this change, you feel that you are able to make this change because (first part of 1 or 2) You believe you could increase your confidence if (insert comments from last part 9 or 10).

It seems you are ready to make this change and are committed to making this change.

\*Note, if they have two goals, go through both motivation and confidence for each.

#### 15 minutes

- Record **Readiness** # in Redcap
- Record **Motivation** # in Redcap
- Record Confidence # in Redcap
- Record **Barriers** in Redcap
- Record **Facilitators** in Redcap



#### Plan for Meal Prep Session

At the next visit we are going to talk about planning and preparing meals and ways to involve your child. We will also prepare a quick nutritious dish for your family with your child and a culinary student from Johnson and Wales University. Here are some quick and healthy recipes that we can choose from.

Here are some recipes that we would be able to bring for you.

Show recipe for "black bean salad" and "lentil soup"

What recipe would you like to try with your family?

#### 5 minutes



Recipe list

Record Home Food Prep in Redcap

#### Wrap up

Let's schedule our next visit. What days of the week or times of day work best for you, keeping in mind that we will be preparing a meal and the visit will take 60-90 minutes.

Also, we will have our culinary intern from Johnson and Wales who will be coming to help prepare a meal. She will bring the food from the recipe you selected. She will come with me at the beginning of our next session and will set up in the kitchen area. After we talk and set a goal you, [child's name] and I will all join her to prepare the dish you chose together.

Just a reminder that you will receive text messages with helpful tips and recipes 2 x/week. Can I confirm the best number to reach you at? If you are interested in more information or want to connect with other parents of children ages 2-5 you can also check out our Facebook group.

To end, we would just like to ask you a couple of questions about today's visit, would that be ok? I will be giving you the IPAD so I don't see your answers.

Complete Visit Satisfaction Questionnaire

Thank you for taking the time to meet with me, I will see you in the next visit.

#### 5 minutes

- Record **Next Visit** in Redcap & Google Calendar
- Have participants complete satisfaction questionnaire



#### Recorder Script

(Prior to turning on recorder)

Hello, it's nice to see you again. This is Haley, who is going to be joining us today, she is a culinary nutrition intern from Johnson and Wales who is helping with our food preparation. Just as a reminder we are going to be doing a food preparation session today, would it be ok if we just put our things in the kitchen?

I wanted to remind you that I will be recording the session. The recording will be used to make sure each session is delivered the same way to each family. As stated in the consent form, all of the recordings will be kept in a secure place and destroyed once we complete the study. The information from the recordings will only be shared with study staff. If you are ready I will turn on the recorder now.

#### Introduction

During our meeting today, we will

- 1. Check in about your goals from last visit.
- 2. Talk about preparing and shopping for meals and how to involve your child.
- 3. Set goals for the next visit.
- 4. Prepare a meal together.

What questions do you have?

If you have questions as we go, feel free to stop and ask me.

#### Assess

Tell me what you remember from our last talk about healthy ways to feed your child.

Affirm Reflect 2-5 minutes

2 Minutes



Helpful to bring copies of visit 1 handout to provide if requested.



Thank you for sharing your experiences. It is helpful to know. It sounds like... Summarize Reassess 10 minutes Last time we talked you identified \_\_\_\_\_ as a goal you wanted to work on. Visit 1 Goal Sheet available in Last time you said this was X/10 important to you. How Redcap under Home Visit 1 encounter. consistent is that with how you currently feel? **Key Points:** Last time you said you were x/10 confident, how consistent is Identify and elicit change talk. that with how you currently feel? DESIRE: Want, wish, like ABILITY: Can, could, able What were some of the changes you came up with at/after our REASON: Specific reason for change last visit? NEED: Need to, have to, must, important, etc. (without stating specific reason) How did that work for you and your child? COMMITMENT: Will, intend to, going to, etc. How satisfied are you with what you tried? ACTIVATION: Ready to, willing to (without specific commitment) What helped you try this new (insert strategy/goal name)? TAKING STEPS: Reporting recent specific action (step) toward change Responding to Change Talk: What got in the way or made it hard? Explore. Ask for elaboration: how, in what ways, why? Ask for examples: Relate to values /goals for family meals when was the last time this happened (e.g., for an adverse consequence). If there were two goals, review both then summarize. Affirm. Express agreement, appreciation, encouragement, etc. for the desire/need/etc. to change. Summarize & Reflect Reflect. This is the most common response to change talk - to offer a It appears there are several things that went well Summarize simple or complex reflection (. "I hear you saying that xxx" or "You feel it is difficult You also discussed some things you want to change Summarize to xx")



like a field of flowers - pick the

Summary. Think about the conversation

sentences you would like to highlight, those that focus on change, and present them back to the family in a Change talk

is also collected in "bouquet" summaries. You can select what to focus on in this process.

#### Grocery Shopping & Preparing meals

Now let's change topics a bit and talk about this visit's topic, shopping for and preparing meals

Tell me a little bit about how you shop for your food?

What challenges do you have shopping for meals?

What works well when you shop for meals?

If it is okay with you, Haley and I would like to share some more information about shopping for meals. We will also talk about ways to include your child.

#### Review visit 2 handouts

Grocery shopping and planning meals can be hard, especially with young kids. This week's handout contains tips for making grocery shopping easier and saving you time and money!

Review Tips for Organizing Grocery Shopping.

As you can see the biggest recommendation is planning ahead so that you know what you need for the week. Here is an example of what 6 days of meals and snacks would look like for a family of 4. Notice how much cheaper the meals are than going to fast food or convenience store.

Review Involve your children at the grocery store

Also, it suggests some tips for involving your kids at the market and at home. We know that it can be challenging to bring young children to the store but here are some ideas to keep them busy and interested in learning about food. Playing games such as I Spy can help keep them busy. If they are asking for food letting

#### 15 minutes

• Tips for organizing grocery shopping

Involve children at the grocery store and improve Eating at Home

Identify and elicit change talk. It may be helpful to check off changes the family is interested in making on the handout for the goal setting activity.



# them help pick out fruits and vegetables. Kids are more likely to eat foods if they are involved in picking them out

Review handout with parent, then ask the following:

#### Which of these strategies have you tried before?

Affirm, reflect

#### What would you be interested in trying?

Affirm, reflect

# What concerns do you have about the recommendations? i.e. possible challenges?

Affirm, reflect

Problem Solving/ Goal Setting.

### Now I would like to talk to you about setting a goal to address the topic you mentioned wanting to change

If parent identified many changes they were interested in making have them rank which are most important to them, choose 1-3.

Can choose from strategies on handout or participants own goal that aligns with best practices.

### Why do you want to make this change? (Desire) (Reflection)

How might you be able to do it? (Ability) (Reflection)

What is one good reason for making the change? (Reasons) (Reflection)

**How important is it, and why?** (0-10) (Need) (Record number) (Reflection)

The goal of this section is to develop a specific goal and identify barriers.

Leave the goal setting sheet with the parent and take a photo this week" to upload later.

#### 15 minutes



**Goal Sheet** 



Keys for Goal Setting: Goals should be:

- Specific: Make sure goals are detailed. (Who, What, When, Where)
- Measurable: Make sure the participant can identify what will happen when they achieve their goal.
- **3.** <u>Achievable</u> Goals should be realistic, not ideal
- **4.** Relevant Goals should relate to best practices for feeding and nutrition 5. Time Bound Goal should have a
- timeline of when it will be met within the next time you meet

\*If parent chooses a behavior (ie modeling healthy behaviors) and a food goal (ie decreasing soda) Ideally combine to one goal "Model healthy eating by not having soda at dinner time this week"



| | Performance Objectives: As part of the study we want participants to achieve the following Increase family meals Increase modeling of healthy foods Increase preparing meals Increase inclusion of vegetables Talk to children about benefits of foods Involve child in food preparation |
|---|---|
| Assess Readiness to Make Change Motivation Now that you have set a goal aboutlinsert topic!for your | Record Readiness in Redcap |
| Now that you have set a goal about _ [insert topic] for your family, I would like to know how you are feeling right now about _ [inset name of goal] | Record Motivation # in Redcap Record Confidence # in Redcap |
| On a scale of 1 to 10 where 1 means you do not want to do this at all and 10 means you really want to do this. How would you rate yourself? (Readiness) | Record <b>Barriers</b> in Redcap Record <b>Facilitators</b> in Redcap |
| What made you pick that number and not a lower number (like 1 or 2)? (Motivation) | Record Facilitators in Redcap |
| Confidence On a scale of 1-10, rate your confidence or ability to [inset name of goal], where 1 means you are not at all confident and 10 means you are very confident you can maintain that change. | |
| How would you rate yourself? | |
| What made you pick that number and not a lower number (like 1 or 2)? (Barriers) | |
| What would it take to get to a higher number (like 8 or 9)? If a 10, what would it take to keep you at a 10? (Facilitators) | |
| Sample Summary: | |


You feel that you are very motivated to make this change because you (first part of rating). You could (insert comments from parent). In terms of being able to make this change, you feel that you are able to make this change because (first part of 1 or 2) You believe you could increase your confidence if (insert comments from last part 9 or 10). It seems you are ready to make this change and are committed to making this change.

Leave the goal setting sheet with the parent.

When we meet next time, we will review this goal so please keep this sheet with your materials.

# Meal Prep Session

Now let's do something different and make a meal together. So, our goal is to involve your child in this session. It can be helpful to get all the materials out ahead of time. *Now let's see if* I can help you get [child's name] involved

Invite child over to help/ Prepare meal.

Haley: So today, we are going to be preparing X recipe today. We want to involve (child's name) today and thought he could help today with (enter name of task). Would that be ok with you?

Begin preparing the recipe together. Take note: you can assess if the parent would like more instruction in preparing the meal or if they already know how to cut allow them to help and you can help with the child involvement.

Walk through the steps as you prepare the meal and share any tips that may be helpful to the parent.

Some important tips to share:

# 30 minutes

Record prepared meal

Recipe Book (recipe & child activity sheet)

Keys for Support Coach
Assist parent in involving child.
Translate for Haley during Spanish
language visit

Identify/Elicit change talk during cooking session.



| 1) | Washing hands- both parent and child-very important | |
|---|---|---|
| 0) | before cooking anything | |
| 2) | Setting up all ingredients and prepping BEFORE | |
| 2) | putting recipe together can save time | |
| 3) | Putting ingredients away and cleaning up as you can | |
| 4) | go can make clean up easier | |
| , | How to cut the onion | |
| | Rolling the lemon/lime before squeezing | |
| 0) | How to safely cut an avocado | |
| Haley | will clean up while coach wraps up with the parent. | |
| Wrap up | | 2 minutes |
| | w cooking session | |
| _ | think having [child's name] involved in the cooking | |
| process work | Ked? | |
| What did yoเ | ı like about it | |
| What didn't y | ou like about it | |
| What might b | be some ways you can do this more often? | |
| Summarize vi | | |
| As a reminder, during our next visit we will do another meal video and review and discuss routines and limits that help children eat healthier. Do you remember how to upload a meal video? Would you be able to send us another video within two weeks? | | 5 minutes |
| Let's schedule our next visit for one week after that. | | Record Next Visit in Redcap & Google calendar |
| | f the week or times of day work best for you, ind that we will take 60 minutes. | |
| | der that you will receive text messages with helpful<br>pes 2 x/week. | |
| Can I confirm | n the best number to reach you at? | |
| | erested in more information or want to connect<br>irents of children ages 2-5 you can also check out<br>k group. | |
| | | 37 |



Thank you for taking the time to meet with me.

# Visit 3 Script

## Recorder Script

(Prior to turning on recorder)

Hello, it's nice to see you again. I wanted to remind you that I will be recording the session. The recording will be used to make sure each session is delivered the same way to each family. As stated in the consent form, all of the recordings will be kept in a secure place and destroyed once we complete the study. The information from the recordings will only be shared with study staff. If you are ready, I will turn on the recorder now.

## •2 Minutes

#### Introduction

During our meeting today, we will

- 1. Check in around your goals and experience from last visit
- 2. Review your mealtime video, like what we did during our first visit
- 3. Talk a little bit about how routines and limits can help children eat healthier
- 4. Discuss if you would like to make any changes on how you feed your child.

What questions do you have?
If you have questions as we go, feel free to stop and ask me.

Assess 2-5 minutes



Tell me what you remember about our last talk about meal preparation, shopping and involving your child.

Helpful to bring copies of visit 1 handout to provide if requested.

Affirm Reflect

Thank you for sharing your experiences. It is helpful to know. It sounds like Summarize

#### Reassess

Last time we talked, you identified \_\_\_\_\_ as a goal you wanted to work on.

Last time you said this was at a level of X in importance for you. How consistent is that with how you currently feel?

Last time you said you were at a level of x confidence in meeting this goal. How consistent is that with how you currently feel?

What were some of the strategies you tried or changes you made at/after our last visit?

How did that work for you and your child?

How satisfied are you with the change you tried?

What helped you try the new (insert strategy/goal name)?

What got in the way or made it hard?

Relate to values /goals for family meals

## Summarize & Reflect

It appears there are several things that went well. You also discussed some things you want to change/areas with room for desire/need/etc. to change. improvement.

# 10 minutes

Visit 1 Goal Sheet available in Redcap under Home Visit 1 encounter.



**Key Points:** 

Identify and elicit change talk.

DESIRE: Want, wish, like ABILITY: Can, could, able

REASON: Specific reason for change

NEED: Need to, have to, must,

important, etc. (without stating specific reason)

COMMITMENT: Will, intend to, going to, etc.

ACTIVATION: Ready to, willing to (without specific commitment) TAKING STEPS: Reporting recent specific action (step) toward change

Responding to Change Talk: Explore. Ask for elaboration: how, in what ways, why? Ask for examples: when was the last time this happened

(e.g., for an adverse consequence). Affirm. Express agreement, appreciation,

encouragement, etc. for the

Reflect. This is the most common response to change talk – to offer a simple or complex reflection (. "I hear you saying that xxx" or "You feel it is difficult to xx")





Summary. Think about the conversation like a field of flowers – pick the sentences you would like to highlight. those that focus on change, and present them back to the family in a Change talk is also collected in "bouquet" summaries. You can select what to focus on in this process. Review Video Now let's take a minute to watch two clips that were chosen 15 minutes from your family meal video. We will stop between each clip and discuss what you think. Remember, only you know what's best for your family. I'm here to talk about your thoughts and Feedback Sheet experiences when feeding your child.

Play clip 1 (Positive Practices). Pause when the screen says clip 2, explore and provide feedback.

## What sticks out from the video?

Elicit thoughts about the videos process (filming a family meal and send it in to the researchers).

Prompts to explore \* if parent has already offered the information you do not need to ask the question.

What surprises you, if anything? Why?

What, if anything, did you do to get your child to eat?

What, if anything worked?

What, if anything, might you want to do differently in the future?

If it's okay with you, I would like to share some thoughts on the meal.

Wait for affirmation then share feedback on positive meal practices.

What are your thoughts about these ideas?

Now let's take a look at the second clip.

Play the second clip.



Mealtime Video Clips on I-PAD



Key Points:

Identify and elicit and respond to change talk.



## What sticks out from the video?

Elicit thoughts about the videos process (filming a family meal and send it in to the researchers).

Prompts to explore \* if parent has already offered the information you do not need to ask the question.

What surprises you, if anything? Why?

What, if anything, did you do to get your child to eat?

What, if anything worked?

What, if anything, might you want to do differently in the future?

If it's okay with you, I would like to share some thoughts on the meal.

Wait for affirmation then share feedback on negative meal practices.

What are your thoughts about these ideas?

## Summarize Feedback session

It appears there are several things that you are doing well and ...

We also discussed some areas with room for improvement and you feel this information is ...

Thank you for sending this video in.

This was a great discussion. I also have some printed materials that you might be interested in.



## Routines & Limits

The topics for this week's materials are - routines and limits.

Tell me a little bit about your family's meal / snack routine?

What challenges do you have sticking with a routine?

What helps keep your child on a routine?

What limits or rules do you have about food or meals in your house?

How do those limits or rules work for your family?

If it is okay with you, I would like to share some information about how routines and limits can help children learn and grow into healthy eaters.

# Review Visit 3 handout

Routines and limits can be hard to start, but can make things much easier for you, your child and your family in the long run. This visit's handout has some tips for creating routines and setting limits around meals and snack times.

> Review handout with parent, "structure for strong families-Tips for planning a routine

We hear from many families that getting children to come to the table, or not snack all the time can be really challenging. One thing that can help is having a routine. This is an outline of your time that helps you and your child know what is coming throughout the day. Kids may resist routines at first but often enjoy them, if they go to school they will have to get used to the handout for the goal setting activity. routines there.

Structure for Strong Families Tips for planning a routine Structure for strong families- Rules and limits

Identify and elicit change talk. It may be helpful to check off changes the family is interested in making on the



Every family is different and so are their routines. Some suggestions on the handout include having set times for meals and snacks, having fun routines that your child looks forward to, like walks after dinner or trips to the park. We also know that young children can sometimes have a hard moving from one activity to another, routines can help with this. For example, instead of going straight from playing to dinner you could have a routine such as: turning off the TV, cleaning up, washing hands and setting the table to let kids know that mealtime is coming.

Time Management Tip
Reflections and exploration of parents'
thoughts on the content are written into
the script -- if time is limited would be OK
just to provide the handout with brief
explanation.

What, if any, strategies have your family tried?

Affirm. reflect

What suggestions on here are you interested in trying or have thought about?

Affirm, reflect

What concerns do you have about the recommendations?

Affirm, reflect

Review handout with parent, "structure for strong families-Rules and limits"

Another way to create structure around meals and snacks is by having some family rules. This is a clear statement about the behavior that you expect from your child. This can teach them what behaviors are ok and not ok. Some examples of rules are: screens should be off at meal times, everyone eats together, or everyone helps clean up.

When coming up with rules it is important to explain to your child what you expect of them, follow the rule yourself, and remind them of the rules often. Children will often break the rules or test limits, this is normal. Don't worry if you are consistent with the rules and remind them often they will learn. Here is a place where you could write down which mealtime rules are important to your family.

Show the cartoon on the back of the handout.



Here you can see an example of how a mealtime rule can help children.

What, if any, strategies have your family tried?

Affirm, reflect

What suggestions on here are you interested in trying or have thought about?

Affirm, reflect

What concerns do you have about the recommendations?

Affirm. reflect

# Problem Solving/ Goal Setting

Thinking about what we talked about today; including routines, rules and limits, would you like to set a goal?

If parent identified many changes they were interested in making have them rank which are most important to them, choose 1-2

Can choose from strategies on handout or participants own goal that aligns with performance objectives.

Remember they should choose at least one goal but if they have more than one they have work on two goals.

Why do you want to make this change? (Reflection)

How might you be able to do it? (Reflection)

What is one good reason for making the change? (Reflection)

**How important is it, and why?** (0-10) (Need) (Record number) (Reflection)

What do you intend to do? (Reflection)

#### 15 minutes



**Goal Sheet** 

Keys for Goal Setting: Goals should be:

- Specific: Make sure goals are detailed. (Who, What, When, Where)
- Measurable: Make sure the participant can identify what will happen when they achieve their goal.
- **3.** <u>Achievable</u> Goals should be realistic, not ideal
- 4. Relevant Goals should relate to best practices for feeding and nutrition 5. Time Bound Goal should have a timeline of when it will be met within the

next time you meet

Performance Objectives: As part of the study we want participants to achieve the following

 Determine when and where children eat.

44



# Provide limited and guided What are you ready or willing to do? choices to their child (Reflection) Teach children about healthy meals What have you already done? Limit screens at meals (Reflection) Provide positive reinforcement when eating healthy food Record specific goal (s) from the bottom of the goal setting sheet on the data sheet. The goal of this section is to Record Goal in Redcap Upload develop a specific goal and identify barriers/ strengths. picture of goal sheet (if more than one goal record both) Leave the goal setting sheet (s) with the parent & take a picture. So, your goal is to... (insert goal from last line on goal setting sheet). When I call next month, we will review this goal so keep this sheet with your materials. You can always use your magnet to put it up on the fridge. Assess Readiness to Make Change 15 minutes Record Readiness in Redcap Motivation Now that you have set a goal about \_ [insert topic] family, I would like to know how you are feeling right now about Record **Motivation** # in Redcap [insert name of goal] Record Confidence # in Redcap On a scale of 1 to 10 where 1 means you do not want to do this at all and 10 means you really want to do this. Record Barriers in Redcap How would you rate yourself? (Readiness) What made you pick that number and not a lower number (like 1 Record **Facilitators** in Redcap or 2)? (Motivation) Confidence On a scale of 1-10, rate your confidence or ability to finsert name \_, where 1 means you are not at

all confident and 10 means you are very confident you can

maintain that change.

How would you rate yourself?



What made you pick that number and not a lower number (like 1 or 2)? (Barriers)

What would it take to get to a higher number (like 8 or 9)? If a 10 What would it take to keep you at a 10? (Facilitators)

# Sample Summary

You feel that you are very motivated to make this change because you (first part of rating). You could (insert comments from parent). In terms of being able to make this change, you feel that you are able to make this change because (first part of 1 or 2) You believe you could increase your confidence if (insert comments from last part 9 or 10). You think that (barrier) may make it challenging but identified (solution) as something that could help.

# Wrap up

It has been a pleasure meeting with you and your family. I will be checking in by phone for the next 3 months to check in on goals, problem solve and cheer you on. Are there good days of 5 minutes the week or times of day to call? Can I confirm the best number to reach you at?

Just a reminder that you will continue to receive text messages with helpful tips and recipes 2 x/week. If you are interested in more information or want to connect with other parents of children ages 2-5 you can also check out our Facebook group.

Record Next Visit in Redcap & Google calendar

Thank you for taking the time to meet with me. Before I leave, we would like to ask you to answer some questions on the IPAD.

Complete Visit Satisfaction Questionnaire

Phone Call Script



| Recorder Script | | | |
|---|---|---|---|
| (Prior to turi | ning on recorder) | | |
| | | | 5 Minutes |
| Families Start at F<br>calling to do our n<br>today. I wanted to<br>ready I will turn or<br>the mail, if you ha<br>you have your goa<br>Introduction | name is name is nome Study with the Univers nonthly phone call. Thank you remind you that I will be red the recorder now. We sent we them around we can refer al setting sheet, we will also to know if you received your | ity of Rhode Island. I amou for talking with me cording the call. If you are you some materials over to them during the call. If be using it during the call. | Goal Sheet available in Redcap under previous Home Visit encounter. |
| Record Red | Cap: Yes / No read through the newsletter? | | Key Points:<br>Restate goal, and review<br>motivation and confidence. |
| Do you have any o | questions about the newslett | ers? | Record if read |
| useful, a little, or r | ne newsletter? Would you sa<br>not at all useful?<br>select one of the response op | | newsletter and texts.<br>Record their usefulnes <b>s</b> . |
| Did you receive th<br>Record: Yes | e text messages?<br>s / No | | Record on redcap if they met their goal: Circle Yes/ No |
| Did you read the to<br>Record: Yes | ext messages? If no, why nos / No | t? | |
| useful, a little, or r | he messages? Would you sanot at all useful? select one of the response op | | |
| | issues or questions?<br>eview of the goal you talked ab | oout in the last visit. | |

Example: "Last time we spoke, you mentioned that you wanted to prepare more meals with your child. You hoped this would get child's name excited about trying new vegetables. Your goal was to prepare a



meal together 2 x/week You also said that you were somewhat motivated to make this change (rated at 7) but did not feel very confident that you could do it every week (rated at 3). How did you do with your goal?

On a scale of 1 to 10, What would you say your motivation level is now for preparing meals with your child? What would you say your confidence level is now?

Use a reflection or an open-ended question to increase your understanding of how the participant is working on the goal. If the participant had problems with the goal:

What do you think you could try differently next time?
Wrap up the topic

Provide summary of progress and transition to the next goal.

Example: It sounds like you were able to meet your goal on this topic and are pleased with your progress. How do you feel about the material you got in the mail?

# Review New Topic

We sent some information on (insert handout name). It reviews some of the topics we talked about during our sessions including (insert topics from targeted handout).

How do you feel about setting a goal for this topic?

Performance Objectives: As part of the study we want participants to achieve the following.

- Increase fruits and vegetables, whole grains, lean proteins served
- Increase accessibility of fruits and vegetables
- Decrease accessibility of treat foods
- Offer choices of healthy options
- Increase family meals/ role modeling
- Have a set location where the family eats, like a table or counter.
- Limit distractions like the TV, tablet, or computer
- Serve small portions and practice letting the child decide when he/she's full.
- Increase family meals
- Increase modeling of healthy foods
- Increase preparing meals
- Increase inclusion of vegetables

2 minutes



Month 4 handout Month 5 handout Month 6 handout



Identify and elicit change talk. It may be helpful to check off changes the family is interested in making on the handout for the goal setting activity.



- Talk to children about benefits of foods
- Involve child in food preparation
- Determine when and where children eat.
- Provide limited and guided choices to their child
- Teach children about healthy meals
- Limit screens at meals
- Provide positive reinforcement when eating healthy food

# Problem Solving/ Goal Setting

Now I would like to talk to you about setting a goal to address the next/new topic you selected (repeat the topic and objective here).

Why do you want to make this change? (Desire) (Reflection)

How might you be able to do it? (Ability) (Reflection)

What is one good reason for making the change? (Reasons) (Reflection)

**How important is it, and why?** (0-10) (Need) (Record number) (Reflection)

What do you intend to do? (Commitment) (Reflection)

What are you ready or willing to do? (Activation) (Reflection)

What have you already done? (Taking Steps) (Reflection)

Record specific goal on the bottom of the goal setting sheet. Record this specific goal on the redcap. The goal of this section is to develop a specific goal and identify barriers.

So, your goal is to: (insert goal from last line on goal setting sheet).

# 15 minutes



**Goal Sheet** 



1. Specific: Make sure goals are detailed. (Who, What, When, Where)
2. Measurable: Make sure the participant can identify what will happen when they achieve their goal.

Setting: Goals should be:

- Achievable Goals should be realistic, not ideal
- 4. Relevant Goals should relate to best practices for feeding and nutrition 5. Time Bound Goal should
- have a timeline of when it will be met within the next time you meet



| What might get in the way of you meeting your goal to {restate goal}? | Record <b>Goal</b> in Redcap<br>Upload picture of goal<br>sheet (if more than one<br>goal record both) |
|---|---|
| Motivation Now that you have set a goal about _ [insert topic], I would like to know how you are feeling right now about _ [insert name of goal] | 15 minutes Record Readiness in Redcap Record Motivation # in |
| On a scale of 1 to 10 where 1 means you do not want to do this and 10 means you really want to do this. How would you rate yourself? What made you pick that number and not a lower number (like 1 or 2)? What would it take to get to a higher number (like 8 or 9)? If a 10 What would it take to keep you at a 10? | Redcap Record Confidence # in Redcap Record Barriers in Redcap Record Facilitators in Redcap |
| On a scale of 1-10, rate your confidence or ability to, where 1 means you are not at all confident | · |
| and 10 means you are very confident you can maintain that change. How would you rate yourself? | |
| What made you pick that number and not a lower number (like 1 or 2)? | |
| What would it take to get you to a higher number (like 8 or 9)? | |
| Sample Summary You feel that you are very motivated to make this change because you (first part of rating). You could (insert comments from caregiver). | |



In terms of being able to make this change, you feel that you are able to make this change because (first part of 1 or 2) You believe you could increase your confidence if (insert comments from last part 9 or 10). It seems you are ready to make this change and are committed to making this change. Wrap up 2 minutes You will receive a handout mailing in about 1-2 weeks. You will also continue to receive the text messages. You can also check out our Facebook page for tips, recipes, and to connect with other caregivers. About 2 weeks after you will receive another newsletter, I will call you again to review your goal and discuss the next topic you want to work on Record **Next Visit** on and set some new goals for that topic. Be sure to have your goal setting redcap and Google sheet to fill out during our phone call. calendar. What would be the best day and time for our next call? \*Note for last phone call \_\_\_\_ (Note date of call) schedule per data Best phone number: \_ collection team calendar Thank you for taking the time to meet with me. I will talk with you again soon by phone.



# Intervention Text Messages

| Message Delivery Scheduled | Message Content English |
|---|---|
| Week 1 - Welcome | *****welcome***** |
| Week 1 - Message 1 | Food tastes best when we're hungry! If your kids are starving when they come home from school, try serving sliced fruits and vegetables. |
| Week 1 - Message 2 | Whole grains are inexpensive and very nutritious! Check out this link for whole grains that cook in less than 15 minutes for a quick healthy dinner. <a href="https://wholegrainscouncil.org/blog/2015/09/whole-grains-quick-and-easy">https://wholegrainscouncil.org/blog/2015/09/whole-grains-quick-and-easy</a> |
| Week 2 - Message 1 | Did you know beans, peas, and nuts are great sources of protein? Add them to dishes like tacos, pastas, and soups for a nutrition boost. |



| Week 2 - Message 2 | Parents provide, and kids decide! If you are offering healthy meals and snacks to your child, you are doing your job! It's up to them to eat it. or not. |
|---|---|
| Week 3 - Message 1 | Raising healthy eaters isn't easy, but it's worth it. You're doing a great job! |
| Week 3 - Message 2 | Soups are a great way to use up leftover vegetables before they go bad. Try this recipe, kids can help strain the beans. <a href="https://youtu.be/wjk4QanUJak">https://youtu.be/wjk4QanUJak</a> |
| Week 4 - Message 1 | Remember that you decide when, where and what your child eats but it's up to them if they will eat it. It is normal for appetites to change a lotdon't worry if they don't eat much at one meal. |
| Week 4 - Message 2 | Frozen broccoli is just as healthy as fresh broccoli! Microwave until tender & toss with some olive oil, lemon juice, garlic powder, salt & pepper! |
| Week 5 - Message 1 | Your kids look up to you! Set another good example for your kids by eating fruits and vegetables every day. |



| Week 5 - Message 2 | https://www.youtube.com/watch?time_continue=55&v=qN566WU5U Try to make this yummy salad with your kids this week. Kids can tear up the kale, squeeze the lemon, and mix the ingredients. |
|---|---|
| Week 6 - Message 1 | Try to plan 2-3 dinners for this week. Ask your kids to pick a vegetable dish to go on the side. |
| Week 6 - Message 2 | Do you worry your child won't believe you when you tell them how great fruits and vegetables are? Maybe they will listen to their peers. Check out this video of kids in RI talking about their favorite healthy foods. <a href="https://www.youtube.com/watch?v=m4u0pjjaSik">https://www.youtube.com/watch?v=m4u0pjjaSik</a> |
| Week 7 - Message 1 | Preparing foods in different ways can totally change the way it tastes! Pick a vegetable as a family and try it raw, roasted, grilled, steamed, or sautéed. Don't be afraid to add your favorite seasonings or dressings, vegetables can taste yummy! |
| Week 7 - Message 2 | Serving new vegetables with foods kids already like is one way to help them try and enjoy these foods. Check out this recipe that combines pasta, cheese and broccoli all together! <a href="https://youtu.be/oPVd7YfW4rU">https://youtu.be/oPVd7YfW4rU</a> |
| Week 8 - Message 1 | Did you know that kids need to taste foods up to 8 times before they know whether or not they like it? Even tiny bites help get their taste buds used to new foods. |



| Week 8 - Message 2 | Kids eat things that are easy to get. Having peeled oranges or sliced pepper strips in the refrigerator can make after school snacking easy and healthy! |
|---|---|
| Week 9 - Message 1 | Shopping lists can help us be prepared and save money! Use our paper template, the notes section on your phone or try an app like Yummy or OutofMilk. Many grocery stores even have their own apps or websites! |
| Week 9- Message 2 | Check out our facebook page to see what families are doing to stay healthy! https://www.facebook.com/groups/680745735718231/ |
| Week 10- Message 1 | Does your child constantly ask for treats like chips, cookies, or soda? The best way to avoid arguments about these foods is to keep them out of your home. |
| Week 10- Message 2 | Kids who eat more meals with their families do better in school, have higher self-esteem and lower risks of depression. |
| Week 11- Message 1 | Family meals don't have to be fancy! The important thing is that you eat together. |
| Week 11- Message 2 | Kids are easily distracted! Turning off the TV or tablet can help them focus. |
| Week 12- Message 1 | Avoid bribes and rewards for eating. Although it might be tempting to offer a cookie if your child eats 3 bites of spinach, this makes kids think that "treats" are more valuable than mealtime food. |
| Week 12- Message 2 | There are no perfect parents, and there are no perfect children, but there are plenty of perfect moments along the way Dave Willis |



| Week 13- Message 1 | Be prepared - children don't always follow the rules!! Show them what you want them to do and remind them often. It will get easier! |
|---|---|
| Week 13- Message 2 | It is hard to get dinner on the table every night! Check out our recipe book for dinners you can prepare in less than 30 minutes! |
| Week 14- Message 1 | Think beyond a single meal. Keep in mind what your child eats over the course of a week. |
| Week 14- Message 2 | Serve new foods with foods your child already likes. If your child's favorite vegetable is corn they might like this recipe! English <a href="https://www.foodnetwork.com/videos/bean-corn-and-tomato-salad-0274222">https://www.foodnetwork.com/videos/bean-corn-and-tomato-salad-0274222</a> |
| Week 15- Message 1 | Let go a little to gain a lot. Giving your child choices and allowing them to decide how much to eat will help them grow into adventurous healthy eaters |
| Week 15- Message 2 | New foods take time. Offer new foods with foods your child already likes so they can fill their bellies and explore the new food at their own pace. |
| Week 16- Message 1 | Patience works better than pressure when it comes to feeding young children. |
| Week 16- Message 2 | Cook together. Eat together. Talk together. Make mealtime family time. |
| Week 17- Message 1 | They learn from watching you. Eat fruits and veggies and your kids will too |
| Week 17- Message 2 | Take it with you. Show your child how whole fruit is a great snack to eat at the park or in the mall. Put apples, oranges, or bananas in your bag for quick snacks |
| Week 18- Message 1 | Feed your child's independence at meal time. Let them choose from the healthy foods you offer. |
| Week 18- Message 2 | Offer young kids the same healthy food the rest of the family is having. Your child may not like everything offered but that is OK |
| Week 19-Message 1 | It's normal for 2-5-year olds to be "picky" eaters. Help them increase the types of fruits and vegetables they eat by eating them yourself! |
| Week 19-Message 2 | Water doesn't have to be boring. Add sliced citrus or frozen berries to water to add flavor without added sugar. |
| Week 20- Message 1 | Make meals and memories together. It's a lesson they'll use for life! |
| Week 20- Message 2 | Pass the Pasta – Try different shapes and colors of whole wheat pasta. Sprinkle it with a little olive oil and low-fat cheese. Add chopped veggies and spices or tomato sauce for a quick lunch or dinner. |



| | Structure helps parents and their kids. Kids feel safe and secure because |
|---|---|
| Week 21- Message 1 | they know what to expect. Parents feel confident because they know |
| | how to respond, and they respond the same way each time |
| | Many parents have a hard time getting their kids to come to the dinner |
| Week 21-Message 2 | table. Routines such as washing hands and setting the table before sitting |
| | can help kids transition from one activity to the next. |
| Wook 22 Mossage 1 | Keep chips and sweets out of the house. It will help kids learn that these |
| Week 22- Message 1 | foods are not meant to be eaten every day. |
| Week 22 Messes 2 | Make your own trail mix by combining whole grain cereal, nuts or seeds |
| Week 22- Message 2 | and dried fruit. It is a yummy snack that is easy to bring on the go. |
| Wash 22 Massas 4 | Starting with small portions on the plate can help you avoid wasting food |
| Week 23- Message 1 | if your child isn't hungry at meal time. |
| | Kids can make good choices if you give them a chance! Let them choose |
| Week 23- Message 2 | how to try new foods, "Do you want to try broccoli cooked with your |
| | pasta or raw with dip" |
| | Try this: At family mealtime, have questions for everyone to answer, for |
| Week 24- Message 1 | example: What is your favorite food tonight? or What was the best part |
| | of your day? |
| Week 24- Message 2 | Healthy meals can be easy and quick to prepare. Try eggs, beans, salsa |
| Week 24- Wessage 2 | and low-fat cheese with a tortilla for a My Plate meal everyone will love. |
| Week 25- Message 1 | Prioritize a pleasant meal—don't worry about counting bites or worrying |
| Week 25- Wessage 1 | about what your child has (or hasn't) eaten. |
| | Nobody's got time for a second job as a short-order cook. Serve the same |
| Week 25- Message 2 | foods to everyone in the family. If your child doesn't like a dish, try |
| | serving a side that they like such as fruit or beans |
| | Your job is to offer a variety of foods. Your child's job is deciding how |
| Week 26- Message 1 | much to eat. There will be days when they only want to eat one food and |
| WEEK 20- WIESSAGE 1 | that's OK. As long as you continue to provide healthy meals and snacks |
| | they will get what they need. |
| Week 26- Message 2 | Thank you for participating in the Strong Families Start at Home Study! |



# Materiales para la Intervención en Español

Nota: Para todos los guiones del estudio, la "negrita" o bolding se utiliza para indicar lo que la consejera debe estar diciendo y las frases "en cursiva" o italics son instrucciones para el entrenador



# Guión de Grabación:

(Antes de encender grabadora)

Muchas gracias por reunirse conmigo el dia de hoy. Le quiero recordar que estaré grabando esta sesión. Esta grabación será utilizada para asegurarnos que cada sesión es llevada a cabo de la misma manera con cada familia. Como se indica en el formulario de consentimiento, todas las grabaciones se mantendrán en un lugar seguro y serán destruidas una vez que completemos el estudio. La información de las grabaciones será únicamente compartida con el personal del estudio. Si está listo encenderé la grabadora ahora.

## Introducción

Hola Señor/ Señora \_\_\_\_\_ mi nombre es \_\_\_\_\_ y soy su consejera del estudio Familias Fuertes Comienzan en Casa de la Universidad de Rhode Island. El día de hoy nos reuniremos por alrededor de 1 hora. Estaremos viendo cortos de los videos que nos mandó y discutiremos sus opiniones y las inquietudes que tenga sobre la alimentación de su hijo(a). También estaremos hablando sobre alimentación saludable y estrategias para ayudarle a que su hijo(a) coma saludablemente.

Refiérase a Cronograma del estudio:

Después de la reunión de hoy, nos reuniremos una vez al mes por los próximos dos meses para discutir la preparación de alimentos, compra de comida y estrategias para ayudarle a alimentar a su hijo(a). También recibirá mensajes de texto con información para usted y su hijo(a). Después de la tercera visita, en vez de venir a su casa, lo/la estaré llamando una vez

#### 5 Minutos



Utilice el cronograma del estudio



al mes para revisar sus metas, resolver problemas y darle ánimos. También le estaremos mandando por correo materiales adicionales y al finalizar el estudio, usted recibirá una visita final con el personal de investigación para recolectar la misma información que en la primera visita.

¿Qué preguntas tiene sobre el estudio?

# Día Típico

Primero, me gustaría conocer un poco acerca de las comidas de su familia.

¿Cómo describiría una comida típica con (nombre del niño(a)? problemas, nuestra meta es: Recopilar Si el participante no está seguro de cómo responder:

¿Cuénteme sobre la cena de ayer? o Comparta conmigo cualquier cosa que considere importante acerca de sus comidas con (nombre del niño(a)

> Pídale al participante que le cuente su historia. Interrumpa lo menos posible. Utilice preguntas abiertas para que sigan hablando (ejemplo "¿Qué pasa después?", "Cuéntame más.")

Cuando piensa en una comida típica con (nombre del niño(a), ¿qué partes/momentos de la comida funcionan bien?

Interrumpa lo menos posible. Utilice preguntas abiertas para que sigan hablando (ejemplo "¿Qué pasa después?", "Cuéntame más."

Al pensar en una comida típica con (nombre del niño(a), ¿qué partes/momentos de la comida no funcionan tan bien?

Utilice preguntas abiertas para que sigan hablando (ejemplo "¿Qué pasa después?", "Cuéntame más."

Gracias por compartir sus experiencias. Siento que entiendo mucho mejor sus comidas. Pareciera que...

Resuma la descripción general de las comidas, destacando las fortalezas and barreras.

#### 5 minutos



Puntos Claves: No intente resolver problemas, nuestra meta es: Recopilar información y hacerles saber que se les está escuchando. Presta atención a sus retos y preocupaciones.

Transmite un tono sin criticar.



## Revisión del Video

Ahora tomemos unos minutos para ver dos clips que fueron elegidos del video de su comida familiar. Haremos pausas entre cada corto/clip y discutiremos lo que usted piensa sobre el corto/clip. Recuerde, sólo usted sabe lo que es mejor para su familia. Estoy aquí para hablar con usted de lo que piensa y sus experiencias al alimentar a su hijo(a).

Reproduzca el corto/clip 1 (Practicas Positivas). Haga una pausa cuando la pantalla diga corto/clip 2, explore y provea retroalimentación.

# ¿Qué sobresale del video?

Obtenga las ideas y opiniones sobre el proceso de filmación (filmar una comida familiar y mandarla a los investigadores).

Indicaciones para explorar \*si el padre ya ha brindado la información, no necesita hacer la pregunta.

#### Explore:

¿Qué le sorprende? ¿Por qué?

¿Qué hizo para que su hijo(a) comiera?

¿Qué funcionó?

¿Qué es lo que, en todo caso, querría hacer de manera diferente en el futuro?

Si te parece bien, me gustaría compartir algunas ideas sobre este tiempo de comida.

Espere la afirmación, luego comparta retroalimentación sobre prácticas de comidas positivas.

¿Qué piensas de estas ideas?

Ahora, observemos el segundo clip.

Reproduzca el segundo clip del video.

¿Qué sobresale del video?

#### 15 minutos



Use la hoja con retroalimentación

Cortos del video de comida familiar en el I-PAD



#### **Puntos Claves**

Identificar y provocar el cambio en la conversación.

<u>DESEO</u>: Querer, desear, gustar HABILIDAD: Poder, podria

RAZON: Razon especifica para el cambio NECESIDAD: Necesitar, tener que, deber, importante, etc. (sin indicar la razón específica)

COMPROMISO: Voluntad, intención de, ir a. etc.

ACTIVACIÓN: Listo para, dispuesto a (sin compromiso específico)

TOMANDO MEDIDAS: Reportar acción específica reciente (paso) hacia el cambio Respondiendo a plática de cambio:

Explorar. Pida una explicación: ¿cómo, de ¿qué manera, por qué? Pida ejemplos: cuándo fue la última vez que sucedió esto? (por ejemplo, para una consecuencia adversa).

<u>Afirmar.</u> Expresar acuerdo, agradecimiento, ánimo, etc. para el deseo/necesidad de cambio.

Reflexionar. Esta es la respuesta más común sobre la conversación de cambio: ofrecer una reflexión simple o compleja. ("Lo escucho decir que xxx" o "Siente que es difícil xx")

Resumen. Piense en la conversación como un campo de flores: elija las oraciones que



Obtenga las ideas y opiniones sobre el proceso de filmación (filmar una comida familiar y mandarla a los investigadores).

Indicaciones para explorar \*si el padre ya ha brindado la información, no necesita hacer la pregunta.

desea resaltar, las que se centran en el cambio y preséntalas a la familia en un resumen como en un "ramo". Puedes seleccionar en qué enfocarte en este proceso.

Explore:

¿Qué le sorprende? ¿Por qué?

¿Qué hizo para que su hijo/a comiera?

¿Qué funcionó?

¿Qué es lo que, en todo caso, querría hacer de manera diferente en el futuro?

Si te parece bien, me gustaría compartir algunas ideas sobre la comida.

Espere la afirmación, luego comparta retroalimentación sobre prácticas de comidas negativas.

¿Qué piensas de estas ideas?

Resumen de la sesión de comentarios

Parece que hay varias cosas que está haciendo bien y ... También discutimos algunas áreas con margen de mejora y usted siente que esta información es ...

Gracias por enviar este video.

Esta fue una gran discusión. También tengo algunos materiales impresos que le pueden interesar.



# Revisión de materiales impresos

Durante esta parte de la visita, usted proporcionará información y proporcionará algunos materiales.

Hemos escuchado de otros padres que las comidas a veces pueden ser estresantes. Algunos estudios sugieren que entendiendo cuáles son los roles de los padres y los niños durante las comidas puede hacer que las comidas sean menos estresantes.

# ¿Puedo compartir un poco más sobre esto?

Proporcione "¡Criar un niño sano no tiene que ser estresante!"

Esta primera página dice que el rol de los padres es decidir qué, dónde y cuándo comen los niños. Usted está a cargo de la comida que entra a su casa y de lo que su hijo come durante las meriendas y las comidas.

Si le preocupa que su hijo no coma lo que usted eligió, hay algunas cosas que puede hacer para ayudarlo. Puede ofrecerle opciones saludables, servir nuevos alimentos con alimentos que ya le gustan a su hijo y modelar hábitos alimenticios saludables - los niños siempre quieren copiar a sus padres.

También dice que su hijo es el responsable de decidir cuánto come y de aprender a comportarse durante las comidas. Puede ser difícil permitir que su hijo decida cuánto va a comer, ya que muchos padres se preocupan de si su hijo/a va a comer lo suficiente. Recuerde que si les proporciona 3 comidas y 2-3 meriendas al día, ellos obtendrán suficientes alimentos para crecer y mantenerse sanos.

El folleto también ofrece algunos consejos para hacer que las comidas sean más agradables.

Por ejemplo, comer con su hijo tan a menudo como sea posible, tener horarios específicos para las comidas y las

#### 15 minutos

¡Criar un niño sano no tiene que ser estresante!



Identifique y promueva conversación de cambio. Puede ser útil marcar las estrategias que la familia hace o ha intentado. Destaque los cambios que la familia está abierta / interesada en hacer.



meriendas, tener un lugar definido para comer como el comedor o la cocina, limitar distracciones como la TV, tableta o la computadora, y colocar pequeñas porciones en el plato de su hijo y dejar que pida más si todavía tiene hambre.

Puede ver un ejemplo en la parte posterior de la hoja de como ofrecer opciones guiadas puede ayudar a los niños a tomar decisiones saludables.

Enseñe a los padres la caricatura en la parte de atrás de la hoja.

Explore opiniones e ideas sobre el folleto.

¿Qué piensa sobre esto?

¿Qué preocupaciones tiene sobre las recomendaciones?

¿Qué estrategias, si las hay, ha intentado su familia?

¿Qué sugerencias está interesado o ha pensado en probar?

Enseñe folleto "La Alimentación Saludable Comienza en Casa- Mi Plato"

También sabemos que muchos padres quieren saber cuáles alimentos son saludables para sus hijos. Este segundo folleto habla un poco más sobre la alimentación saludable y cómo mantener a su familia sana. Se basa en "Mi Plato", el cual nos dice que lo que comemos debería ser principalmente granos enteros, frutas, vegetales, proteínas magras o sin grasa, y lácteos sin grasa o con poca grasa. También incluye consejos acerca cómo incluir más de estos alimentos saludables en la alimentación de su familia.

En el otro lado del folleto, se habla acerca de cómo limitar los alimentos que no son tan saludables para nosotros, como alimentos con azúcares agregados y grasas, por ejemplo, postres, chips o papitas, gaseosas, jugos/refrescos y comidas frita. Esto hace que sea más fácil para tus hijos limitar estos alimentos al mantenerlos afuera de tu hogar. Al

La Alimentación Saludable Comienza en Casa- Mi Plato

Consejo para manejo del tiempo:
Las reflexiones y la exploración de los
pensamientos y opiniones de los padres
sobre el contenido están en el guión - si el
tiempo es limitado, está bien proporcionar
solamente una breve explicación del folleto.



no tenerlos cerca, puede evitar que sus hijos estén pidiendo siempre dulces o chips. También hay algunos consejos sobre cómo puede modelar una alimentación saludable, la cual es una manera de ayudar a sus hijos a comer de manera saludable.

Enseñe folleto "La Alimentación Saludable Comienza en Casa" (con sandía)

Explore opiniones e ideas sobre el folleto.

¿Qué piensas sobre esto?

¿Cuáles son sus pensamientos sobre esto?

¿Qué preocupaciones tiene sobre las recomendaciones?

¿Qué estrategias, si las hay aquí, ha intentado su familia?

¿Qué sugerencias de aquí está interesado en probar o ha pensado en probar?

# Folletos específicos

Si al(la) niño(a) se le ha asignado un rasgo apetitivo, lea el guión correspondiente y proporcione un folleto adicional. Esto no es para todos los niños.

¿Estaría bien compartir alguna información adicional específica para su hijo(a)?

Espere respuesta



## Inquietud por la comida

En nuestra primera visita, le pedimos que respondiera algunas preguntas sobre la alimentación de su hijo(a). En base a esas respuestas, su hijo(a) tiene tendencias de ser "caprichoso con la comida".

Ser caprichoso con la comida es una etapa normal para muchos niños. Por lo general, es peor a los 2 años y disminuye a los 5 años. Pero su encuesta nos dice que su



# Folleto para cada rasgo

Consejos útiles para niños caprichosos con la comida



hijo(a) puede ser más caprichoso con la comida que otros niños. Esto quiere decir que a ellos solo les pueden gustar ciertos alimentos o tienen miedo de probar nuevos alimentos. ¡Su hijo(a) puede rechazar alimentos o incluso dejar de comer alimentos que solía amar!

A los padres les preocupa que a niños que tienen esta tendencia reciban suficiente nutrición. A veces los padres intentan que sus hijos coman, forzándolos a comer lo que hay en el plato. Pero, por lo general, eso hace que los caprichos con la comida empeoren a largo plazo.

Proporcione el folleto de "Consejos útiles para niños que siempre quieren comida."

Sensibilidad a la saciedad

En nuestra primera visita, le pedimos que respondiera algunas preguntas sobre la alimentación de su hijo(a). Basándose en esas respuestas, su hijo(a) puede tener más problemas para sentir saciedad después de comer. La sensibilidad a la saciedad es lo que permite que un niño(a) sepa si está lleno o tiene hambre. Algunos niños pueden tener dificultades para saber cuándo están llenos. Puede ser tentador restringir su alimentación para ayudarlos, pero esto puede ser perjudicial.

Proporcione el folleto de "Consejos para ayudar a tu hijo con una alimentación consciente"



Respuesta de Alimentos

En nuestra primera visita, le pedimos que respondiera algunas preguntas sobre la alimentación de su hijo(a). Basándose en esas respuestas, para su hijo es difícil resistir comidas deliciosas cuando están en su alcance. Comparado a otros niños, su hijo(a) puede reaccionar más fuertemente a los alimentos que ve o huele. A muchos padres les preocupa que estos niños coman demasiados alimentos que saben

Consejos para ayudar a tu hijo con una alimentación consciente

Consejos útiles para niños que siempre quieren comida.



bien pero que no son saludables (como dulces o papas fritas). Los padres pueden intentar restringir estos alimentos, pero esto puede ser perjudicial. A medida que los niños se sienten más restringidos, ¡sienten que quieren esos alimentos aún más!

Proporcione folleto "¿Cómo hacer que tu entorno funcione para ti y tu familia?"

Resolución de problemas / establecimiento de metas

Ahora me gustaría hablar con usted sobre el establecimiento de una meta para abordar el tema que mencionó que desea cambiar

Si los padres identificaron varios cambios que le interesaron, haz que clasifiquen los más importantes para ellos, desde el más importante al menos importante para ellos, elija 1-2

Puede elegir entre las estrategias del folleto o entre las metas propias de los participantes que se alinean con los objetivos de desempeño.

Deben centrarse en 1 meta, pero si deciden trabajar en 2 metas, escriba ambas y haga las mismas preguntas para cada uno.

¿Por qué quiere hacer este cambio? (Deseo) (Reflexión)

¿Cómo podría hacerlo? (Capacidad) (Reflexión)

¿Cuál es una buena razón para hacer el cambio? (Razones) (Reflexión)

¿Qué tan importante es, y por qué? (0-10) (Necesidad) (Número de registro)

## 15 minutos

Hoja de establecimiento de metas y los materiales de la sesión 1

ŧ

Guía para el establecimiento de metas. Las metas deberían ser:

- 1. Específico: Asegúrese de que las metas estén detallados. (Quien, que, cuando, donde)
- 2. Medible: Asegúrese de que el participante pueda identificar lo que sucederá cuando logre su meta.
- 3. Realizable: Las metas deben ser realistas, no ideales.
- Relevante: Las metas deben relacionarse con las mejores prácticas de alimentación y nutrición.
- 5. Límite de Tiempo:La meta debe tener un plazo de tiempo de cuándo se cumplirá (para la próxima visita)
- \*Si los padres escogen un comportamiento (por ejemplo, modelar o ejemplificar un comportamiento saludable) y una meta



# (Reflexión)

Registre la meta específica en la parte inferior de la hoja de establecimiento de metas en la hoja de datos. La meta de esta sección es desarrollar una meta específica e identificar barreras. Deje la hoja de determinación de metas con el padre y tome una foto.

relacionado a un alimento (por ejemplo, disminuir bebidas gaseosas), lo ideal sería combinarlos a una sola meta: "Modele una alimentación saludable al no toma bebidas gaseosas durante la cena".

Objetivos de rendimiento: como parte del estudio, queremos que los participantes cumplan lo siguiente:

 Incrementar frutas y verduras, granos integrales, proteínas magras servidas.

Aumentar la accesibilidad de frutas y

- verduras.
- Disminuir la accesibilidad de los alimentos procesados y golosinas
- Ofrecer opciones saludables.
- Aumentar las comidas familiares / modelando los roles
- Tener un lugar fijo donde la familia come, como la mesa o el mostrador.
- Limitar las distracciones como televisión, tableta o computadora
- Servir porciones pequeñas y dejar que el/la niño/a decida cuándo esté lleno/a

Registre **Meta y su importancia** en Redcap. Suba una foto de la hoja de metas (si es más de 1 meta, registre ambas)



| Evaluar la preparación para hacer el cambio | 15 minutos |
|---|---|
| Motivación | Registre # Preparación en Redcap |
| Ahora que ha establecido una meta sobre _ [insertar tema] para su familia, me gustaría saber cómo se siente en este momento acerca de [insertar nombre de la meta] En una escala de 1 al 10, donde 1 significa que no quiere hacer esto y 10 significa que realmente quiere hacer esto. ¿Cómo se calificaría? (Preparación) ¿Qué le hizo elegir ese número y no un número más bajo (como 1 ó 2)? (Motivación) | Registre # Motivación en Redcap Registre # Confianza en Redcap Registre Barreras en Redcap Registre Facilitadores en Redcap |
| Confianza En una escala del 1 al 10, califique su confianza/seguridad o capacidad para [insertar el nombre de la meta], donde 1 significa que no está del todo seguro y 10 significa que está muy seguro de que puede mantener ese cambio. | |
| ¿Cómo se calificaría? | |
| ¿Qué te hizo elegir ese número y no un número más bajo (como 1 ó 2)? (Facilitadores) | |
| ¿Qué se necesita para llegar a un número más alto (como 8 ó<br>9)? | |
| Si es un 10, ¿qué necesitarías para mantenerte en un 10? | |
| Resumen de la muestra: Siente que está muy motivado para hacer este cambio porque usted (primera parte de la calificación). Usted podría (insertar comentarios de los padres). En términos de poder hacer este cambio, siente que puede hacerlo porque (primera parte de 1 ó 2). Cree que podría aumentar su confianza si (inserte comentarios de la última parte 9 o 10). Parece que está listo y comprometido a hacer este cambio. | |
| *Nota: si los padres tienen dos metas, evalúe motivación v | |

confianza para ambas.



# Plan para la sesión de preparación de comidas

En la próxima visita hablaremos sobre la planificación y preparación de las comidas y las formas de cómo involucrar a su hijo/a. También prepararemos un plato rápido y nutritivo para su familia con su hijo y un estudiante culinario de la Universidad de Johnson and Wales. Aquí hay algunas recetas rápidas y saludables de las cuales podemos elegir.

Aquí hay algunas recetas que podríamos traerle

Muestre la receta para "ensalada de frijoles" and "sopa de lentejas"

¿Qué receta le gustaría probar con su familia?

# 5 minutos



Lista de recetas

Registre Home Food Prep in Redcap

#### Cierre

Vamos a programar nuestra próxima visita.

¿Qué días de la semana y cuáles horas son las mejores para usted?, teniendo en cuenta que prepararemos una comida y que la visita durará entre 60 y 90 minutos.

También tendremos una pasante de la escuela culinaria Johnson and Wales, quien vendrá para ayudarnos a preparar una receta. Ella traerá los alimentos para preparar la receta que usted escogió. Ella vendrá conmigo al inicio de la siguiente sesión, se instalará y prepará todo en el área de la cocina. Después que hablemos y establezcamos las metas, usted, [nombre del niño(a)] y todos nos iremos a la cocina para preparar la receta juntos.

También quiero recordarle que recibirá mensajes de texto con consejos y recetas útiles 2 veces por semana.

¿Puedo confirmar el número para contactarlo/a? Si está interesado/a en obtener más información o desea conectarse con otros padres de niños de 2 a 5 años, también puede consultar nuestro grupo de Facebook.

Gracias por tomarse el tiempo para reunirse conmigo. También, le queremos pedir si por favor puede responder algunas preguntas en el IPAD de las sesión de hoy.

Completar el cuestionario de satisfacción

#### 5 minutos

- Registre **Siguiente Visita** en RedCap y Google Calendar "Home Visit and Phone Call Schedule" "Home Visit and Phone Call Checklist and Satisfaction Questionnaire
- Pida a los participantes que completen el cuestionario de satisfacción



# Visit 2 Script

# Guión de Grabación

(Antes de encender la grabadora)

Hola, es bueno verlo(a) de nuevo. Muchas gracias por reunirse conmigo el dia de hoy. Ella es Haley, va estar con nosotros hoy, está haciendo su internado culinario en Johnson and Wales y nos va estar ayudando a preparar un comida el día de hoy. Quería recordarle que vamos a estar preparando una comida hoy, podríamos poner nuestras cosas en la cocina?

Quería recordarle que voy a grabar la sesión. La grabación se utilizará para asegurarse que cada sesión se realice de la misma manera con cada familia. Como se indica en el formulario de consentimiento, todas las grabaciones se guardarán en un lugar seguro y se destruirán una vez que completamos el estudio. La información de las grabaciones solo se compartirá con el personal del estudio. Si está listo(a), encenderé la grabadora ahora.

#### Introducción

Durante nuestra reunión de hoy, haremos lo siguiente:

- 1. Revisar sus metas de la última visita.
- 2. Hablar sobre cómo preparar y comprar comidas y cómo involucrar a su hijo(a).
- 3. Establecer metas para la próxima visita.
- 4. Preparar una comida juntos.

¿Qué preguntas tiene?

Si tiene alguna pregunta en cualquier momento siéntase libre de pararme y preguntarme.

#### Evaluar

obre

2-5 minutos

2 Minutos

Dígame lo que recuerda de nuestra última conversación sobre maneras saludables de alimentar a su hijo/a

Afirme


#### Reflexione

Gracias por compartir sus experiencias. Es útil saberlo. Suena como.... Resuma

Llevar copias de los folletos de la visita 1 por si fueran solicitados de nuevo.

#### Reevaluar

La última vez que hablamos, usted identificó \_\_\_\_\_ como una meta en la que quería trabajar.

La última vez dijo que esto tenía un X/10 en importancia para usted. ¿Qué tan consistente es eso con la forma en la que se siente actualmente?

La última vez dijo que tenía un X/ 10 en confianza (seguridad en que puede hacer), ¿qué tan consistente es eso con la forma en la que se siente actualmente?

¿Cuáles fueron algunos de los cambios después de nuestra última visita?

¿Cómo funcionó eso para usted y su hijo/a?

¿Qué tan satisfecho está con lo que intentó?

¿Qué le ayudó a probar este nuevo

Insertar estrategia / nombre de meta?

¿Qué se interpuso o lo hizo difícil?

Relacione con valores / metas para las comidas familiares. Si tenía 2 metas, revise ambas y resuma.

Resuma y reflexione

Parece que hay varias cosas que salieron bien. Resuma

También discutió algunas cosas que quiere cambiar. Resuma

#### 10 minutos

Utilizar metas de visita 1, disponible en Redcap bajo la opción Home Visit 1 encounter.



Puntos clave:

Identifique y promueva conversación de cambio.

<u>DESEO:</u> Querer, desear, gustar HABILIDAD: Poder, podria

RAZÓN: Razon especifica para el cambio

NECESIDAD: Necesitar, tener que, deber, importancia, etc. (sin indicar la razón específica)

<u>COMPROMISO:</u> Voluntad, intención de, ir a, etc.

ACTIVACIÓN: Listo para, dispuesto a (sin compromiso específico)

TOMANDO PASOS: Reportar acción específica reciente (paso) hacia el cambio

•Respondiendo a plática de cambio:

<u>Explorar</u>. Pida una explicación: ¿cómo, de qué manera, por qué? Pida ejemplos: cuándo fue la última vez que sucedió esto (por ejemplo, para una consecuencia adversa).

<u>Afirmar</u>. Expresar acuerdo, agradecimiento, ánimo, etc. para el deseo/necesidad de cambio.



Reflexionar. Esta es la respuesta más común sobre la conversación de cambio: ofrecer una reflexión simple o compleja. ("Lo escucho decir que xxx" o "Siente que es difícil xx")

Resumen. Piense en la conversación como un campo de flores: elija las oraciones que desea resaltar, las que se centran en el cambio y preséntalas a la familia en un resumen como en un "ramo". Puedes seleccionar en qué enfocarte en este proceso.

# Compra y Preparación de Comida

Ahora cambiemos un poco de tema y hablemos sobre el tema de esta visita, que es sobre la compra y preparación de las comidas.

Cuénteme un poco acerca de cómo compra su comida.

¿Qué desafíos tiene al comprar o preparar las comidas?

¿Qué funciona bien cuando compra y prepara las comidas?

Si usted está de acuerdo, Haley y yo queremos compartir más información sobre cómo comprar alimentos; también vamos a compartir algunas formas en las que puede incluir a su hijo/a.

#### Revisión de Folleto Segunda Visita

Ir de compras y planificar las comidas puede ser difícil, especialmente con los niños pequeños. ¡El folleto de esta semana contiene consejos para facilitar las compras y ahorrarle tiempo y dinero!

Revisar folleto "Consejos para organizar la compra de comestibles."

Como puede ver, una de las recomendaciones principales es planificar con anticipación, para que sepa lo que necesita para la semana.

#### 15 minutos

Consejos para organizar la compra de comestibles.

Involucra a los niños en el supermercado y mejora la alimentación en el hogar

Identifique y promueva conversación de cambio. Puede ser útil marcar las estrategias que la familia está interesada en probar en el folleto de establecimiento de metas.



Aquí hay un ejemplo de cómo se ven 6 días de meriendas y comidas para una familia de 4 personas. Observe cuánto más baratas son las comidas en comparación a la comida rápida o las tiendas de conveniencia. Además, incluye algunos consejos para involucrar a sus hijos en el mercado y en el hogar.

Sabemos que puede ser un desafío llevar niños pequeños al supermercado, pero acá hay algunas ideas para mantenerlos ocupados e interesados en aprender acerca alimentos. Jugar juegos como "Yo espío" puede mantenerlos ocupados. Si están pidiendo comida, deje que ellos escojan frutas y vegetales. Es más probable que los niños coman los alimentos que ellos escogieron.

Revise el folleto con los padres, luego pregunte lo siguiente

¿Cuál de estas estrategias probó antes?

Afirme. reflexione

¿Qué le gustaría probar?

Afirme, reflexione

¿Qué preocupaciones tiene sobre las recomendaciones?, es decir, ¿posibles desafíos?

Afirme, reflexione

Resolución de problemas / establecimiento de metas:

Ahora me gustaría hablar con usted sobre el establecimiento de una meta para abordar el tema que mencionó que desea cambiar

> Si los padres identificaron varios cambios que le interesaron, haz que clasifiquen los más importantes para ellos, desde el más importante al menos importante para ellos, elija 1-2.

Puede elegir entre las estrategias del folleto o entre las metas propias de los participantes que se alinean con los objetivos de desempeño.

¿Por qué quiere hacer este cambio? (Deseo) (Reflexión)

#### 15 minutos



Folleto con metas

Guía para el establecimiento de metas. Las metas deberían ser:

- 1. Específico: Asegúrese de que las metas estén detalladas. (Quien, que, cuando, donde)
- 2. Medible: Asegúrese de que el participante pueda identificar lo que sucederá cuando logre su meta.



# ¿Cómo podría hacerlo? (Capacidad) (Reflexión) ¿Cuál es una buena razón para hacer el cambio? (Razones) (Reflexión) ¿Qué tan importante es, y por qué? (0-10) (Necesidad) (Registre Número)

específica e identificar barreras.

(Reflexión)

El objetivo de esta sección es desarrollar una meta

Deje la hoja de determinación de metas con el padre y tome una foto.

- 3. Realizable: Las metas deben ser realistas, no ideales.
- 4. Relevante: Las metas deben relacionarse con las mejores prácticas de alimentación y nutrición.
- 5. Limite de Tiempo:La meta debe tener un plazo de tiempo de cuándo se cumplirá (para la próxima visita)

\*Si los padres escogen un comportamiento (por ejemplo, modelar o ejemplificar un comportamiento saludable) y una meta relacionado a un alimento (por ejemplo, disminuir bebidas gaseosas), lo ideal sería combinarlos a una sola meta: "Modele una alimentación saludable al no toma bebidas gaseosas durante la cena"

Objetivos de rendimiento: Como parte del estudio, queremos que los participantes logren lo siguiente:

- Incrementar las comidas familiares.
- Ser un modelo a seguir
- Preparar comidas
- Incluir verduras
- Hablar con los niños sobre los beneficios de los alimentos.
- Involucrar al niño en la preparación de alimentos.

Evaluar la preparación para hacer el cambio

Motivación

Ahora que ha establecido una meta sobre \_ [insertar tema] \_\_\_\_
para su familia, me gustaría saber cómo se siente en este
momento acerca de \_\_\_\_ [insertar nombre de la meta]
\_\_\_\_ En una escala de 1 al 10, donde 1 significa que no
quiere hacer esto y 10 significa que realmente quiere hacer
esto. ¿Cómo se calificaría? (Preparación)

\*15 minutos

Registre Preparación en Redcap

Registre # Motivación en Redcap

Registre # Confianza en redcap



¿Qué le hizo elegir ese número y no un número más bajo (como 1 ó 2)? (Motivación)

Registre **Barreras** en Redcap

Registre **Facilitadores** en Redcap

#### Confianza

En una escala del 1 al 10, califique su confianza o capacidad para [insertar el nombre de la meta]

donde 1 significa que no está del todo seguro y 10 significa que está muy seguro de que puede mantener ese cambio.

¿Cómo se calificaría?

¿Qué te hizo elegir ese número y no un número más bajo (como 1 ó 2)? (Barreras)

¿Qué se necesita para llegar a un número más alto (como 8 o 9)? O, si un 10 ¿Qué haría falta para mantenerte en un 10? (Facilitadores)

Resumen de la muestra

Siente que está muy motivado para hacer este cambio porque su (primera parte de la calificación). Usted podría (insertar comentarios de los padres).

En términos de poder hacer este cambio, siente que puede hacerlo porque (primera parte de 1 ó 2).

**Cree que podría aumentar su confianza si** (inserte comentarios de la última parte 9 ó 10).

Parece que está listo y comprometido a hacer este cambio.

Deje la hoja de establecimiento de metas con el padre y tome foto.

Cuando nos reunamos la próxima vez, revisaremos esta meta, entonces por favor mantenga esta hoja con sus materiales.

Sesión de Preparación de Comida

Ahora haremos algo diferente. Vamos a hacer una comida juntos. Nuestro objetivo es involucrar a su hijo(a) en esta sesión. Puede ser útil tener todos los alimentos, equipo u otros materiales listos previamente. Ahora veamos si puedo ayudarle a involucrar a [nombre de niño(a)].

Invite al niño(a) a que participe y ayude a preparar la receta.

# 30 minutos

Registrar Prepared Meal



\*\*\*Community Health Worker can translate this section\*\*\*

Note: Translate for Haley as she does activity.

Haley: So today, we are going to be preparing X recipe today.

We want to involve [child's name] today and thought he could help today with [enter name of task]. Would that be ok with you?

Begin preparing the recipe together. Take note: you can assess if the parent would like more instruction in preparing the meal or if they already know how to cut allow them to help and you can help with the child involvement.

Walk through the steps as you prepare the meal and share any tips that may be helpful to the parent.

Some important tips to share:

- 1) Washing hands- both parent and child-very important before cooking anything
- 2) Setting up all ingredients and prepping BEFORE putting recipe together can save time
- 3) Putting ingredients away and cleaning up as you can go can make clean up easier
- 4) How to cut the onion
- 5) Rolling the lemon/lime before squeezing
- 6) How to safely cut an avocado

Clean up while CHW wraps up with the parent.

Libro de Recetas (recetas y folleto de Preparación de comidas para niños)



Puntos Claves para consejera:

- Ayudar a los padres a involucrar al niño(a)
- Traducir la conversación entre Haley y los padres y/o niño(a)
- Identificar y promover el cambio durante la sesión de cocina.

Cierre

Repaso de la Sesión de Comida

¿Cómo cree que tener a [nombre del niño (a)] involucrado en el proceso de preparación de la comida funcionó?

¿Qué le gustó sobre eso?

¿Qué es lo que no le gustó de eso?

2 minutos



¿Cuáles podrían ser algunas formas en que podría hacer esto regularmente?

#### Resumen de la visita

En la próxima visita, revisaremos otro video de un tiempo de comida y discutiremos las rutinas y los límites que ayudan a los niños a comer de manera más saludable. ¿Recuerda cómo subir un video con su teléfono? ¿Podría enviarnos otro video a lo largo de estas 2 próximas semanas?

Programemos nuestra próxima visita para una semana después de eso. ¿Qué días de la semana y horas del día funcionan mejor para usted, teniendo en cuenta que la sesión tardará 60 minutos?

Además, recuerde que recibirá mensajes de texto con consejos y recetas útiles 2 veces por semana. ¿Puedo confirmar el número para contactarlo(a)? Si está interesado(a) en obtener más información o desea conectarse con otros padres de niños de 2 a 5 años, también puede consultar nuestro grupo de Facebook.

Gracias por tomarse el tiempo para reunirse conmigo.

5 minutos

Registre **Siguiente Visita** en RedCap y Google Calendar "Home Visit and Phone Call Schedule" "Home Visit and Phone Call Checklist and Satisfaction Questionnaire



# Guión de grabación

(Antes de encender la grabadora)

Hola, es bueno verlo(a) de nuevo. Quería recordarle que voy a grabar la sesión. La grabación se utilizará para asegurarse que cada sesión se desarrolle de la misma manera con cada familia. Como se indica en el formulario de consentimiento, todas las grabaciones se guardarán en un lugar seguro y se destruirán una vez completemos el estudio. La información de las grabaciones solo se compartirá con el personal del estudio. Si está listo(a), encenderé la grabadora ahora.

#### Introducción

Durante nuestra reunión de hoy, vamos a

- 1. Revisar sus metas y la experiencia de la última visita
- 2. Revisar tu video de la hora de comida
- 3. Hablar un poco sobre cómo las rutinas y los límites pueden ayudar a los niños a comer de manera más saludable
- 4. Discutir si le gustaría hacer algún cambio en la forma en que alimenta a su hijo(a).

¿Qué preguntas tiene?

Si tiene preguntas a medida que avanzamos siéntase libre de parar y preguntarme.

#### -valuar

Cuénteme lo que recuerde de nuestra última visita sobre la preparación de comidas, las compras y la participación de su hijo.

Afirme, reflexione
Gracias por compartir tus experiencias. Es útil saberlo.
Suena como... resuma

2-5 Minutos

2 Minutos

Llevar copias de los folletos de la visita 1 por si fueran solicitados de nuevo.

Reevaluar 10 Minutos



La última vez que hablamos, identificó \_\_\_\_ como una meta en la que quería trabajar.

La última vez dijo que esto era "X" de importante para usted. ¿Qué tan consistente es eso con la forma en la que se siente actualmente?

La última vez que dijo que estaba en un nivel de confianza "X" para alcanzar esta meta. ¿Qué tan consistente es eso con la forma en la que se siente actualmente?

¿Cuáles fueron algunas de las estrategias que probó o los cambios que realizó en / después de nuestra última visita?

¿Cómo funcionó eso para usted y su hijo/a?

¿Qué tan satisfecho está con el cambio que intentó?

¿Qué le ayudó a probar el nuevo

(inserte estrategia / nombre de meta)?

¿Qué se interpuso o lo hizo difícil?

Relacione con valores / metas para las comidas familiares.

#### Resuma y Reflexione

Parece que hay varias cosas que salieron bien. También mencionó algunas cosas que desea cambiar / áreas para mejorar. Utilizar metas de visita 1, disponible en Redcap bajo la opción Home Visit 1 encounter.



Puntos clave:

Identifique y promueva conversación de cambio.

<u>DESEO:</u> Querer, deseo, gusto
<u>HABILIDAD:</u> puede, podría, apto
<u>RAZÓN:</u> Motivo específico del cambio.
<u>NECESIDAD:</u> Necesito, tengo que, debo, importante, etc. (sin indicar razón específica)

<u>COMPROMISO:</u> Voluntad, intención, ir a, etc

ACTIVACIÓN: Listo para, dispuesto a (sin compromiso específico).

TOMANDO PASOS: Reporta acción específica reciente (paso) hacia el cambio

•Respondiendo a plática de cambio:

<u>Explora.</u> Pida una explicación: ¿cómo, de qué manera, por qué? Pida ejemplos: cuándo fue la última vez que sucedió esto (por ejemplo, para una consecuencia adversa).

<u>Afirma.</u> Expresa acuerdo, agradecimiento, ánimo, etc. for el deseo/necesidad/etc de cambiar.

<u>Reflexiona.</u> Esta es la respuesta más común para cambiar la conversación, para ofrecer una reflexión simple o compleja. ("Te escucho decir que xxx o que es difícil xxx").

Resumen. Piense en la conversación como un campo de flores: elija las oraciones que desea resaltar, las que se centran en el cambio y preséntalas a la familia en un resumen como en un



'ramo". Puedes seleccionar en qué enfocarte en este proceso. Revisión de Video 15 minutos Ahora tomemos unos minutos para ver dos clips que fueron elegidos del video de su comida familiar. Haremos pausas entre cada corto/clip y discutiremos acerca de lo que usted piensa sobre el corto/clip. Recuerde, sólo usted sabe lo que es mejor Use la hoja con retroalimentación para su familia. Estoy aquí para hablar sobre sus pensamientos y experiencias al alimentar a su hijo(a). Reproduzca el corto/clip 1 (Practicas Positivas). Haga una pausa cuando la pantalla diga corto/clip 2, explore y provea Cortos del video de comida retroalimentación. familiar en el I-PAD ¿Qué sobresale del video? Obtenga las ideas y opiniones sobre el proceso de filmación Puntos clave (filmar una comida familiar y mandarla a los investigadores). Identificar y provocar el cambio en la Explora: \*si el padre ya brindó esta información, no necesita conversación. preguntar otra vez. ¿Qué le sorprendió? Por qué? ¿Qué hizo para intentar que su hijo(a) comiera alimentos saludables? ¿Qué funcionó bien? ¿Qué es lo que, si hay algo, querrá hacer de manera diferente en el futuro? Si le parece bien, me gustaría compartir algunas ideas sobre la comida. Espere la afirmación, luego comparta retroalimentación sobre las prácticas de comidas positivas. ¿Qué piensas de estas ideas? Ahora, observemos el segundo clip.

Reproduzca el segundo clip del video.



# ¿Qué sobresale del video?

Obtenga las ideas y opiniones sobre el proceso de filmación (filmar una comida familiar y mandarla a los investigadores).

Explora: \*si el padre ya brindó esta información, no necesita preguntar otra vez.

# ¿Qué le sorprendió? Por qué?

¿Qué hizo para intentar que su hijo/a comiera alimentos saludables?

¿Qué funcionó bien?

¿Qué es lo que, si hay algo, querrá hacer de manera diferente en el futuro?

Si le parece bien, me gustaría compartir algunas ideas sobre la comida.

Espere la afirmación, luego comparta retroalimentación sobre las prácticas de comidas positivas.

# Resumen de la sesión de retroalimentación.

Parece que hay varias cosas que está haciendo bien y ... También discutimos algunas áreas con espacio para mejorar y siente que esta información es ...

Gracias por enviar este video. Fue una gran discusión. También tengo algunos materiales impresos en los que podría estar interesado.



# Rutinas y Límites

Los temas para los materiales de esta semana son: rutinas y límites.

Cuénteme un poco sobre la rutina de comidas / bocadillos de tu familia?

¿Qué retos tiene para llevar a cabo una rutina?

¿Qué le ayuda a mantener a su hijo(a) en una rutina?

¿Qué límites o reglas tiene sobre la comida o las comidas en su casa?

¿Cómo funcionan esos límites o reglas para su familia?

Si está de acuerdo, me gustaría compartir información sobre cómo las rutinas y los límites pueden ayudar a los niños a aprender y convertirse en niños que comen saludable.

# Repasar folleto de visita 3

Las rutinas y los límites pueden ser difíciles de establecer, pero pueden facilitar mucho las cosas para usted y su hijo(a) a largo plazo. El folleto de esta visita contiene consejos para crear rutinas y establecer límites alrededor de los horarios de comidas y refrigerios.

Revise el folleto "Estructura para Familias Fuertes- consejos para planificar una rutina" con los padres.

Escuchamos de muchas familias que hacer que los niños vayan a la mesa a comer o que no "piquen" y merienden todo el tiempo puede ser realmente un desafío. Una cosa que puede ayudar es tener una rutina. Este es un esquema o bosquejo de tu tiempo que ayuda a que a usted y su hijo sepan lo que va pasar a lo largo del día. Los niños pueden resistirse a las

Estructura para Familias Fuertes-consejos para planificar una rutina

Identifique y promueva conversación de cambio. Puede ser útil marcar las estrategias que la familia está interesada en probar en el folleto con el establecimiento de metas.

Consejo para manejo del tiempo: Las reflexiones y la exploración de los pensamientos y opiniones de los padres sobre el contenido están en el guión - si el tiempo es limitado, está bien



rutinas al inicio, pero a menudo las disfrutan; si van a la escuela ellos tendrán que acostumbrarse a las rutinas.

proporcionar solamente una breve explicación del folleto.

Cada familia es diferente, al igual que sus rutinas. Algunas sugerencias en el folleto son establecer horarios definidos para las comidas y las meriendas, tener rutinas divertidas que sus hijos esperen, cómo hacer caminatas después de la cena o paseos al parque.

También sabemos que puede ser difícil para los niños pequeños pasar de una actividad a otra, las rutinas pueden ayudar con esto. Por ejemplo, en lugar de pasar directamente de jugar a cenar, se puede incluir una rutina como la siguiente: apagar la TV, limpiar, lavarse las manos y ayudar a poner la mesa para hacer saber a los niños que se acerca la hora de la comida.

¿Qué estrategias ha probado antes?

Afirma, reflexiona

¿Qué sugerencias del follleto esta interesado o le gustaría probar?

Afirma, reflexiona

¿Qué preocupaciones tiene sobre las recomendaciones?

Afirma, reflexiona

Revisa el folleto "Estructura para familias fuertes - reglas y límites" con los padres

Otra forma de crear estructura alrededor de las comidas y las meriendas es tener algunas reglas familiares. Esta es una declaración clara acerca del comportamiento que espera de su hijo. Esto les puede enseñar cuáles comportamientos están bien y cuáles no están bien. Algunos ejemplos de reglas son: las pantallas deben estar apagadas a la hora de comer, todos comen juntos, o todos ayudan a limpiar. Cuando establezca las reglas es importante: explicarle a sus hijos qué es lo que espera de ellos, que usted también siga la regla y que les recuerde las reglas frecuentemente. Los niños rompen las reglas y ponen a prueba los límites frecuentemente, esto es



normal. No se preocupe, si es consiste con las reglas y les recuerda frecuentemente, ellos aprenderán. Aquí hay un espacio en donde puede escribir cuáles reglas a la hora de comer son importantes para su familia.

Muestre la caricatura en la parte posterior del folleto.

Aquí hay un ejemplo de cómo una regla a la hora de comer puede ayudar a los niños.

¿Qué estrategias ha probado antes?

Afirma, reflexiona

¿Qué sugerencias del follleto esta interesado o le gustaría probar?

Afirma, reflexiona

¿Qué preocupaciones tiene sobre las recomendaciones?

Afirma, reflexiona

Resolución de Problemas / Establecimiento de Metas

Pensando en lo que hablamos hoy, incluyendo rutinas, reglas y límites, ¿le gustaría establecer una meta?

Si los identificaron muchos varios que le interesaron, haz que metas clasifiquen los más importantes para ellos, desde el más importante al menos importante para ellos, elija 1-2)

Puede elegir entre las estrategias del folleto o entre las metas propias de los participantes que se alinean con los objetivos de desempeño.

Recuerde que deben escoger al menos 1 meta, pero si tienen más de uno, pueden trabajar en 2 metas.

¿Por qué quiere hacer este cambio? (Deseo) (Reflexión)

¿Cómo podría hacerlo? (Capacidad) (Reflexión)

15 Minutos

Use la hoja de establecimiento de

Guía para el establecimiento de metas. Las metas deberían ser:

1. Específico: Asegúrese de que las metas estén detallados. (Quien, que, cuando, donde)

2. Medible: Asegúrese de que el participante pueda identificar lo que sucederá cuando logre su meta.

3. Realizable: Las metas deben ser realistas, no ideales.



| ¿Cuál es una buena razón para hacer el cambio? (Razones) | 4. Relevante: Las metas deben |
|---|---|
| (Reflexión) | relacionarse con las mejores prácticas |
| | de alimentación y nutrición. |
| ¿Qué tan importante es, y por qué? (0-10) (Necesidad) (Anota el | 5. Limite de Tiempo:La meta debe tener |
| número) | un plazo de tiempo de cuándo se |
| (Reflexión) | cumplirá (para la próxima visita/llamada) |
| ¿Qué es lo que va a hacer? (Compromiso) | |
| (Reflexión) | |
| (1.10.110.11) | <u> </u> |
| ¿Qué está listo y dispuesto a hacer? (Activación) | Objetivos de Rendimiento: como |
| (Reflexión) | parte del estudio queremos que los |
| | participantes logren lo siguiente: |
| ¿Qué has hecho ya? (Tomando pasos) | Determinar cuándo y dónde |
| (Reflexión) | comen los niños. |
| | <ul> <li>Proporcionar opciones limitadas</li> </ul> |
| Registre la meta específica de la parte inferior de la hoja de | guiadas al niño/a |
| establecimiento de metas en la hoja de datos. El objetivo de | Enseñar sobre comidas |
| esta sección es desarrollar una meta específica e identificar | saludables a los niños |
| barreras. | <ul> <li>Limitar las pantallas en las</li> </ul> |
| | comidas |
| Deje la hoja de establecimiento de metas con el padre y | <ul> <li>Proporcionar un refuerzo positivo</li> </ul> |
| tome una foto. | cuando comen alimentos |
| Por lo tanto, su meta es: (insertar la meta de la última línea en la | saludables |
| hoja de establecimiento de metas). | |
| noja ao ostablosimismo ao metasji | Anote <b>Meta</b> en Redcap |
| Cuando lo llame el siguiente mes, revisaremos esta meta, así | Suba una foto de la hoja de metas (si |
| | más de una, suba ambas) |
| puerta del refrigerador. | |
| Evaluar la Preparación Para Hacer el Cambio | 15 Minutos |
| | Anote la Preparación en Redcap |
| Motivación | Anote la Preparación en Redeap |
| Ahora que ha establecido una meta sobre _ [insertar tema] | |
| para su familia, me gustaría saber cómo se siente en este<br>momento acerca de [insertar el nombre de la meta] | Anote el # Motivación en Redcap |
| Inomento acerca de [insertar el nombre de la meta] | |
| En una escala de 1 a 10, donde 1 significa que no quiere hacer | Anote el # Confianza en Redcap |
| esto y 10 significa que realmente quiere hacer esto. ¿Cómo te | , wiete ein Germania en reedeap |
| calificarías? (Preparación) | |
| ( | Anota las <b>barreras</b> en Redcap |
| ¿Qué te hizo elegir ese número y no un número más bajo (como | _ |
| 1 ó 2)? (Motivación) | Anote a los facilitadores en Redcap |
| | · |
| Confianza | |



| En una escala del 1 al 10, califique su confianza/seguridad o capacidad para[insertar el nombre de la meta], donde 1 significa que no está del todo seguro y 10 significa que está muy seguro de que puede mantener ese cambio. | |
|---|---|
| ¿Cómo te calificarías? | |
| ¿Qué te hizo elegir ese número y no un número más bajo (como 1 ó 2)? (Barreras) | |
| ¿Qué necesita para llegar a un número más alto (como 8 ó 9)?<br>Si un 10 ¿Qué haría falta para mantenerte en un 10?<br>(Facilitadores) | |
| Resumen de la muestra | |
| Sientes que estás muy motivado para hacer este cambio porque tú (primera parte de la calificación). | |
| Usted podría (insertar comentarios de los padres). | |
| En términos de poder hacer este cambio, siente que puede hacerlo porque (primera parte de 1 ó 2). | |
| Usted cree que podría aumentar su confianza si (inserte comentarios de la última parte 9 ó 10). | |
| Piensas que (barrera) puede hacer que sea desafiante pero (solución) fue identificado como algo que podría ayudar. | |
| <u>Cierre</u> | 5 Minutos |
| Ha sido un placer conocer y reunirme con usted y su familia.<br>Estaré en contacto por teléfono durante los próximos 3 meses<br>para verificar las metas, resolver problemas y animarlo. | Registre <b>Siguiente visita</b> en RedCap<br>y Google Calendar |
| ¿Qué días de la semana y horas del día está disponible para recibir llamadas? ¿Puedo confirmar el mejor número para comunicarme con usted? | |
| Solo para recordarle que continuará recibiendo mensajes con consejos y recetas útiles 2 veces por semana. Si está interesado en obtener más información o desea conectarse con otros padres de niños de 2 a 5 años, también puede consultar nuestro grupo de Facebook. | |



| Como la ultima visita, si por favor podria responder estas |
|-----------------------------------------------------------------|
| preguntas en el IPAD.<br>Llenar el cuestionario de satisfacción |
| Gracias por tomarse el tiempo para reunirse conmigo. |



# Phone Call Script

| Guión de grabación | | 5 minutos |
|---|---|---|
| (Antes de encender la grabadora) | | |
| Universidad de Rhode Island. Lo/<br>telefónica del mes. Gracias por su ti<br>que estaremos grabando esta sesi<br>grabadora ahora. Le enviamos unos | mi nombre es<br>Fuertes Comienzan en Casa de la<br>la llamo para hacer nuestra sesión<br>empo el dia de hoy. Quería recordarle<br>ón. Si está listo/a voy a encender la<br>s materiales por correo, si los tiene a<br>s durante la llamada. También vamos | Hoja de metas en<br>Redcap en el anterior<br>Home Visit Encounter. |
| <u>Introducción</u> | | Puntos clave:<br>Reafirme la meta y<br>chequee motivación y |
| Para comenzar, quería saber Respuesta: Sí/No | | confianza. |
| ¿Pudo leer la hoja de información?<br>Respuesta: Sí / No | | Registre si leyó folleto de información y textos, y |
| ¿Tiene alguna pregunta acerca de e | sa información? | si le parecieron útiles. |
| ¿Qué tan útil le fue esta hoja de info<br>algo útil, un poco útil, o para nada ú | | |



Haga que seleccione una de las opciones de respuesta y registre la respuesta en Redcap

Registre en Redcap si se cumplió su meta: seleccione Sí/ No

# ¿Recibió los mensajes de texto?

Respuesta: Sí / No

# Leyó los mensajes de texto? Si no, por qué no?

Respuesta: Sí / No Si sí, pregunte:

# ¿Qué tan útiles fueron los mensajes de texto? Diría que fueron: muy útiles, algo útiles, un poco útiles, o para nada útiles?

Haga que seleccione una de las opciones de respuesta y registre la respuesta en Redcap.

# ¿Tuvo algún problema o pregunta?

Proporcione un resumen de la meta de la que se habló en la última visita.

<u>Ejemplo:</u> "La última que que hablamos, usted mencionó que quería preparar más comidas con su hijo(a). Usted pensaba que esto haría que "nombre del niño(a)" se emocionara mas al probar nuevos vegetales. Su meta era preparar las comidas junto con su hijo(a) dos veces por semana. También dijo que estaba algo motivado(a) por hacer este cambio (calificado con un 7) pero no se sentía tan seguro que podría hacerlo cada semana (calificado con un 3). ¿Cómo le fue con esta meta?

En una escala del 1 al 10, ¿cuál diría que es su nivel de motivación ahora al preparar las comidas junto a su hijo(a)? ¿Cuál diría que es su nivel de confianza/seguridad ahora?

Reflexione **o** haga una pregunta abierta para entender mejor cómo el participante está trabajando para alcanzar su meta:

Si el participante tuvo problemas con la meta:

¿Qué cree que podría hacer de manera diferente la próxima vez?"

#### Cerrar el tema

Proporcione un resumen del progreso y haga una transición a la próximo meta

Ejemplo:Parece que pudo alcanzar su meta en este tema y está satisfecho con su progreso.

¿Cómo se siente acerca del material que recibió en su correo?



# Revise Tema Nuevo

Nosotros le enviamos información sobre (insertar nombre del folleto).

Este le explica algunos de los temas de los que hablamos durante nuestras sesiones, incluyendo (insertar temas del folleto).

¿Cómo se siente al establecer una meta para este tema?

Objetivos de rendimiento: como parte del estudio, queremos que los participantes cumplan lo siguiente:

- Incrementar frutas y verduras, granos integrales, proteínas magras servidas.
- Aumentar la accesibilidad de frutas y verduras.
- Disminuir la accesibilidad de los alimentos procesados y golosinas
- Ofrecer opciones saludables.
- Aumentar las comidas familiares / modelando los roles
- Tener un lugar fijo donde la familia come, como la mesa o el mostrador.
- Limitar las distracciones como televisión, tableta o computadora
- Servir porciones pequeñas y dejar que el/la niño/a decida cuándo esté lleno/a
- Incrementar las comidas familiares.
- Ser un modelo a seguir
- Preparar comidas
- Incluir verduras
- Hablar con los niños sobre los beneficios de los alimentos.
- Involucrar al niño en la preparación de alimentos.
- Determinar cuándo y dónde comen los niños.

#### 2 minutos



Folleto mes 4 Folleto mes 5 Folleto mes 6



Identifique y promueva conversación de cambio. Puede ser útil marcar las estrategias que la familia está interesada en probar en el folleto que incluye el establecimiento de metas.



- Proporcionar opciones limitadas y guiadas al niño/a
- Enseñar sobre comidas saludables a los niños
- Limitar las pantallas en las comidas
- Proporcionar un refuerzo positivo cuando comen alimentos saludables

# Resolución de Problemas/ Establecimiento de Metas

Ahora me gustaría hablarle acerca de establecer una meta para abordar el nuevo/siguiente tema que seleccionó (repita el tema y el meta aquí).

¿Por qué quiere hacer este cambio? (Deseo) (Reflexión)

¿Cómo podría hacerlo? (Capacidad) (Reflexión)

¿Cuál es una buena razón para hacer este cambio? (Razones) (Reflexión)

¿Qué tan importante es, y por qué? (0-10) (Necesidad) (Registre Número) (Reflexión)

¿Que intentará hacer? (Compromiso) (Reflexión)

¿Qué está listo o dispuesto a hacer? (Activación) (Reflexión)

¿Qué ha hecho ya? (Pasos tomados) (Reflexión)

Registre la meta específica en la parte inferior de la hoja de establecimiento de metas. Registre esta meta específica en Redcap. El objetivo de esta sección es desarrollar una meta específica e identificar los obstáculos.

#### 15 minutes



Hoja de metas



Puntos clave:

Guía para el establecimiento de metas. Las metas deberían ser:

- Específico: Asegúrese de que las metas estén detallados. (Quien, que, cuando, donde)
- 2. Estimable: Asegúrese de que el participante pueda identificar lo que sucederá cuando logre su meta.
- 3. <u>Realizable:</u> Las metas deben ser realistas, no ideales.
- 4. <u>Relevante</u>: Las metas deben relacionarse con las mejores prácticas de alimentación y nutrición.
- 5. <u>Limite de Tiempo</u>: La meta debe tener un plazo de tiempo de cuándo se



| Entonces, su meta es: (Insertar meta de la última línea de la hoja de establecimiento de metas). | cumplirá (para la próxima<br>visita/llamada) |
|---|---|
| Evaluando Obstáculos | Objetivos de |
| ¿Qué podría interponerse en su camino para cumplir su meta (replantear meta)? | Rendimiento: como parte del estudio queremos que |
| Cuando volvamos a hablar por teléfono, revisaremos esta meta, así que guarde esta hoja con sus materiales. | los participantes logren lo siguiente: Determinar cuándo y dónde comen los niños. Proporcionar opciones limitadas y guiadas al niño/a Enseñar sobre comidas saludables a los niños Limitar las pantallas en las comidas Proporcionar un refuerzo positivo cuando comen alimentos saludables |
| | Suba una foto de la hoja<br>de metas (si más de una,<br>suba ambas) |
| Evaluar la Preparación para hacer el Cambio | 15 minutos |
| Motivación Ahora que ya ha establecido la meta acerca de[insertar tema], me gustaría saber como se siente acerca de[insertar nombre de la meta] En una escala del 1 al 10, en donde 1 significa que no quiere hacer esto y 10 significa que realmente quiere hacer esto. | Registre <b>Preparación</b> en Redcap Registre <b># Motivación</b> en Redcap |
| ¿Cómo se calificaría? | Registre <b># Confianza</b><br>en Redcap |
| ¿Qué le hizo elegir ese número y no un número más bajo (como 1 ó 2)? | |



| ¿Qué necesitaría para llegar a un número más alto (como 8 ó 9)? Si un<br>10, ¿qué necesitaría para mantenerse en un 10? | Registre <b>Barreras</b> en Redcap |
|---|---|
| Confianza | Registre <b>Facilitadores</b> en Redcap |
| En una escala del 1-10, califique su confianza o habilidad para, en donde 1 significa que no se siente seguro de sí mismo y 10 significa que está muy seguro de que podrá mantener el cambio. | |
| ¿Cómo se calificaría? | |
| ¿Qué le hizo elegir ese número y no un número más bajo (como 1 ó 2)? | |
| ¿Qué necesitaría para llegar a un número más alto (como 8 ó 9)? Si un 10, ¿Qué se necesitaría para mantenerse en un 10? | |
| Resumen de Ejemplo: Sientes que estás muy motivado para hacer este cambio porque tú (primera parte de la calificación). Usted podría (insertar comentarios del cuidador). En términos de poder hacer este cambio, siente que puede hacerlo porque (primera parte de 1 ó 2). Cree que podría aumentar su confianza si (inserte comentarios de la última parte 9 ó 10). Parece que está listo para hacer este cambio y está comprometido a hacer este cambio. | |
| <u>Cierre</u> | 2 minutos |
| Usted recibirá un folleto en el correo en 1-2 semanas. Usted también<br>seguirá recibiendo mensajes de texto. También puede revisar nuestra<br>página de facebook para consejos, recetas, y para comunicarse con<br>otros padres. | Registre <b>Siguiente</b><br><b>Visita</b> en Redcap y Google<br>Calendar |
| maniale de nuevo para levisar la meia y discum sobre el broximo lema | *Nota para calendario de la<br>próxima llamada telefónica,<br>según el equipo de<br>recolección de datos |
| ¿Cuál sería el mejor día y hora para nuestra próxima<br>llamada? (Anote la fecha de la llamada)<br>Mejor número de teléfono: | |



| Gracias por tomarse el tiempo para reunirse conmigo. Me estaré<br>comunicando pronto con usted por teléfono. |
|---|

# **Text Messages**

| Message Delivery Scheduled | Message Content Spanish |
|---|---|
| Week 1 - Welcome | **** Bienvenidos **** |
| Week 1 - Message 1 | Los alimentos saben mejor cuando tenemos hambre! Si tus hijos llegan a casa con mucha hambre de la escuela, sírveles rodajas de vegetales y frutas. |
| Week 1 - Wiessage 1 | Les granes integrales can harates y muy putritives! Mire este enlace |
| | Los granos integrales son baratos y muy nutritivos! Mira este enlace sobre diferentes formas en las que puedes incorporar granos enteros en cada tiempo de comida. |
| Mark 1 Marrage 2 | https://wholegrainscouncil.org/resources/recursos-en- |
| Week 1 - Message 2 | espa%C3%B1ol/granos-enteros-todos-los-d%C3%ADas |
| Week 2 - Message 1 | ¿Sabías que los frijoles, guisantes/chícharos y las nueces son una<br>buena fuente de proteína? Agrégalos a platillos como tacos, pastas<br>y sopas para que sean más nutritivos. |



| | Los padres y madres ofrecen y los hijos deciden! Si estás ofreciendo |
|---|---|
| Week 2 - Message 2 | comidas y meriendas saludables a tu hijo, estás cumpliendo con tu tarea! Es decisión de ellos comérselos o no. |
| Week 3 - Message 1 | Criar niños con hábitos saludables no es fácil, pero vale la pena. ¡Estás haciendo un excelente trabajo! |
| Week 3 - Message 2 | Las sopas son una excelente manera de usar los sobrantes de vegetales Prueba esta receta, los niños pueden ayudar a colar los frijoles. <a href="https://youtu.be/kW6JV4DsTFc">https://youtu.be/kW6JV4DsTFc</a> |
| Week 4 - Message 1 | Recuerda que tú decides cuándo, dónde y qué come tu hijo, pero es decisión de ellos si lo comen o no. Es normal que el apetito cambie mucho - no te preocupes si no comen mucho durante una de las comidas. |
| Week 4 - Message 2 | ¿Sabías que los frijoles, guisantes/chícharos y las nueces son una<br>buena fuente de proteína? Agrégalos a platillos como tacos, pastas<br>y sopas para que sean más nutritivos. |
| Week 5 - Message 1 | ¡Tus hijos te imitan! Sé un buen ejemplo para tus hijos y come frutas y verduras todos los días. |
| Week 5 - Message 2 | https://youtu.be/RaLEPfuojWg Prueba esta deliciosa ensalada con<br>tus hijos esta semana. Los niños pueden rasgar la lechuga, exprimir<br>los limones y mezclar los ingredientes. |
| Week 6 - Message 1 | Intenta planear entre 2-3 cenas para esta semana. Pídele a tus niños que escojan una verduras para acompañar el plato |
| Week 6 - Message 2 | ¿Estás preocupado porque tu hijo no te cree cuando le dices que las frutas y vegetales son geniales? Tal vez debería escuchar a otros niños. Mira este video de niños en RI hablando sobre sus alimentos saludables favoritos. <a href="https://www.youtube.com/watch?v=m4u0pjjaSik">https://www.youtube.com/watch?v=m4u0pjjaSik</a> |
| Week 7 - Message 1 | Preparar alimentos de maneras distintas puede cambiar totalmente<br>su sabor! Entre todos en la familia, escojan un vegetal y pruébenlo<br>crudo, asado, a la parrilla, al vapor o salteado! No tengas miedo de<br>agregar tus condimentos o aderezos favoritos! |
| Week 7 - Message 2 | Servir vegetales nuevos con alimentos que ya le gustan a los niños es una manera en la que pueden probarlos y disfrutarlos! Mira esta receta que combina pasta, queso y brócoli! |



| | https://www.h-/DUCCTV/-UDI |
|---|---|
| | https://youtu.be/BIj66TVrHPI |
| | ¿Sabías que los niños necesitan probar una comida por lo menos 8 |
| | veces antes que sepan si les gusta o no? Incluso los pequeños bocados ayudan a que las papilas gustativas se acostumbren a los |
| Week 8 - Message 1 | nuevos alimentos |
| | Los niños comen todo lo que sea fácil de obtener. Ten listo naranjas |
| | peladas o tiritas de pimientos en el refrigerador para hacer que la |
| Week 8 - Message 2 | merienda después de la escuela sea fácil y saludable. |
| | Las listas de compras nos ayudan a estar preparados y a ahorrar |
| | dinero! Usa lápiz y papel, tu celular o una aplicación como Yummly o |
| Week 9 - Message 1 | OutOfMilk. Muchos supermercados tienen sus propias apps o páginas web! |
| | ¡Revisa nuestro sitio en Facebook para ver lo que están haciendo |
| Week 9- Message 2 | otras familias para mantenerse saludables! |
| | ¿Tu hijo pide constantemente golosinas como chips, galletas o |
| | gaseosas? La mejor manera de enseñarles cómo limitar estas |
| Week 10- Message 1 | comidas es mantenerlas fuera de tu casa. |
| | Los niños que comen en familia, se desempeñan mejor en la |
| Week 10- Message 2 | escuela, tienen una mejor autoestima y un menor riesgo de sufrir depresión. |
| Week 10- Wessage 2 | <u>'</u> |
| Week 11- Message 1 | ¡Las comidas en familia no tienen que ser lujosas! Lo importante es que coman juntos. |
| | ¡Los niños se distraen fácilmente! Apagar el televisor o la tableta |
| Week 11- Message 2 | puede ayudarles a concentrarse. |
| | Evita los sobornos y las recompensas por comer. Aunque podría ser |
| | tentador ofrecer una galleta si tu hijo come 3 bocados de espinaca, |
| Mook 12 B4 4 | esto hace que los niños piensen que las golosinas son más |
| Week 12- Message 1 | importantes que las comidas a la hora de comer. |
| Week 12- Message 2 | No hay padres perfectos, y no hay hijos perfectos, pero hay muchos momentos perfectos en el caminoDave Willis |
| WCCK 12- WICSSASC Z | ¡Prepárate! ¡Los niños no siempre siguen las reglas! ¡Muéstrales lo |
| Week 13- Message 1 | que quieres que hagan y recuérdales a menudo! |
| | 1 - |



| | ¡Es difícil sentarse a la mesa a cenar todas las noches! ¡Mira |
|---|---|
| | nuestro libro de recetas para cenas que puedes preparar en menos |
| Week 13- Message 2 | de 30 minutos! |
| | Piensa más allá de una sola comida. Ten en cuenta lo que tu hijo |
| Week 14- Message 1 | come a lo largo de la semana. |
| | Sirve alimentos nuevos con alimentos que ya le gusten a tu hijo ¡Si |
| Week 14- Message 2 | la verdura favorita de su hijo es el maíz, esta receta podría gustarles! https://www.youtube.com/watch?v=Hy-I7MweYCc |
| | Darle opciones a tu hijo y permitir que decida cuánto comer, le |
| Week 15- Message 1 | ayudará a convertirse en un niño saludable y aventurero. |
| | Incluir alimentos nuevos toma tiempo. Ofrece nuevos alimentos con |
| | alimentos que ya le gustan a tu hijo(a) para que puedan llenar sus |
| Week 15- Message 2 | barrigas y explorar alimentos nuevos a su propio ritmo |
| Magle 10 B4 1 | La paciencia funciona mejor que la presión cuando se trata de |
| Week 16- Message 1 | alimentar a los niños pequeños. |
| Week 16- Message 2 | Cocinen juntos. Coman juntos. Hablen juntos. Haz que la hora de comer sea un tiempo familiar |
| Treek Is message I | Ellos aprenden observándote. Come frutas y verduras y sus hijos |
| Week 17- Message 1 | también lo harán. |
| | Llévalas contigo. Enséñale a tu hijo(a) que la fruta entera es una |
| | gran merienda para comer en el parque o en el centro comercial.<br>Pon manzanas, naranjas o bananas en tu bolso para una merienda |
| Week 17- Message 2 | rápida. |
| - | Fortalece la independencia de tu hijo(a) a la hora de la comida. |
| Week 18- Message 1 | Permite que elijan entre los alimentos saludables que le ofreces. |
| | Ofrece a los niños pequeños la misma comida saludable que al |
| Week 10 B4 3 | resto de tu familia. Puede que a tu hijo(a) no le guste todo lo que le |
| Week 18- Message 2 | ofreces pero eso es normal. |
| | Es normal que los niños entre 2 y 5 años sean caprichosos con la comida. Ayúdales a aumentar los tipos de frutas y vegetales que |
| | comen al comerlos tú mismo! |
| | https://www.youtube.com/watch?v=VxgVxidCecM&feature=youtu.be |
| Week 19-Message 1 | |
| W. J. 40.55 | El agua no tiene porqué ser aburrida. Agrega rebanadas de frutas |
| Week 19-Message 2 | cítricas o bayas congeladas al agua para agregar sabor sin azúcar |



| | agregada. |
|---|---|
| Week 20- Message 1 | ¡Hagan comidas y recuerdos juntos! Es una lección para toda la vida! |
| Week 20- Message 2 | Pasa la pasta alrededor - Prueba pasta integral de diferentes formas y colores. Agrega un poco de aceite de oliva, queso bajo en grasa, verduras picadas y especias, o salsa de tomato para un almuerzo rápido o una cena. |
| Week 21- Message 1 | La estructura ayuda a los padres y a sus hijos. Los niños se siente seguros porque saben qué esperar. Los padres se sienten seguros porque saben cómo responder y responden de la misma manera todas las veces. |
| Week 21-Message 2 | Muchos padres tienen dificultades para que sus hijos se sienten en la mesa. Rutinas, como lavarse las manos y poner la mesa antes de sentarse, pueden ayudar a los niños a pasar de una actividad a otra. |
| Week 22- Message 1 | Mantén las papitas fritas y dulces fuera de la casa. Esto le enseñará a los niños que estos alimentos no se deben comer todos los días. |
| Week 22- Message 2 | Haz tu propio "trail mix" al combinar cereal integral, semillas o nueces y frutos secos. Es una merienda deliciosa que es fácil de llevar. |
| Week 23- Message 1 | Comenzar con porciones pequeñas en el plato puede ayudarle a evitar el desperdicio de comida si su hijo no tiene hambre. |
| Week 24- Message 1 | Intenta esto: a la hora de comer, ten preguntas para todos, por ejemplo: ¿Cuál es tu comida favorita de esta noche? o ¿Cuál fue la mejor parte de tu día? |
| Week 23- Message 2 | ¡Los niños pueden tomar buenas decisiones si les das una oportunidad! Deja que ellos elijan cómo probar nuevos alimentos: "¿Quieres probar el brócoli cocinado con su pasta o crudo con salsa?" |
| Week 24- Message 2 | ¡Las comidas saludables pueden ser fáciles y rápidas de preparar!<br>Prueba una tortilla con huevos, frijoles, salsa y queso bajo en grasa<br>para una comida MiPlato que a todos les encantará. |
| Week 25- Message 1 | Prioriza una comida placentera - no te preocupes por contar bocados ni te preocupes por lo que tu hijo ha comido (o no comido) |



| Week 25- Message 2 | Nadie tiene tiempo para un segundo trabajo como cocinero de todos. Sirve los mismos alimentos a todos en la familia. Si a tu hijo no le gusta un plato, intenta servir un acompañamiento que le guste, como fruta o frijoles. |
|---|---|
| Week 26- Message 1 | Tu trabajo es ofrecer una variedad de alimentos. El trabajo de tu hijo es decidir cuánto quiere comer. Habrá días en los que quiera comer solo un alimento y eso está bien. Mientras continúes brindando comidas y meriendas saludables, ellos obtendrán lo que necesitan. |
| Week 26- Message 2 | Gracias por participar en "Una Familia Fuerte Comienza en Casa" |

# **Control Materials English**



# Visit 1 Script

# Recorder Script:

(Prior to turning on recorder)

Thank you for meeting with me today. I wanted to remind you that I will be recording the session. The recording will be used to make sure each session is delivered the same way to each provider. As stated in the consent form, all of the recordings will be kept in a secure place and destroyed once we complete the study. The information from the recordings will only be shared with study staff. If you are ready I will turn on the recorder now.

# <u>Introduction</u>

Just a reminder, my name is XX – I am the support coach working with the University of Rhode Island. Thank you for participating in this study and opening your home to me. Your thoughts and experiences are important. Today we will meet for about 1 hour.

Before we get started, I would like to take a moment to talk about confidentiality or keeping your information private. Everything we discuss and all the questions you answer are private and confidential. We don't use your name or your child's name in our materials. What questions do you have about confidentiality?

# 5 Minutes



Study timeline handout





The main reason we are meeting today is to review the recording of you and your child that you sent us and discuss your thoughts about how you can engage with your child around reading. We will also discuss if you would like to make any changes to how you engage with your child around reading related activities.

Whether you make any changes to how you engage with your child around reading related activities is totally up to you. I am not here to judge you or talk you into making any changes. Remember, only you know what works best for you and your child. I am here to give you a chance to talk about your experiences and to see if what you are doing now fits with what you want for your child's future.

What questions do you have? If you have any questions during our talk please feel free to ask me.

Refer to Study timeline

After this first meeting today, I will be coming back in one month to discuss how you are doing and to do a special activity with your child around reading readiness and after that we will meet once more in your home. After the home visits, we will be calling you over the phone once a month for three more months and you will be receiving informative texts to accompany the newsletters each month. This information will help you make successful changes.

Do you have any questions for me?

Typical Day

To get started, you mentioned you have \_\_\_\_ child/ren.

What does a typical day look like for you and your child/ren?

Affirm and reflect statements regarding positive aspects of the participant's day with her child (children).

What about activities related to reading, tell me about some activities that you do with them.

Affirm and reflect statements regarding positive aspects of the participant's meal with her child (children)

When thinking about engaging with your child around reading related activities, are there are any challenges?

Tell me more about that. Affirm and reflect.

5 minutes



Key points: Do not try to solve problems -- our goal is to: Gather information let families know you are listening Hear their challenges and concerns Convey a non-judgmental tone.

Time management: If they share multiple changes:





# What parts work well? What else? or Tell me more about that. Affirm and reflect.

# What do you think helps you engage with your child around reading readiness activities?

Affirm and reflect self-motivational statements. Summarize Reading Readiness Activities Overview.

It sounds like you several changes, which one is the most important to vou?

Importance of participants role in creating a healthy environment

- Positive aspects of reading readiness activities with child/ren
- Confidence that she can make choices about what is right for her
- Intentions to want to do more reading readiness activities to engage children

# Review Video and Feedback Form:

The next section will focus on the target child from the video (not all children).

Now let's take a few minutes to review the recording that you sent

As a reminder, I'm not here to judge you or how you interact with your child. Only you know what's best for you and your child. I'm here to talk about your thoughts and experiences about engaging with your child around reading related activities.

> Play selected video segments (approx. 5 minutes of segment time).

# What sticks out from the video? What surprised you? What else?

If participant is unable to come up with anything or looks lost then say.

#### I'd like to share with you what I noticed if that's okay?

Wait for affirmation, then discuss participant strengths/areas where she demonstrated helpful reading activities.

If participant is unable to come up with anything or has misinformation then say If it's okay with you, I can share ways others have found helpful. Provide information with permission. Illicit participants thoughts on the information presented.

Tell me about the strategies you use to read with your child? Reflect.

#### 15 minutes



Feedback Sheet



Reading Video Clips on I-



Key Points:

Identify and elicit change talk. DESIRE: Want, wish, like ABILITY: Can, could, able REASON: Specific reason for change

NEED: Need to, have to, must, important, etc. (without stating specific reason)

COMMITMENT: Will, intend to,

going to, etc.

ACTIVATION: Ready to, willing to (without specific commitment) TAKING STEPS: Reporting recent specific action (step) toward change Responding to Change Talk:





What are some of the good things about those strategies? What else?

Reflect.

Affirm and reflect self-motivational statements: Summarize the Recording Review

Explore. Ask for elaboration: how, in what ways, why? Ask for examples: when was the last time this happened (e.g., for an adverse consequence).

Affirm. Express agreement, appreciation, encouragement, etc. for the desire/need/etc. to change. Reflect. This is the most common response to change talk – to offer a simple or complex reflection (. "I hear you saying that xxx" or "You feel it is difficult to xx") Summary. Think about the conversation like a field of flowers pick the sentences you would like to highlight, those that focus on change, and present them back to the family in a Change talk is also collected in "bouquet" summaries. You can select what to focus on in this process.

Set agenda & Review Handout

Asking Permission

Today we are going to talk about Why Reading is Important

The best practice for this topic is to introduce reading to children from an early age and make reading a part of each day.

Introduce Handout

15 minutes

Why is Reading Important

Identify and elicit change talk. It may be helpful to check off changes the family is interested in making on the handout for the goal setting activity.

Problem Solving/ Goal Setting

Now I would like to talk to you about setting a goal to introduce reading to children from an early age make reading a part of each



**Goal Sheet** 





day. You can set your own goal based on some of the materials we provided for you.

Why do you want to make this change? (Desire) (Reflection)

**How might you be able to do it? (**Ability) (Reflection)

What is one good reason for making the change? (Reasons) (Reflection)

How important is it, and why? (0-10)(Need) (Reflection)

What do you intend to do? (Commitment) (Reflection)

What are you ready or willing to do? (Activation) (Reflection)

What have you already done? (Taking Steps) (Reflection)

Record specific goal from the bottom of the goal-setting sheet on the data sheet. The goal of this section is to develop a specific goal and identify barriers. Leave the goal-setting sheet with the parent. They should choose one goal but can choose two if they would like. Please have a separate sheet for each goal.

We use this sheet to help people think about plans they may want to make. Keep in mind that your plan does not have to be a commitment to do something. It might be a plan to think about a way to make reading every day part of your routine. It's up to you to decide whether or not you want to make any changes – only you can make that decision.

If participant decides to make a plan say.

I can do all the writing, so you can concentrate on your plan.

Keys for Goal Setting: Goals should be:

- 1. Specific: Make sure goals are detailed. (Who, What, When, Where)
- 2. Measurable: Make sure the participant can identify what will happen when they achieve their goal.
- 3. <u>Achievable:</u> Goals should be realistic, not ideal
- 4. Relevant: Goals should relate to best practices for feeding and nutrition
- 5. <u>Time Bound:</u> Goal should have a timeline of when it will be met within the next time you meet

Performance Objectives: As part of the study we want participants to achieve the following If they have trouble coming up with their own goal here are some options:

- establish a daily reading routine with your child
- talk to your child all the time
- sing song with your child
- tell stories to your child
- something else related to getting your child ready to read, e.g



Guide participant with the following parts of the plan:

- · What is the plan
- · Reasons for the plan/why it is important
- Steps she can take to accomplish the plan
- · Barriers to the plan
- Possible solutions to the barriers
- Why she can do the plan

Summarize the plan.

Affirm plan and express optimism about change.

I think you have done a great job of coming up with ideas for your plan – I believe this plan can help you achieve the goals you have set for yourself.

Assess Readiness to Make Change

#### Motivation

Now that you have set a goal about reading in your home, I would like to know how are you feeling right now about \_[insert name of goal]

On a scale of 1 to 10 where 1 means you do not want to do this and 10 means you really want to do this. How would you rate yourself?

What made you pick that number and not a lower number (like 1 or 2)?

What would it take to get to a higher number (like 8 or 9)? If a 10

What would it take to keep you at a 10?

# Confidence

On a scale of 1-10, rate your confidence or ability to
\_\_\_\_\_in your home, where 1 means you are
not at all confident and 10 means you are very confident you can
maintain that change. How would you rate yourself?

What made you pick that number and not a lower number (like 1 or 2)?

What would it take to get you to a higher number (like 8 or 9)? If a 10 What would it take to keep you at a 10?

Summarize Example

# 15 minutes

- Record **Readiness** # in Redcap
- Record **Motivation #** in Redcap
- Record Confidence # in Redcap
- Record **Barriers** in Redcap
- Record **Facilitators** in Redcap



You feel that you are very motivated to make this change because you (first part of rating). You could...
In terms of being able to make this change, you feel that you are able to make this change because (first part of 1 or 2) You

able to make this change because (first part of 1 or 2) You believe you could increase your confidence if (insert comments from last part 9 or 10).

It seems you are ready to make this change and are committed to making this change.

#### Wrap up

We've covered a lot during our session – it has been great talking with you. If it's okay with you, I would like to take a moment to summarize our session today.

Use participant's words, highlight the major points and affirm commitment to change.

Before we finish, what questions might you have? Thank you for your time – I appreciate you welcoming me into your home.

Let's schedule our next appointment. Just as a reminder during our next visit, we will complete an activity with your child.

Thank you for taking the time to meet with me. I will see you again in one month but please call or text me if you have any questions before then.

Complete Visit Satisfaction Questionnaire

#### 5 minutes

- Record **Next Visit** in Redcap & Google Calendar
- Have participants complete satisfaction questionnaire



#### Recorder Script

Prior to turning on recorder

Hello, it's nice to see you again. I wanted to remind you that I will be recording the session. The recording will be used to make sure each session is delivered the same way to each family. As stated in the consent form, all of the recordings will be kept in a secure place and destroyed once we complete the study. The information from the recordings will only be shared with study staff. If you are ready I will turn on the recorder now.

Introduction

During our meeting today, we will

- 1. Check in around your goals from last visit
- 2. Talk about the joys of reading, wordless picture books and the importance of talking to your child
- 3. Set goals.
- 4. Do an activity together with you and your child

What questions do you have?

If you have questions as we go feel free to stop and ask me.

Assess

Tell me what sticks out from our last talk about the importance of reading with your child.

Afirm

Reflect

Thank you for sharing your experiences. It is helpful to know what types of successes and challenges you have faced as we begin to talk about preparing your child for reading and writing. It sounds like, Summarize

Reassess

Last time we talked you identified \_\_\_\_ & \_\_\_ as things you 10 minutes wanted to work on.

Last time you said this was X importance for you. How consistent is that with how you currently feel?

2 Minutes

2-5 minutes



Helpful to bring copies of visit 1 handout to provide if requested.






Last time you said you were x confidence how consistent is that with how you currently feel.

What were some of the strategies you came up with last visit.

How did trying the new strategies go for you and your child?

How satisfied are you with the new strategies you tried?

What is it about you that helped you try the new strategies?

What got in the way?

Relate to values /goals for reading readiness

#### Summarize & Reflect

It appears there are several things that went well You also discussed some areas with room for improvement

Redcap under Home Visit 1 encounter.



**Key Points:** 

Identify and elicit change talk. DESIRE: Want, wish, like

ABILITY: Can, could, able REASON: Specific reason for

change

NEED: Need to, have to, must, important, etc. (without stating

specific reason)

COMMITMENT: Will, intend to,

going to, etc.

ACTIVATION: Ready to, willing to (without specific

commitment)

TAKING STEPS: Reporting recent specific action (step)

toward change

Responding to Change Talk: Explore. Ask for elaboration: how, in what ways, why? Ask for examples: when was the last time this happened (e.g., for an adverse consequence). Affirm. Express agreement, appreciation, encouragement. etc. for the desire/need/etc. to change.

Reflect. This is the most common response to change talk – to offer a simple or complex reflection (. "I hear you saying that xxx" or "You feel it is difficult to xx") Summary. Think about the conversation like a field of flowers – pick the sentences you would like to highlight, those that focus on change. and present them back to the family in a Change talk is also collected in "bouquet"



summaries. You can select what to focus on in this process.

#### **Review Handout**

Can you tell me a little bit about how you interact with your child with words? How often/when do you talk to them?

What challenges do you have to engage them in talking?

What do you do well when you engage your child in talking/reading?

If it is okay with you, I would like to share some information about engaging with your child around talking to them. We will also talk about ways to include your child.

#### Review visit 2 handout

Review handout with parent, then ask the following:

Is there anything on here that you do already?

Afirm, reflect

Is there anything on here you are interested in or wanting to try?

Afirm, reflect

What concerns do you have about some of the recommendations?

Afirm, reflect

#### Problem Solving/ Goal Setting

Now I would like to talk to you about setting a goal to address what we have discussed today.

Why do you want to make this change? (Desire) (Reflection)

How might you be able to do it? (Ability) (Reflection)



Identify and elicit change talk. It may be helpful to check off changes the family is interested in making on the handout for the goal setting activity.

#### **@**15 minutes



Goal Sheet



Keys for Goal Setting: Goals should be:



What is one good reason for making the change? (Reasons) (Reflection)

**How important is it, and why?** (0-10)(Need) (Record number) (*Reflection*)

What do you intend to do? (Commitment) (Reflection)

What are you ready or willing to do? (Activation) (Reflection)

What have you already done? (Taking Steps) (Reflection)

Record specific goal from the bottom of the goal setting sheet on the data sheet. The goal of this section is to develop a specific goal and identify barriers. Leave the goal setting sheet with the parent.

So, your goal is to: (insert goal from last line on goal setting sheet). When we meet next time we will review this goal so keep this sheet with your materials.

- 1. Specific: Make sure goals are detailed. (Who, What, When, Where)
- 2. Measurable: Make sure the participant can identify what will happen when they achieve their goal.
- **3.** <u>Achievable</u> Goals should be realistic, not ideal
- **4.** Relevant Goals should relate to best practices for feeding and nutrition
- 5. <u>Time Bound</u> Goal should have a timeline of when it will be met within the next time you meet

Performance

Objectives: As part of the study we want participants to achieve the following:

Χ



| Assess Readiness to Make Change | 15 minutes |
|---|---|
| Motivation Now that you have set a goal about _[insert topic] for your family, I would like to know how are you feeling right now about _[inset name of goal] | Record <b>Readiness</b> in Redcap Record <b>Motivation #</b> in Redcap |
| On a scale of 1 to 10 where 1 means you do not want to do this and 10 means you really want to do this. How would you rate yourself? | Record Confidence # in Redcap |
| What made you pick that number and not a lower number (like 1 or 2)? | Record <b>Barriers</b> in Redcap |
| What would it take to get to a higher number (like 8 or 9)? If a 10 What would it take to keep you at a 10? | Record <b>Facilitators</b> in Redcap |
| Confidence On a scale of 1-10, rate your confidence or ability toi where 1 means you are not at all confident and 10 means you are very confident you can maintain that change. How would you rate yourself? | |
| What made you pick that number and not a lower number (like 1 or 2)? | |
| What would it take to get you to a higher number (like 8 or 9)? If a 10 What would it take to keep you at a 10? | |
| Sample Summary: You feel that you are very motivated to make this change because you (first part of rating). You could (insert comments from parent). In terms of being able to make this change, you feel that you are able to make this change because (first part of 1 or 2) You believe you could increase your confidence if (insert comments from last part 9 or 10). It seems you are ready to make this change and are committed to making this change. | |



#### Activity Now let's switch gears and do an activity. We can choose @30 minutes from these two activities. Is there one that you prefer? Allow parent to choose an activity from reading activities listed on the next pages. Wrap up Review Activity **@5** minutes How do you think xx worked? Are there things you liked about it? Things you didn't like about it? Is there anything you would do differently next time? Record Next Visit in Summarize visit Redcap & Google calendar Let's schedule our next visit. Just as a reminder we will **Recap Forms:** be doing another video feedback. What days of the week "Home Visit and Phone Call or times of day work best for you, keeping in mind that we Schedule" "Home Visit and will take 60 minutes. Phone Call Checklist and Satisfaction Questionnaire Just a reminder that you will receive text messages with helpful tips and recipes 2 x/week. Can I confirm the best number to reach you at? Also, we would like to ask you to complete a short survey on the IPAD about today. Provide IPAD to participant.

Thank you for taking the time to meet with me.



# Get Ready to Read!

Try this activity with the children to practice repetition and acting.

### Poetry in Motion

When children "act out" a poem, they learn to love its rhyme and rhythm. They connect feelings with the written word.

#### What you'll need:

Poems that rhyme, tell a story, and/or are written from a child's point of view.

#### What to do:

- Read a poem slowly to the children child. Be dramatic when you read. (In other words, "ham it up.")
- If there is a poem the children like, suggest acting out a favorite line.
- Suggest acting out a verse, a stanza, or the entire poem.
- Ask the children to make a face the way the character in the poem is feeling. Remember that facial expressions bring emotion into the performer's voice.

- Be an enthusiastic audience for the children. Applause is always nice.
- Mistakes are a fact of life, so ignore them.
- Poems are often short. This makes them easy for young children to repeat or remember lines and helps to build their confidence.







# Scribble, Draw, Write!

### Early writing activities!

Teaching young children writing skills helps them develop small motor skills. Children learn to hold pencils and crayons and control their drawing.

Try these activities with children to encourage early writing and reading readiness:

#### Sidewalk Chalk

Summer is great to practice drawing and writing skills outdoors.

You can buy colorful sidewalk chalks at a variety of stores.

- Be sure to get sidewalk chalk and not regular chalk. It is larger, sturdier and easier for young children to grip and use.
- Help children write their name.
- Draw pictures of things you see outside like trees, bugs, or your home.
   Label them, helping older children to spell out the letters as you write them.



#### Scribble Time

Make writing a daily activity along with reading.

Gather cheap paper tools. This includes newspapers, brown paper bags, or used wrapping paper.

- Let children use pencils, pens, markers or crayons to draw, scribble or decorate.
- Older toddlers can keep a notebook that is just for their "writing."
- Young toddlers should be allowed to scribble and draw unguided. This will help them become comfortable holding and controlling their writing tools.

You can guide preschoolers (3- and 4-years-old) by writing a letter for them and then having them practice writing it themselves.





# Play and Pretend!

Try this activity: TAKE A BOW!

Best for children ages 3-5

When children act out a poem or story, they show their own understanding of what it is about. They also grow as a reader by connecting emotions with written words.

Play-acting helps a child learn that there are more and less important parts to a story. They also learn how one thing in a story follows another.

#### What You Need:

Poems or stories written from a child's point of view. Things to use in a child's play (dress-up clothes, puppets).

#### What to Do:

- Read a poem or short story slowly.
   Read it with feeling, making the words seem important.
- Ask them to make a face to show the way the character in the poem is feeling. Making different faces adds emotion to the performer's voice. After the performance, praise the child for doing a good job.
- Have your child perform for you and the rest of the family.
   When the child finishes their performance, have them to take a bow. Clap and cheer loudly.
- Encourage your child to make up their own play from a story
  that they have read or heard. Tell them that it can be makebelieve or from real life. Help them to find or make things to go
  with the story—a pretend crown, stuffed animals, a broomstick,
  or whatever the story needs.



www.aplaceofourown.org



#### Visit 3 Script

#### Recorder Script:

(Prior to turning on recorder)

It's nice to see you again. I wanted to remind you that I will be recording the session. The recording will be used to make sure each session is delivered the same way to each family. As stated in the consent form, all of the recordings will be kept in a secure place and destroyed once we complete the study. The information from the recordings will only be shared with study staff. If you are ready I will turn on the recorder now.

#### 5 Minutes

#### Introduction

During our meeting today, we will

- 1. Check in around your goals from last visit
- 2. Review and Discuss Video-Recording that you sent
- 3. Review typical language development milestones and how your child gets ready to write
- 4. Set some goals

What questions do you have?

If you have questions as we go feel free to stop and ask me.

#### Assess

Tell me what sticks out from our last talk about the joys of reading, wordless picture books and the importance of talking to your child.

Helpful to bring copies of visit 1 handout to provide if requested.

Afirm Reflect

Thank you for sharing your experiences. It is helpful to know what types of successes and challenges you have faced as we begin to talk about preparing your child for reading and writing. It sowns you?

Time management: If they share multiple changes: It sounds like you several changes, which one is the most important to you?



### Review Video and Feedback Form

The next section will focus on the target child from the video (not all children).

Now let's take a few minutes to review the recording that you sent us.

As a reminder, I'm not here to judge you or how you interact with your child. Only you know what's best for you and your child. I'm here to talk about your thoughts and experiences about engaging with your child around reading related activities.

Play selected video segments (approx. 5 minutes of segment time).

What sticks out from the video?

What surprised you?

What else?

If participant is unable to come up with anything or looks lost then say:

I'd like to share with you what I noticed if that's okay?

Wait for affirmation, then discuss participant strengths/areas where she demonstrated healthy practices.

Set agenda & Review Handout

Asking Permission.

Today we are going to talk about Review typical language development milestones and how your child gets ready to write

Introduce Handout and discuss.

#### **@15** minutes



Feedback Sheet



Reading Video Clips on I-

PAD



Key Points:

Identify and elicit and respond to change talk.



Reading Aloud



Identify and elicit change talk. It may be helpful to check off changes the family is interested in making on the handout for the goal setting activity.





Time Management Tip
Reflections and exploration of
parents' thoughts on the content are
written into the script -- if time is
limited would be OK just to provide
the handout with brief explanation.

#### Problem Solving/ Goal Setting

Now I would like to talk to you about setting a goal to introduce reading to children from an early age make reading a part of each day. See performance objectives to help guide goals

Why do you want to make this change? (Desire) (Reflection)

**How might you be able to do it?** (Ability) (Reflection)

What is one good reason for making the change? (Reasons) (Reflection)

How important is it, and why? (0-10)(Need) (Reflection)
What do you intend to do? (Commitment) (Reflection)

What are you ready or willing to do? (Activation) (Reflection)

What have you already done? (Taking Steps) (Reflection)

Record specific goal from the bottom of the goal-setting sheet on the data sheet. The goal of this section is to develop a specific goal and identify barriers. Leave the goal-setting sheet with the parent.

#### 15 minutes



Goal Sheet



Keys for Goal Setting: Goals should be:

- 1. Specific: Make sure goals are detailed. (Who, What, When, Where)
- 2. Measurable: Make sure the participant can identify what will happen when they achieve their goal.
- 3. Achievable Goals should be realistic, not ideal
- **4.** Relevant Goals should relate to best practices for feeding and nutrition
- 5. <u>Time Bound</u> Goal should have a timeline of when it will be met within the next time you meet



We use this sheet to help people think about plans they may want to make. Keep in mind that your plan does not have to be a commitment to do something. It might be a plan to think about a way to make reading every day part of your routine. It's up to you to participants to achieve the following decide whether or not you want to make any changes - only you can make that decision.

Performance Objectives: As part of the study we want

- Establish a daily reading routine with your child
- Talk to your child all the time

Sing to your child

Record **Goal** in Redcap Upload picture of goal sheet (if more than one goal record both)

Guide participant, with the following parts of the plan:

- What is the plan
- Reasons for the plan/why it is important
- Steps she can take to accomplish the plan
- Barriers to the plan
- Possible solutions to the barriers
- Why she can do the plan

Summarize the plan.

Affirm plan and express optimism about change.

I think you have done a great job of coming up with ideas for your plan – I believe this plan can help you achieve the goals you have set for yourself.

Assess Readiness to Make Change Record **Readiness** in Redcap Motivation Now that you have set a goal about reading in your home, I would Record **Motivation** # in Redcap like to know how are you feeling right now about [inset name of Record Confidence # in Redcap goal] On a scale of 1 to 10 where 1 means you do not want to do this Record Barriers in Redcap and 10 means you really want to do this. How would you rate vourself? Record **Facilitators** in Redcap What made you pick that number and not a lower number (like 1 or 2)?

What would it take to get to a higher number (like 8 or 9)? If a 10

What would it take to keep you at a 10?

Confidence



On a scale of 1-10, rate your confidence or ability to in your home, where 1 means you are

not at all confident and 10 means you are very confident you can maintain that change. How would you rate yourself?

What made you pick that number and not a lower number (like 1 or 2)?

What would it take to get you to a higher number (like 8 or 9)? If a 10. What would it take to keep you at a 10?

Summarize

Example:

You feel that you are very motivated to make this change because you (first part of rating). You could...

In terms of being able to

make this change, you feel that you are able to make this change because (first part of 1 or 2) You believe you could increase your confidence if (insert comments from last part 9 or 10).

It seems you are ready to make this change and are committed to making this change.

#### Wrap up

We've covered a lot during our session – it has been great talking 5 minutes with you. If it's okay with you, I would like to take a moment to summarize our session today.

Use participant's words, highlight the major points and affirm commitment to change.

Before we finish, what questions might you have?

Thank you for your time - I appreciate you welcoming me into your home.

Let's schedule our next appointment, which will be over the phone. When would be a good time to call you. Also, could you please complete this short survey on the IPAD.

Complete Visit Satisfaction Questionnaire

Record Next Visit in Redcap & Google calendar

#### Recap Forms:

"Home Visit and Phone Call Schedule" "Home Visit and Phone Call Checklist and Satisfaction Questionnaire



### Phone Call Script

| Recorder Script | |
|---|---|
| (Prior to turning on recorder) | |
| | 5 Minutes |
| Hi Mr./Ms name is from the Strong | |
| materials to have ready during the call. | Goal Sheet available in Redcap under previous Home Visit encounter. |
| Introduction | <del></del> |
| To start, I wanted to know if you received your newsletter? Record: Yes / No | Key Points: |



#### Were you able to read through the newsletter?

Record: Yes / No

How useful was the newsletter? Would you say: very useful, somewhat useful, a little, or not at all useful?

Have them select one of the response options and record it on the Redcap.

#### Did you receive the text messages?

Record: Yes / No

#### Did you read the text messages? If no, why not?

Record: Yes / No If yes, ask:

How useful were the messages? Would you say: very useful, somewhat useful, a little, or not at all useful?

Have them select one of the response options and record it on the Redcap.

#### Did you have any issues or questions?

Provide a review of the topic you talked about in the last visit.

<u>Example:</u> "Last time we spoke, you mentioned that you wanted to prepare read with your child. You hoped this would get child's name excited about reading. Your goal was to read together 3 x/week. You also said that you were somewhat motivated to make this change (rated at 7) but did not feel very confident that you could do it every week(rated at 3). How did you do with your goal?

## On a scale of 1 to 10, What would you say your motivation level is now for XXX? What would you say your confidence level is now?

Use a reflection <u>or</u> an open-ended question to increase your understanding of how the participant is working on the goal:

If the participant had problems with the goal:

#### What do you think you could try differently next time?

Wrap up the topic:

Provide summary of progress and transition to next goal.

Restate goal, and review motivation and confidence.

Record if read newsletter and texts.
Record their usefulness.

Record on redcap if they met their goal: Circle Yes/ No



Example: It sounds like you were able to meet your goal on this topic and are pleased with your progress. How do you feel about the material you got in the mail?

#### Review New Topic:

We sent some information on (insert handout name). It reviews some of the topics we talked about during our sessions including (insert topics from targeted handout).

How do you feel about setting a goal for this topic?

#### 2 minutes



Month 4 handout Month 5 handout Month 6 handout

Identify and elicit change talk. It may be helpful to check off changes the family is interested in making on the handout for the goal setting activity.

#### Problem Solving/ Goal Setting:

Now I would like to talk to you about setting a goal to address the next/new? topic you selected (repeat the topic and objective here).

Why do you want to make this change? (Desire) (Reflection)

How might you be able to do it? (Ability) (Reflection)

What is one good reason for making the change? (Reasons) (Reflection)

#### 15 minutes



Goal Sheet



Keys for Goal Setting: Goals should be: 1. Specific: Make sure goals are detailed. (Who, What, When, Where) 2. Measurable: Make sure the participant can identify

123



| How important is it, and why? (0-10)(Need) (Record number) (Reflection) What do you intend to do? (Commitment) (Reflection) What are you ready or willing to do? (Activation) (Reflection) | what will happen when they achieve their goal. 3. Achievable Goals should be realistic, not ideal 4. Relevant Goals should relate to best practices for feeding and nutrition 5. Time Bound Goal should have a timeline of when it will be met within the next time you meet |
|---|---|
| What might get in the way of you meeting your goal to {restate goal}? | Record <b>Goal</b> in Redcap<br>Upload picture of goal<br>sheet (if more than one<br>goal record both) |
| Assess Readiness to Make Change | 15 minutes |
| Motivation Now that you have set a goal about _[insert topic] in your home daycare, I would like to know how are you feeling right now about _[inset] | Record <b>Readiness</b> in Redcap Record <b>Motivation</b> # in |
| name of goal] On a scale of 1 to 10 where 1 means | Redcap |
| you do not want to do this and 10 means you really want to do this. How | Redcap |
| you do not want to do this and 10 means you really want to do this. How would you rate yourself? What made you pick that number and not a lower number (like 1 or 2)? | Redcap Record Confidence # |



| Confidence On a scale of 1-10, rate your confidence or ability to, where 1 means you are not at all confident | |
|---|---|
| and 10 means you are very confident you can maintain that change. How | |
| would you rate yourself? | |
| What made you pick that number and not a lower number (like 1 or 2)? | |
| What would it take to get you to a higher number (like 8 or 9)? | |
| If a 10 What would it take to keep you at a 10? | |
| Sample Summary: You feel that you are very motivated to make this change because you (first part of rating). You could (insert comments from caregiver). In terms of being able to make this change, you feel that you are able to make this change because (first part of 1 or 2) You believe you could increase your confidence if (insert comments from last part 9 or 10). It seems you are ready to make this change and are committed to making this change. | |
| Wrap up You will receive a newsletter mailing in about 1-2 weeks. You will also continue to receive the text messages. | 2 minutes |
| Best phone number:(Note date of call) Thank you for taking the time to meet with me. I will talk with you again soon by phone. | Record <b>Next Visit</b> on redcap and Google calendar. <b>Recap Forms:</b> "Home Visit and Phone Call Schedule" "Home Visit and Phone Call Checklist and Satisfaction Questionnaire |



| *Note for last phone call<br>schedule per data<br>collection team calendar |
|---|



### **Control Text Messages**

| Message | |
|---|---|
| Delivery | |
| Scheduled | Message Content English |
| Week 1 - | |
| Welcome | *****welcome***** |
| Week 1 - | |
| Message 1 | Remember that reading introduces new sounds and words to children. |
| Week 1 - | |
| Message 2 | Reading can help your child expand their vocabulary once they start talking. |
| Week 2 - | Reading can help your child recognize new words which will set the foundation for |
| Message 1 | writing. |
| Week 2 - | Does your child have a favorite book? Reread it! Maybe your child will catch |
| Message 2 | something he/she didn't notice the first time. |
| | Regardless of language, reading, talking and singing to your child helps children use |
| Week 3 - | language. |
| Message 1 | |
| Week 3 - | Make some time to visit the library this week. Encourage your child to pick out a few |
| Message 2 | books. |
| Week 4 - | Reading can help children learn about printed words and how they are organized on a |
| Message 1 | page. |
| Week 4 - | |
| Message 2 | While reading, try to connect parts of the story to your child's life. |
| Week 5 - | When you're outside with your child, point out things such as stop signs. This will |
| Message 1 | allow your child to make the connection between words and their definitions. |
| Week 5 - | |
| Message 2 | This is your reminder to read for at least 15 minutes every day. |
| Week 6 - | Picture books are just as effective as regular books. They will teach your child to |
| Message 1 | comprehend the pictures. |
| Week 6 - | |
| Message 2 | Tell your child a story today. This will help give your child a headstart with reading. |
| Week 7 - | Read books with a repeated rhyme or phrase. Your child will begin to learn what |
| Message 1 | comes next . |
| Week 7 - | |
| Message 2 | Hi! This is your weekly reminder to read for at least 15 minutes every day. |



| Week 8 - | |
|---|---|
| Message 1 | Game time: Read a poem to your child and have him/her reenact the scenes. |
| Week 8 - | Activity of the week: After finishing a book, have a short discussion on the plot and |
| Message 2 | characters with your children. Compare your different perspectives. |
| Week 9 - | Label everyday things in your some, such as a chair or a table, to teach your child |
| Message 1 | which words connect to which objects. |
| Week 9- | Remember that the first three years are crucial to a child's language development. |
| Message 2 | Make the most of each day. |
| Week 10- | |
| Message 1 | Just a reminder to read for at least 15 minutes today. |
| Week 10- | |
| Message 2 | As you read, point out important words and how they are pronounced. |
| Week 11- | |
| Message 1 | Read books based on the alphabet. This will help your child learn each letter. |
| Week 11- | Spend some time teaching your child to spell his/her name out. Teach them how to |
| Message 2 | write other words too. |
| Week 12- | Play a guessing game with different letters. For example, "name animals whose |
| Message 1 | names start with the letter 'A'. " |
| Week 12- | |
| Message 2 | Read a wordless picture book and show your child how to interpret each picture. |
| Week 13- | Try this: Write down a set of words on a page and have your child outline each letter. |
| Message 1 | After each word is outlined, go over the pronunciation and meaning of that word. |
| Week 13- | |
| Message 2 | Try to always read with expression. This will keep your child focused and interested. |
| Week 14- | Look at the cover of each book you read together and try to predict what the story |
| Message 1 | will be about. |
| Week 14- | While reading, point out the difference between capital and lowercase letters. Explain |
| Message 2 | when each one should be used. |
| Week 15- | Talk out loud to your child from an early age so he/she will be able to use words |
| Message 1 | sooner. |
| Week 15- | Remember that most words in a child's vocabulary come from everyday encounters |
| Message 2 | with language. |
| Week 16- | Have a conversation with your child as you do every day things. For example, talk |
| Meesage 1 | about how coffee is usually hot and bananas are most often yellow. |
| Week 16- | |
| Message 2 | Always ask simple questions such as the color or shape of an object |



| Week 17- | |
|---|---|
| Message 1 | Create a routine, read to your child every night before going to bed! |
| Week 17- | |
| Message 2 | Language comes from many sources. Try to maximize encounters with these sources. |
| Week 18- | Have your child make up a story. This teaches children how to place their thoughts in |
| Message 1 | order |
| Week 18- | Encourage early writing skills. Help your child learn to scribble, draw and write a |
| Message 2 | letter. |
| Week 19- | It is important that your child understand that writing is simply "talking written |
| Message 1 | down". |
| Week 19- | Show your child how to hold a pencil. This is a necessary skill that will be introduced |
| Message 2 | when he/she starts school. |
| Week 20- | Encourage early writing skills by scheduling "scribble time" so your child can write |
| Message 1 | freely. |
| Week 20- | Children who know the letter of the alphabet before they go to kindergarten will do |
| Message 2 | better in school. |
| Week 21- | |
| Message 1 | Encourage your child to draw and scribble whenever possible. |
| Week 21- | Point to each word as you read so your child can associate the spoken word to its |
| Message 2 | respective written word. |
| Week 22- | Activity idea: purchase sidewalk chalk and help your child create masterpieces outside |
| Message 1 | on warm days. |
| Week 22- | Learning how to scribble and draw goes hand-in-hand with learning how to read. |
| Message 2 | Make sure it is a priority in your child's life. |
| Week 23- | |
| Message 1 | Encourage creative play to get children talking, inventing and exploring. |
| Week 23- | Play is a very important part of learning. "Play" helps children remember what they |
| Message 2 | learn. |
| Week 24- | |
| Message 1 | Activity Idea: Put together a puzzle with your child today. |
| Week 24- | |
| Message 2 | Point out words and signs you see and describe each one to your child. |
| Week 25- | When you have the opportunity, ask your child simple questions such as "what letter |
| Message 1 | does that word begin with?". |
| Week 25- | Try this! Provide empty cereal boxes, plastic bowls and dolls and have your child play |
| Message 2 | "house". |



| Week 26- | Play a board game meant for younger children. They can teach your child about |
|---|---|
| Message 1 | letters, colors, shapes and colors. |
| Week 26- | |
| Message 2 | Congrats! |

# Materiales para control en español



#### Guión de grabación:

(Antes de encender la grabadora)

Gracias por reunirse conmigo hoy. Quería recordarle que grabaré la sesión. La grabación se utilizará para asegurarse de que cada sesión se desarrolle de la misma manera. Como se indica en el formulario de consentimiento, todas las grabaciones se mantendrán en un lugar seguro y se destruirán una vez que completamos el estudio. La información de las grabaciones solo se compartirá con el personal del estudio. Si usted está listo voy a encender la grabadora ahora.

#### Introducción

Sólo un recordatorio, mi nombre es XX – soy una consejera trabajando con la Universidad de Rhode Island. Gracias por participar en este estudio y permitirme entrar a su casa. Lo que usted opina y sus experiencias son importantes. Hoy nos reuniremos durante aproximadamente 1 hora.

Antes de empezar, me gustaría tomar un momento para hablar de confidencialidad o mantener su información privada. Todo lo que discutimos y todas las preguntas que responde es privado y confidencial. No usamos su nombre ni el nombre de su hijo(a) en nuestros materiales. ¿Qué preguntas tiene sobre la confidencialidad?

La razón principal por la que nos encontramos hoy es para revisar la grabación que usted nos envió y discutir sus opiniones de cómo puede participar con su hijo en la lectura. También discutiremos si usted desea hacer cualquier cambio en cómo usted interactúa con su hijo en torno a la lectura y actividades relacionadas.

#### 5 Minutes



Utilice cronograma del



Si realiza cambios en la forma en que interactúa con su hijo(a) en torno a la lectura y actividades relacionadas, depende totalmente de usted. No estoy aquí para juzgarlo ni para convencerlo de que hagas cambios. Recuerde, sólo usted sabe lo que funciona mejor para usted y su hijo(a). Estoy aquí para darle la oportunidad de hablar sobre sus experiencias y ver si lo que está haciendo ahora encaja con lo que desea para el futuro de su hijo(a).

¿Qué preguntas tiene? Si tiene alguna pregunta durante nuestra Hablar por favor, siéntase libre de preguntarme.

Refiérase al cronograma del estudio:

Después de esta primera reunión de hoy, volveré en un mes para discutir su progreso y para realizar una actividad especial con su hijo(a) alrededor de la preparación para la lectura y después de eso nos reuniremos una vez más en su hogar. Después de las visitas al hogar, le llamaremos por teléfono una vez al mes durante tres meses más y va a recibir textos informativos para acompañar los boletines cada mes. Esta información le ayudará a realizar cambios exitosos.

¿Tiene alguna pregunta para me?

Día típico

Para empezar, mencionaste que tienes \_\_\_\_\_ hijo(s)(as).

¿Cuénteme acerca de un un día típico para usted y su hijo(s)(as)?

Afirme y reflexione sobre declaraciones de aspectos positivos del día del participante con su hijo(s)(as).

¿Cuénteme acerca de algunas de las actividades que hace con su les está escuchando. Presta atención hijo/a relacionado a la lectura?

Afirme y reflexione sobre declaraciones de aspectos positivos del día del participante con su hijo(s)(as).

Al pensar en interactuar con su hijo en torno a la lectura y actividades relacionadas, ¿hay algún desafío? Cuéntame más sobre eso.

Afirme y reflexione.

¿Qué partes funcionan bien? ¿Qué más? O Cuéntame más sobre cambios, ¿cuál es el más importante eso.

Afirme y reflexione.

5 minutos



#### **Puntos clave:**

No intente resolver problemas, nuestro objetivo es: Recopilar información y hacerles saber que se les está escuchando. Presta atención a sus retos y preocupaciones.

Transmite un tono sin criticar.

Gestión de tiempo: Si los padres comparten varios cambios: parece ser que le gustan varios cambios, ¿cuál es el más importante para usted?



¿Qué crees que te ayude a interactuar con tu hijo(a) en actividades para la preparación para la lectura?

Afirme y reflexione declaraciones automotivacionales.

Resuma visión general de actividades de preparación de lectura.

Importancia del rol de los participantes en la creación de un ambiente saludable.

Aspectos positivos de las actividades de la preparación para la lectura.

Confianza de que el padre puede tomar decisiones sobre lo que es correcto para su familia.

Intenciones de realizar más actividades de preparación para la lectura

#### Revisión de Video

La siguiente sección se centrará en el niño objetivo del video (no todos los niños).

Ahora vamos a tomar unos minutos para observar el video que nos envió.

Como recordatorio, no estoy aquí para juzgarte ni cómo interactúas con tu hijo. Sólo usted sabe lo que es mejor para usted y su hijo(a). Estoy aquí para hablar sobre sus opiniones y experiencias acerca de cómo interactuar con su hijo alrededor de la lectura y actividades relacionadas.

> Reproduce segmentos de vídeo seleccionados (aprox. 5 minutos de tiempo de segmento).

¿Qué sobresale del video?

¿Qué te sorprendió?

¿Qué más?

Si el participante no dice nada o parece perdido, entonces

Si está de acuerdo, me gustaría compartir con ustedes lo que noté del video

> Espere la afirmación y luego analice las fortalezas/áreas de los acción específica reciente (paso) participantes, donde ella/él demostró prácticas positivas.

#### 15 minutos



Hoja con retroalimentación



Observar video clips en I-

PAD



Puntos claves:

Identificar y provocar el cambio en la conversación.

DESEO: Querer, desear, gustar HABILIDAD: Poder, podria

RAZÓN: Razon especifica para el cambio

NECESIDAD: Necesitar, tener que, deber, importante, etc. (sin indicar la razón específica)

COMPROMISO: Voluntad, intención de, ir a, etc.

ACTIVACIÓN: Listo para, dispuesto a (sin compromiso específico) TOMANDO MEDIDAS: Reportar

hacia el cambio



¿Me puede contar acerca de las estrategias que usas para leer con tu hijo(a)? Reflexione

¿Cuáles son algunas de las cosas buenas de esas estrategias? ¿Qué más? Reflexione

Afirme y reflexione con declaraciones de automotivación. Resuma el Guión de grabación con el segundo video. Respondiendo a plática de cambio:

<u>Explorar.</u> Pida una explicación:
¿cómo, de ¿qué manera, por qué?
Pida ejemplos: cuándo fue la última
vez que sucedió esto? (por ejemplo,
para una consecuencia adversa).

<u>Afirmar.</u> Expresar acuerdo,
agradecimiento, ánimo, etc. para el
deseo/necesidad de cambio.

<u>Reflexionar.</u> Esta es la respuesta más
común sobre la conversación de
cambio: ofrecer una reflexión simple o
compleja. ("Lo escucho decir que xxx"
o "Siente que es difícil xx")

Resumen. Piense en la conversación como un campo de flores: elija las oraciones que desea resaltar, las que se centran en el cambio y preséntalas a la familia en un resumen como en un "ramo". Puedes seleccionar en qué enfocarte en este proceso.

Establecer agenda y revisión de folletos

Pedir permiso:

Hoy vamos a hablar de ¿Por qué leer es importante?

El procedimiento recomendado para este tema es para introducir la lectura a los niños desde una edad temprana y hacer que la lectura de una parte de cada día.

Presentar el folleto.

Resolución de problemas/establecimiento de metas:

Ahora me gustaría hablar con usted acerca de establecer una meta para introducir la lectura a los niños desde una edad temprana, que la lectura sea parte de cada día. Usted puede establecer sus propias metas basándose en cada uno de los materiales que le hemos dado.

¿Por qué quiere hacer este cambio? (Deseo)

#### 15 minutos



¿Por qué leer es importante?

Identifique y promueva conversación de cambio. Puede ser útil registrar los cambios que la familia está interesada en hacer en la hoja de establecimiento de metas.

#### 10 Minutos



Hoja de metas



Puntos clave: Guía para el establecimiento de metas. Las metas deberían ser:

134



(Reflexión)

¿Cómo podría hacerlo? (Capacidad)

(Reflexión)

¿Cuál es una buena razón para hacer el cambio? (Razones) (Reflexión)

¿Qué tan importante es, y por qué? (0-10) (Necesidad) (Anota el número)

(Reflexión)

¿Qué es lo que va a hacer? (Compromiso) (Reflexión)

¿Qué está listo y dispuesto a hacer? (Activación) (Reflexión)

¿Qué has hecho ya? (Tomando pasos) (Reflexión)

Registre la meta específico de la parte inferior de la hoja de establecimiento de metas en la hoja de datos. El objetivo de esta sección es desarrollar una meta específica e identificar barreras. Deje la hoja de establecimiento de metas con los padres. Ellos deben escoger una meta pero pueden escoger dos si quisieran. Tenga una hoja separada para cada meta.

Usamos esta hoja para ayudar a las personas a pensar en los planes que podrían querer hacer. Tenga en cuenta que su plan no tiene que ser un compromiso para hacer algo. Podría ser un plan para pensar en una manera de hacer que la lectura diaria sea parte de su rutina. Depende de usted decidir si desea o no hacer cambios -sólo usted puede tomar esa decisión.

Guíe a los participantes con las siguientes partes del plan:

- · ¿Cuál es el plan?
- · Razones para el plan/por qué es importante
- Pasos que puede seguir para lograr el plan
- · Las barreras para cumplir el plan
- Posibles soluciones a las barreras
- · ¿Por qué puede hacer el plan?

Resuma el plan.

- 1. Específico: Asegúrese de que las metas estén detallados. (Quien, que, cuando, donde)
- 2. Estimable: Asegúrese de que el participante pueda identificar lo que sucederá cuando logre su meta.
- 3. Realizable: Las metas deben ser realistas, no ideales.
- 4. Relevante: Las metas deben relacionarse con las mejores prácticas de alimentación y nutrición.
- 5. <u>Limite de Tiempo:</u>La meta debe tener un plazo de tiempo de cuándo se cumplirá (para la próxima visita)

Objetivos de Rendimiento: como parte del estudio queremos que los participantes logren lo siguiente:

- Establecer una rutina diaria de lectura con su hijo (a).
- Hablar con su hijo(a) todo el tiempo
- Cantar canciones con su hijo(a)
- Contarle historias o cuentos a su hijo (a)
- Algo relacionado con preparar a su hijo a la lectura



Afirme el plan y exprese optimismo sobre el cambio, Creo que has hecho un gran trabajo al desarrollar estas ideas para plan – creo que este plan puede ayudarte a alcanzar las metas que te has propuesto. Evalúe la preparación para hacer cambio 15 minutos Registre # Preparación en Motivación Redcap Ahora que ha establecido una meta sobre leer en su casa, me gustaría saber cómo te estás sintiendo ahora mismo sobre Registre Motivación en Redcap [nombre inserto de la meta] Registre Confianza en Redcap En una escala de 1 a 10 donde 1 significa que no quieres hacer Registre Barreras en Redcap esto y 10 significa que realmente quieres hacer esto. ¿Cómo te calificarías? Registre Facilitadores en Redcap ¿Qué te hizo elegir ese número y no un número más bajo (como 1 ó 2)? ¿Qué necesitarías para llegar a un número más alto (como 8 ó 9)? Si el 10, ¿ qué necesita para mantenerlo en un 10? Confianza En una escala de 1 a 10, evalúe su confianza/seguridad o la en su casa, donde 1 significa que no está seguro y 10 significa que está muy seguro de que puede mantener ese cambio. ¿Cómo se calificaría? ¿Qué te hizo elegir ese número y no un número más bajo (como 1 ó 2)? ¿Qué necesitarías para llegar a un número más alto (como 8 ó 9)? Si el 10, ¿qué necesita para mantenerlo en un 10? Resuma Eiemplo: Usted siente que está muy motivado para hacer este cambio porque usted (primera parte de la calificación). Podrías... En cuanto a poder hacer este cambio, usted siente que es capaz de hacer este cambio porque (primera parte de 1 ó 2) Usted cree que podría aumentar su confianza insertar comentarios de la última parte 9 ó 10).



| Parece que está listo para hacer este cambio y se compromete a haciendo este cambio. | |
|---|---|
| <u>Cierre</u> | 5 minutos |
| Hemos cubierto mucho durante nuestra sesión - ha sido muy<br>bueno hablar con usted. Si le parece bien, quisiera tomar un<br>momento para resumir nuestra sesión de hoy. | Registrar <b>Próxima visita en</b><br>Redcap y Google Calendar |
| Utilice las palabras del participante, resalte los puntos principales y afirme el compromiso de cambiar. | Los participantes deben completar cuestionario de satisfacción. |
| Antes de terminar, ¿qué preguntas podrías tener?<br>Gracias por su tiempo – le agradezco que me den la bienvenida a<br>su hogar. Programemos nuestra próxima cita. | |
| Gracias por tomarse el tiempo para reunirse conmigo. Nos veremos de nuevo en un mes, pero por favor llameme o envieme un mensaje de texto si tiene alguna pregunta antes de entonces. Antes de que me vaya si por favor puede completar estas preguntas en el IPAD. | |
| Completar cuestionario de satisfacción de visita. | |

Visit 2 Script

| Guión de grabación Antes de encender el grabador | 2 minutos |
|---|---|
| Hola, me alegro de verte de nuevo. Quería recordarle que grabaré la sesión. La grabación se | |



utilizará para asegurarse de que cada sesión se desarrolle de la misma manera con cada familia.

Como se indica en el formulario de consentimiento, todas las grabaciones se mantendrán en un lugar seguro y se destruirán una vez que completemos el estudio. La información de las grabaciones solo se compartirá con el personal del estudio. Si estás listo(a) voy a encender la grabadora ahora.

#### Introducción:

Durante nuestra reunión de hoy, vamos a

- 1. Repasar sus metas de la última visita
- 2. Hablar sobre las alegrías de leer, libros de imágenes sin palabras y la importancia de hablar con su hijo(a).
- 3. Establecer metas.
- 4. Hacer una actividad juntos con usted y su hijo(a).

¿Qué preguntas tienes?

Si tienes preguntas, siéntete libre de detenerme y preguntarme.

#### **Evaluar**

Dime lo que sobresale de nuestra última charla sobre la importancia de leer con su hijo(a).

Afirme, reflexione

Gracias por compartir sus experiencias. Es útil saber qué tipos de éxitos y desafíos ha enfrentado a medida que empezamos a hablar sobre cómo preparar a su hijo para comenzar a leer y escribir. Suena como, *Resuma* 

#### 2-5 minutos



Es útil llevar copias de los folletos de la visita 1 por si fueran solicitados de nuevo.

#### Reevaluar

La última vez que hablamos identifiqué \_\_\_ & \_\_\_ como cosas en las que querías trabajar.

La última vez que dijiste que esto era importante para ti. ¿Qué tan consistente es eso con la forma en la que te sientes actualmente?

#### 10 minutos



Visite hoja de metas 1 en Redcap bajo Home Visit 1 encounter.



138



La última vez que dijiste que tenías X seguridad/confianza. ¿Qué tan consistente es eso con la forma en la que te sientes actualmente?

¿Cuáles fueron algunas de las estrategias que surgieron en la última visita?

¿Cómo le fue probando las nuevas estrategias con su hijo?

¿Qué tan satisfecho(a) estás con las nuevas estrategias que has probado?

¿Qué es lo que te ayudó a probar las nuevas estrategias?

¿Qué se interpusuo en el camino?

Relacione con valores/metas para preparación para la lectura

#### Resumir y reflexionar:

Parece que hay varias cosas que les funcionó. También mencionó algunas áreas con espacio para mejorar...



Puntos claves: Identificar y provocar el cambio en la conversación.

<u>DESEO</u>: Querer, desear, gustar <u>HABILIDAD</u>: Poder, podria <u>RAZÓN</u>: Razon especifica para el cambio

NECESIDAD: Necesitar, tener que, deber, importante, etc. (sin indicar la razón específica)

COMPROMISO: Voluntad, intención de, ir a, etc.

ACTIVACIÓN: Listo para, dispuesto a (sin compromiso

específico)
TOMANDO MEDIDAS: Reportar
acción específica reciente (paso)
hacia el cambio

Respondiendo a plática de cambio:

Explorar. Pida una explicación: ¿cómo, de ¿qué manera, por qué? Pida ejemplos: cuándo fue la última vez que sucedió esto? (por ejemplo, para una consecuencia adversa). Afirmar. Expresar acuerdo. agradecimiento, ánimo, etc. para el deseo/necesidad de cambio. Reflexionar. Esta es la respuesta más común sobre la conversación de cambio: ofrecer una reflexión simple o compleja. ("Lo escucho decir que xxx" o "Siente que es difícil xx") Resumen. Piense en la conversación como un campo de flores: elija las oraciones que desea resaltar, las que se centran en el cambio y preséntalas a la familia en un resumen como en un "ramo". Puedes seleccionar en qué enfocarte en este proceso.



#### Revisar el folleto

- ¿Puedes contarme un poco sobre cómo interactúa usted con su hijo(a) usando palabras? ¿Con qué frecuencia/Cuándo hablas con ellos?
- ¿Qué desafíos tienes al hablar con ellos?
- ¿Qué haces bien cuando involucras a su hijo(a) en conversaciones/lectura?

Si te parece bien, me gustaría compartir una información acerca de cómo involucrar a tu hijo en conversaciones y que hables con ellos.

Revise el folleto de la visita 2.

Revise el folleto con el padre, luego pregunte lo siguiente:

- ¿Hay algo en este folleto que ya haces? Afirme. reflexione
- ¿Hay algo aquí que te interese o quieras probar? Afirme, reflexione
- ¿Qué inquietudes tiene acerca de algunas de las recomendaciones?

Afirme, reflexione

Resolución de problemas/establecimiento de metas:

Ahora me gustaría hablar con usted sobre el establecimiento de una meta para abordar lo que hemos discutido hoy.

- ¿Por qué quieres hacer este cambio? (Deseo) Reflexión
- ¿Cómo podrías hacerlo? (Capacidad) Reflexión

#### 5 minutos



Preparado para leer



Identifique y promueva conversación de cambio. Puede ser útil marcar las estrategias que la familia está interesada en probar en el folleto que incluye el establecimiento de metas.

15 minutos



Hoja de metas



Guía para el establecimiento de metas. Las metas deberían ser:

1. <u>Específico</u>: Asegúrese de que las metas estén detalladas. (Quien, que, cuando, donde)





¿Cuál es una buena razón para hacer el cambio? (Razones)

Reflexión

¿Qué tan importante es, y por qué? (0-10) Necesidad (Número de registro) Reflexión

¿Qué es lo que pretendes hacer? (Compromiso) Reflexión

¿Qué estás listo o dispuesto a hacer? (Activación) Reflexión

¿Qué has hecho ya? (Tomando medidas) Reflexión

> Registre la meta específico en la parte inferior de la hoja de establecimiento de metas. La meta de esta sección es desarrollar una meta específica e identificar barreras. Deje la hoja de establecimiento de metas con el padre.

Por lo tanto, su meta es: (insertar la meta de la última línea en la hoja de establecimiento de metas).

Cuando nos reunimos la próxima vez revisaremos esta meta, por lo tanto, mantenga esta hoja con sus materiales.

2. <u>Medible:</u> Asegúrese de que el participante pueda identificar lo que sucederá cuando logre su meta.

- 3. <u>Realizable</u>: Las metas deben ser realistas, no ideales.
- 4. Relevante: Las metas deben relacionarse con las mejores prácticas de alimentación y nutrición.
- 5. <u>Limite de Tiempo</u>:La meta debe tener un plazo de tiempo de cuándo se cumplirá (para la próxima visita)

Objetivos de rendimiento: como parte del estudio, queremos que los participantes cumplan lo siguiente:

Evalúe la preparación para hacer el cambio

Motivación

Ahora que ha establecido una meta acerca de
\_\_\_[Insertar tema]\_\_\_ para su familia, me gustaría
saber ¿cómo te sientes en este momento acerca de
\_\_\_ inserte meta]\_\_

En una escala de 1 a 10 donde 1 significa que no quieres hacer esto y 10 significa que realmente quieres hacer esto. ¿Cómo se calificaría usted mismo?

¿Qué te hizo elegir ese número y no un número más bajo (como 1 ó 2)?

#### 15 minutos

- Registrar **Preparación** en Redcap.
- Registrar **# Motivación** en Redcap.
- Registrar **# Confianza** en Redcap.
- Registrar **Barreras** en Redcap.



¿Qué se necesitaría para llegar a un número más alto (como 8 ó 9)? Si un 10, ¿qué necesita para mantener un 10? Confianza En una escala de 1-10, evalúe su confianza o su capacidad de \_\_\_\_\_ donde 1 significa que no está seguro y 10 significa que está muy seguro de que puede mantener ese cambio. ¿Cómo se calificaría usted mismo? ¿Qué te hizo elegir ese número y no un número más bajo (como 1 ó 2)? ¿Qué necesita para llegar a un número más alto (como 8 o 9)? Si el 10, ¿qué necesita para mantener un 10? Resumen Usted siente que está muy motivado para hacer este cambio porque usted (primera parte de la calificación). Puede (insertar comentarios de padre). En términos de poder hacer este cambio, usted siente que usted es capaz de hacer este cambio porque (primera parte de 1 o 2) usted cree que podría aumentar su confianza si (insertar comentarios de la última parte 9 o 10). Parece que está listo para hacer este cambio y está

#### Actividad

Ahora vamos a cambiar de tema y hacer una actividad. Usted puede escoger una actividad de estas dos.

comprometido a hacer este cambio.

Permite que el padre escoja un actividad de las activades de lectura mencionadas en las siguientes paginas.

#### 20-30 minutos

"Prepárate para leer" "Garabeta, Dibuja, Escribe" "Jugar e Inventar"



Compruebe la lista de los aparatos/utensilios disponibles Etc Libro de recetas

#### ! Puntos clave:

#### Cierre

Actividad de revisión

¿Cómo crees que funcionó la actividad?

¿Hay cosas que te gustaron?

¿Hay algo que no le gusto?

¿Hay algo que haría diferente la próxima vez?

#### Resumir visita

La próxima visita haremos otra revisión del video que nos mande. Programemos nuestra próxima visita. Qué días de la semana o horas del día funcionan mejor para usted, teniendo en cuenta que tomaremos 60 minutos.

Sólo un recordatorio de que usted recibirá mensajes de texto con consejos útiles y recetas 2 x/Week. ¿Puedo confirmar el mejor número para contactarlo? Gracias por tomarse el tiempo para reunirse conmigo.

Antes de que me vaya por favor puede completar este cuestionario en el IPAD.

#### 5 minutos

Registrar **Próxima visita** En Redcap "Home Visit and Phone Call Schedule" "Home Visit and Phone Call Checklist and Satisfaction Questionnaire Google Calendar


# ¡Prepárate para leer!

Intenta esta actividad con tu niño para practicar repetición y actuación.

#### Poesía en movimiento

Cuando los niños "recitan" un poema, aprenden a apreciar su ritmo y rima. Ellos conectan sus sentimientos con las palabras escritas.

#### Lo que necesitarás:

Poemas que rimen, cuenten una historia, y/o que estén escritos desde el punto de vista de un niño.

#### Cómo hacerlo:

- Léele un poema lentamente a los niños. Sé dramático/a cuando leas.
- Si hay un poema que a los niños les gusta, díles que reciten su parte favorita.
- Sugiere que dramaticen o reciten un verso, una estrofa o todo el poema.
- Pídele a los niños que utilicen gestos faciales para expresar cómo se siente el personaje del poema. Recuerda que las expresiones faciales agregan emoción a la voz del que está leyendo.
- Se una audiencia entusiasta para los niños. Los aplausos siempre son agradables.
- Los errores son inevitables, así que, ignóralos.
- Los poemas casi siempre son breves. Estos facilita que los niños repitan o recuerden las líneas y les ayuda a sentirse seguros/confiados.





## Garabatea, Dibuja, Escribe

## ¡Actividades de escritura!

Enseñarle a los niños pequeños habilidades de escritura les ayuda a desarrollar las habilidades motrices finas. Los niños aprenden a sostener lápices o crayones y a controlar sus dibujos.

Prueba estas actividades con los niños para fomentar su preparación para la lectura:

#### Dibujos en la acera:

El verano es fantástico para practicar las habilidades de lectura y escritura al aire libre. Puedes comprar coloridas tizas gruesas en muchas tiendas.



- Asegúrate de comprar tiza gruesa, no tiza común. Es más grande, más resistente y los niños pueden sujetarla y usarla con más facilidad.
- · Ayuda a los niños a escribir sus nombres.
- Haz dibujos de las cosas que ven, como árboles, insectos o su casa.
   Dale un nombre a cada cosa y ayuda a los niños más grandes a deletrear los nombres a medida que tu los escribes.

#### La hora de los garabatos:

Haz que la escritura y la lectura sean actividades diarias. Consigue materiales de papel baratos. Pueden ser periódicos, bolsas de papel marrón o papel para envolver usado.



- Los niños más grandes pueden tener un cuaderno solo para su "escritura."
- Los niños más pequeños deben tener la libertad de garabatear y dibujar sin instrucciones. Esto les ayuda a acostumbrarse a sostener y controlar sus herramientas de escritura.

Puedes orientar a los niños de edad preescolar (3 y 4 años) escribiendo una letra y pidiéndoles que practiquen escribiéndola ellos la mismos.





# Jugar é inventar

## Prueba esta actividad: ¡HAZ UNA REVERENCIA!

Se recomienda para niños entre 3 y 5 años

Cuando los niños dramatizan poemas o historias, demuestran su comprensión sobre lo que trató el cuento. También crecen como lectores cuando conectan sus emociones con las palabras escritas.

El juego de roles ayuda a que un niño aprenda que una historia tiene partes que son importantes y otras que no lo son. También entenderán cómo una parte de la historia lleva a la otra.

#### Lo que necesitas:

Poemas o cuentos escritos desde la perspectiva de un niño. Cosas para usar en una obra de teatro infantil (disfraces, títeres).

#### Cómo juegar:

- Lee lentamente un cuento o poema.
   Lee con sentimiento, para que las palabras parezcan importantes.
- Pídele a los niños que hagan la cara que representa cómo se siente el personaje del poema. Hacer las caras le agrega emoción a la voz del que lee.

Después de la actuación, felicita a los niños por el trabajo que hicieron.

- Pide a un niño que actúe frente a todo el grupo.
   Cuando el niño haya terminado, pide a los demás que le hagan una reverencia. Aplaudan y celebren con mucho ruido.
- Motiva a los niños para que inventen su propia obra con base a un cuento que hayan escuchado o leído.

Diles que la obra puede estar basada en hechos reales o imaginarios. Ayúdales a encontrar o crear cosas que acompañen la historia: una corona de juguete, osos de peluche, un palo de escoba o lo que haga falta para contar la historia.

www.aplaceofourown.org





#### Guión de grabación:

(Antes de encender la grabadora)

Es bueno verte de nuevo. Quería recordarle que grabaré la sesión. La grabación se utilizará para asegurarse de que cada sesión se desarrolle de la misma manera con cada familia. Como se indica en el formulario de consentimiento, todas las grabaciones se mantendrán en un lugar seguro y se destruirán una vez que completemos el estudio. La información de las grabaciones solo se compartirá con el personal del estudio. Si estás listo voy a encender la grabadora ahora.

Durante nuestra reunión de hoy, vamos a

- 1. Repasar las metas de la última visita
- 2. Revisar y discutir la grabación de vídeo que envió
- 3. Revisar los el desarrollo del lenguaje y cómo su hijo(a) se prepara para escribir
- 4. Establecer algunos metas

Qué preguntas tienes?

Si tienes preguntas, siéntase libre de detenerme y preguntarme.

#### Evaluar

Dime lo que sobresale de nuestra última charla sobre las alegrías de leer, libros de imágenes sin palabras y la importancia de hablar con su hijo.

> Afirme Reflexione

Gracias por compartir sus experiencias. Es útil saber qué tipos de éxitos y desafíos ha enfrentado a medida que empezamos a hablar sobre cómo preparar su hijo para leer y escribir. Suena como, Resumir

#### Revisión Video

La siguiente sección se centrará en el(la) niño(a) objetivo del video (no todos los niños).

#### 5 minutos

#### 10 minutos

Llevar copias de los folletos de la visita 1 por si fueran solicitados de nuevo.

Gestión del tiempo: si comparten varios cambios: Suena como que le interesan varios

Suena como que le interesan varios cambios, cuál es el más importante para usted?

#### 15 minutos



Hoja con retroalimentación

147



Ahora vamos a tomar unos minutos para revisar la grabación que nos envió.

Como recordatorio, no estoy aquí para juzgarte ni cómo interactúas con tu hijo. Sólo usted sabe lo que es mejor para usted y su hijo. Estoy aquí para hablar sobre sus pensamientos y experiencias acerca de cómo interactuar con su hijo alrededor de la lectura y actividades relacionadas.

Reproduce segmentos de vídeo seleccionados (aprox. 5 minutos).

¿Qué sobresale del video? ¿Qué te sorprendió? ¿Qué más?

Si el participante no dice nada o parece perdido, entonces diga, Me gustaría compartir con ustedes lo que noté que está bien?

> Espere la afirmación y luego analice las fortalezas/áreas de los participantes donde demostró prácticas positivas. Luego haga lo mismo con las prácticas negativas.

Video Clips del tiempo de



Puntos clave:

Identifique y promueva conversación de cambio.

#### Establecer agenda y revisión de folletos:

Pida permiso:

Hoy vamos a hablar de Revise los hitos típicos del desarrollo del lenguaje y cómo su hijo se prepara para escribir

Presentar el folleto y discutir.

#### 10 minutos

■Ve a través del volante con ellos



Identifique y promueva conversación de cambio. Puede ser útil marcar las estrategias que la familia está interesada en probar en el folleto que incluye el establecimiento de metas.

Consejo para manejo del tiempo: Las reflexiones y la exploración de los pensamientos y opiniones de los padres sobre el contenido están en el guión - si el tiempo es limitado, está bien proporcionar solamente una breve explicación del folleto.



| Resolución de problemas/establecimiento de metas: | 15 minutos |
|---|---|
| Ahora me gustaría hablar con usted acerca de establecer una<br>meta para introducir la lectura a los niños desde una edad<br>temprana y hacer que la lectura sea parte de cada día.<br>Ver objetivos de rendimiento para ayudar a guiar las metas. | Hoja de metas |
| ¿Por qué quieres hacer este cambio? (Deseo)<br>Reflexión | Guía para el establecimiento de metas. Las metas deberían ser: |
| ¿Cómo podrías hacerlo? (Capacidad)<br>Reflexión | 1. Específico: Asegúrese de que las metas estén detalladas. (Quien, que, cuando, donde) |
| ¿Cuál es una buena razón para hacer el cambio? (Razones)<br>Reflexión | 2. Estimable: Asegúrese de que el participante pueda identificar lo que sucederá cuando logre su meta. |
| ¿Qué tan importante es, y por qué? (0-10) Necesidad<br>(Número de registro)<br>Reflexión | 3. Realizable: Las metas deben ser realistas, no ideales. 4. Relevante: Las metas deben |
| ¿Qué es lo que pretendes hacer? (Compromiso)<br>Reflexión | relacionarse con las mejores<br>prácticas de alimentación y nutrición.<br>5. Limite de Tiempo:La meta debe |
| ¿Qué estás listo o dispuesto a hacer? (Activación)<br>Reflexión | tener un plazo de tiempo de cuándo<br>se cumplirá (para la próxima visita) |
| : Qué has hecho va? (Tomando medidas) | |

Reflexión



Registre la meta específica en la parte inferior de la hoja de establecimiento de metas. El objetivo de esta sección es desarrollar una meta específica e identificar barreras. Deje la hoja de establecimiento de metas con el padre.

Usamos esta hoja para ayudar a las personas a pensar en los planes que podrían querer hacer. Tenga en cuenta que su plan no tiene que ser un compromiso para hacer algo. Podría ser un plan para pensar en una manera de hacer que la lectura diaria sea parte de su rutina. Depende de usted decidir si desea o no hacer cambios -sólo usted puede tomar esa decisión.

Si el participante decide hacer un plan, diga:

Yo puedo me puedo encargar de escribir, para que puedas concentrarte en tu plan.

Guíe a los participantes con las siguientes partes del plan:

- · ¿Cuál es el plan?
- · Razones para el plan/por qué es importante
- · Pasos que puede seguir para lograr el plan
- · Las barreras para cumplir el plan
- · Posibles soluciones a las barreras
- ¿Por qué puede hacer el plan?

Resuma el plan.

Afirme el plan y exprese optimismo sobre el cambio:

Creo que has hecho un gran trabajo al desarrollar estas ideas para plan – creo que este plan puede ayudarte a alcanzar las metas que te has propuesto.

Objetivos de Rendimiento: como parte del estudio queremos que los participantes logren lo siguiente:

- Establecer una rutina diaria de lectura con su hijo (a).
- Hablar con su hijo(a) todo el tiempo
- Cantar canciones con su hijo(a)
- Contarle historias o cuentos a su hijo (a)
- Algo relacionado con preparar a su hijo a la lectura

Registre **Meta** en Redcap. Suba una foto de la hoja (si hay más de una meta, registre ambos

#### Evalúe la preparación para hacer cambio

Motivación

Ahora que ha establecido una meta sobre leer en su casa, me gustaría saber como estás sintiendo ahora mismo sobre \_[inserte meta]

En una escala de 1 a 10 donde 1 significa que no quieres hacer esto y 10 significa que realmente quieres hacer esto. ¿Cómo te calificarías?

#### 15 minutos

- Registrar **Preparación** en Redcap
- Registrar # Motivación en Redcap
- Registrar # Confianza en Redcap
- Registrar **Barreras** en Redcap



| ¿Qué te hizo elegir ese número y no un número más bajo (como 1 2)? | Registrar <b>Facilitadores</b> en Redcap |
|---|---|
| ¿Qué se necesitaría para llegar a un número más alto (como 8 ó<br>9)? | . toucup |
| Si el 10 ¿qué necesitas para mantener un 10? | |
| Confianza En una escala de 1-10, evalúe su confianza/seguridad o la capacidad deen su casa, donde 1 significa que no está seguro y 10 significa que está muy seguro de que puede mantener ese cambio. | |
| ¿Cómo se calificaría? | |
| ¿Qué te hizo elegir ese número y no un número más bajo (como 1 ó 2)? | |
| ¿Qué se necesita para llegar a un número más alto (como 8 ó 9)? | |
| Si el 10 ¿Qué necesitas para mantener un 10? | |
| Resuma | |
| Usted siente que está muy motivado para hacer este cambio porque usted (primera parte de la calificación). Podrías | |
| En cuanto a poder hacer este cambio, usted siente que usted es capaz de hacer este cambio porque (primera parte de 1 ó 2) | |
| Usted cree que podría aumentar su confianza insertar comentarios de la última parte 9 ó 10). Parece que está listo para hacer este cambio y se compromete a haciendo este cambio. | |
| <u>Cierre</u> | 5 minutos |
| Hemos cubierto mucho durante nuestra sesión - ha sido una muy buena conversación. Si le parece bien, quisiera tomar un momento para resumir nuestra sesión de hoy. Utilice las palabras del participante, resalte los puntos principales y afirme el compromiso de cambiar. | Registrar <b>Próxima visita</b> en Redcap "Home Visit and Phone Call Schedule" "Home Visit and Phone Call Checklist and Satisfaction Questionnaire" y Google Calendar |
| Antes de terminar, ¿qué preguntas podrías tener? | |
| Gracias por su tiempo – le agradezco que me den la bienvenida a<br>su hogar. La próxima vez, vamos a hablar por teléfono, que día, y | |



qué hora le quedaría bien? También le estaremos mandando materiales.

Antes de que me vaya, si puede completar este cuestionario en el IPAD?

Por favor llámeme o envieme un mensaje de texto si tiene alguna

Completar el cuestionario de satisfacción.

pregunta antes de entonces.



| Recorder Script: | |
|---|---|
| (Antes de prender la grabadora) | |
| Hola Señor/Señora mi nombre es<br>soy del estudio de las Familia Fuertes Comienzan en Casa de la<br>Universidad de Rhode Island. Lo/la llamo para hacer nuestra sesión | Redcap en el anterior |
| telefónica del mes. Gracias por su tiempo el dia de hoy. Quería recordarle que estaremos grabando esta sesión. Si está listo/a voy a encender la grabadora ahora. Le enviamos unos materiales por correo, si los tiene a la mano, nos podemos referir a ellos durante la llamada. También vamos | <b></b> |
| a usar su hoja de metas. | Puntos clave:<br>Reafirme la meta y<br>chequee motivación y |
| | confianza |
| | Registre si leyó folleto de información y textos, y |
| ¿Pudo leer la hoja de información/folleto?<br>Respuesta: Sí / No | si le parecieron útiles. |
| ¿Tiene alguna pregunta acerca de esa información? | Registre en Redcap si<br>se cumplió su meta: |
| 1 A / | seleccione Sí/ No |
| ¿Recibió los mensajes de texto?<br>Respuesta: Sí / No | |
| Leyó los mensajes de texto? Si no, por qué no?<br>Respuesta: Sí / No<br>Si sí, pregunte: | |
| ¿Qué tan útiles fueron los mensajes de texto? Diría que fueron: muy útiles, algo útiles, un poco útiles, o para nada útiles? | |



Haga que seleccione una de las opciones de respuesta y registre la respuesta en Redcap.

#### ¿Tuvo algún problema o pregunta?

Proporcione un resumen del tema del que se habló en la última visita. <u>Ejemplo:</u> "La última que que hablamos, usted mencionó que quería preparar leer más con su hijo(a). Usted pensaba que esto haría que "nombre del niño(a)" se emocionara mas al leer. Su meta era leer junto con su hijo(a) 3 veces por semana. También dijo que estaba algo motivado(a) por hacer este cambio (calificado con un 7) pero no se sentía tan seguro que podría hacerlo cada semana (calificado con un 3). ¿Cómo le fue con esta meta?

En una escala del 1 al 10, ¿cuál diría que es su nivel de motivación ahora para XXX? ¿Cuál diría que es su nivel de confianza/seguridad ahora?

Reflexione **o** haga una pregunta abierta para entender mejor cómo el participante está trabajando para alcanzar su meta: Si el participante tuvo problemas con la meta:

Qué cree que podría hacer de manera diferente la próxima vez?"

#### Cerrar el tema:

Proporcione un resumen del progreso y haga una transición al próximo objetivo o meta

Ejemplo: Parece que pudo alcanzar su meta en este tema y está satisfecho con su progreso.



### Revise Tema Nuevo:

Nosotros le enviamos información sobre (insertar nombre del folleto).

Este le explica algunos de los temas de los que hablamos durante nuestras sesiones, incluyendo (insertar temas del folleto).

¿Cómo se siente al establecer una meta para este tema?

#### 2 minutos



Folleto mes 4 Folleto mes 5 Folleto mes 6

Identifique y promueva conversación de cambio. Puede ser útil marcar las estrategias que la familia está interesada en probar en el folleto que incluye el establecimiento de metas.



#### Resolución de Problemas/ Establecimiento de Metas:

Ahora me gustaría hablarle acerca de establecer una meta para abordar el nuevo/siguiente tema que seleccionó (repita el tema y la meta aquí).

¿Por qué quiere hacer este cambio? (Deseo) (Reflexión)

¿Cómo podría hacerlo? (Capacidad) (Reflexión)

¿Cuál es una buena razón para hacer este cambio? (Razones) (Reflexión)

¿Qué tan importante es, y por qué? (0-10) (Necesidad) (Registre Número) (Reflexión)

¿Que intentará hacer? (Compromiso) (Reflexión)

¿Qué está listo o dispuesto a hacer? (Activación) (Reflexión)

¿Qué ha hecho ya? (Pasos tomados) (Reflexión)

Registre la meta específica en la parte inferior de la hoja de establecimiento de metas. Registre esta meta específica en Redcap. La meta de esta sección es desarrollar una meta específica e identificar los obstáculos.

#### Entonces, su meta es:

Insertar meta de la última línea de la hoja de establecimiento de meta.

#### Evaluando Obstáculos

¿Qué podría interponerse en su camino para cumplir su meta replantear meta

Cuando volvamos a hablar por teléfono, revisaremos esta meta, así que guarde esta hoja con sus materiales.

#### 10 minutos

#### 15 minutes



Hoja de metas



Puntos clave:

Guía para el establecimiento de metas. Las metas deberían ser:

- 1. Específico: Asegúrese de que las metas estén detallados. (Quien, que, cuando, donde)
- 2. Estimable: Asegúrese de que el participante pueda identificar lo que sucederá cuando logre su meta
- 3. <u>Realizable:</u> Las metas deben ser realistas, no ideales.
- 4. Relevante: Las metas deben relacionarse con las mejores prácticas de alimentación y nutrición.
- 5. <u>Limite de Tiempo</u>: La meta debe tener un plazo de tiempo de cuándo se cumplirá (para la próxima visita/llamada)
- Suba una foto de la hoja de metas (si más de una, suba ambas)







| Evalúe la preparación para hacer el cambio | 15 minutos |
|---|---|
| gustaria saber como se siente acerca de[mscrtar nombre de la | Registre <b>Preparación</b><br>en Redcap |
| meta] En una escala del 1 al 10, en donde 1 significa que no quiere hacer esto y 10 significa que realmente quiere hacer esto. | Registre <b># Motivación</b><br>en Redcap |
| ¿Cómo se calificaría? | Registre # Confianza |
| ¿Qué le hizo elegir ese número y no un número más bajo (como 1 ó 2)? | en Redcap |
| ¿Qué necesitaría para llegar a un número más alto (como 8 ó 9)? Si un<br>10, ¿qué necesitaría para mantener un 10? | Registre <b>Barreras</b> en<br>Redcap |
| | Registre Facilitadores en Redcap |
| mismo y 10 significa que está muy seguro de que podrá mantener el cambio. | |
| ¿Cómo se calificaría?<br>¿Qué le hizo elegir ese número y no un número más bajo (como 1 ó 2)? | |
| ¿Qué necesitaría para llegar a un número más alto (como 8 ó 9)? Si un<br>10, ¿Qué necesitarías para mantener un 10? | |
| Resumen de Ejemplo: Sientes que estás muy motivado para hacer este cambio porque tú (primera parte de la calificación). Usted podría (insertar comentarios del cuidador). En términos de poder hacer este cambio, siente que puede hacerlo porque (primera parte de 1 ó 2). Cree que podría aumentar su confianza si (inserte comentarios de la última parte 9 ó 10). Parece que está listo para hacer este cambio y está comprometido a hacer este cambio. | |



| <u>Cierre</u> | 2 minutos |
|---|---|
| Alrededor de 2 semanas después, usted recibirá otro correo y lo/la llamaré de nuevo para revisar la meta y discutir sobre el próximo tema en el que querrá trabajar y para establecer nuevas metas para este tema. Asegúrese de tener la hoja de establecimiento de metas para llenarla durante la llamada | Registre <b>Siguiente Visita</b> en Redcap y Google Calendar *Nota para calendario de la próxima llamada telefónica según el equipo de recolección de datos |
| ¿Cuál sería el mejor día y hora para nuestra próxima llamada? (Anote la fecha de la llamada) Mejor número de teléfono: | |



## **Text Messages**

| Entrega de<br>mensajes<br>programada | Contenido del mensaje inglés |
|---|---|
| Semana 1-<br>Bienvenido | Bienvenido * * * * * |
| Semana 1-mensaje<br>1 | Recuerde que la lectura introduce nuevos sonidos y palabras a los niños. |
| Semana 1-mensaje<br>2 | La lectura puede ayudar a tus hijos a expandir su vocabulario una vez que empiecen a hablar. |
| Semana 2-mensaje<br>1 | La lectura puede ayudar a tu hijo a reconocer palabras nuevas que establecerá las base para la escritura. |
| Semana 2-mensaje<br>2 | ¿Su hijo tiene un libro favorito? Vuelve a leerlo! Tal vez tu hijo notara algo que no notó la primera vez. |
| Semana 3-mensaje<br>1 | Independientemente del idioma, leer, hablar y cantarle a tu hijo le va a ayudar a usar el lenguaje fácilmente. |
| Semana 3-mensaje<br>2 | Haz tiempo para visitar la biblioteca esta semana. Anima a tu hijo para que escoja algunos libros. |
| Semana 4-mensaje<br>1 | La lectura puede ayudar a los niños a aprender sobre las palabras impresas y cómo se organizan en una página. |
| Semana 4-mensaje<br>2 | Mientras lees, intenta conectar partes de la historia a la vida de tu hijo. |



| Semana 5-mensaje<br>1 | Cuando estés afuera con tu hijo, señala cosas como las señales de parada. Esto permitirá que tu hijo haga la conexión entre las palabras y sus definiciones. |
|---|---|
| Semana 5-mensaje<br>2 | Este es tu recordatorio de leer durante al menos 15 minutos todos los días. |
| Semana 6-mensaje<br>1 | Los libros de solo imágenes son tan efectivos como los libros con palabras Le enseñarán a tu hijo a comprender las imágenes. |
| Semana 6-mensaje<br>2 | Cuéntale un cuento a tu hijo hoy. Esto le ayudará a que su hijo comience con la lectura. |
| Semana 7-mensaje<br>1 | Lee libros con una rima o frase repetida. Su hijo comenzará a aprender lo que viene después. |
| Semana 7-mensaje<br>2 | ¡Hola! Este es su recordatorio semanal de leer por lo menos 15 minutos todos los días. |
| Semana 8-mensaje<br>1 | Tiempo para jugar: Leela un poema a tu hijo y pídele que actúe las escenas. |
| Semana 8-mensaje<br>2 | Actividad de la semana: después de terminar un libro, ten una breve discusión con sus hijos sobre la historia y los personajes. Compara sus diferentes perspectivas. |
| Semana 9-mensaje<br>1 | Etiqueta las cosas cotidianas en tu casa, como una silla o una mesa, para enseñarle a tu hijo qué palabras se conectan a qué objetos. |
| Semana 9-mensaje<br>2 | Recuerda que los primeros tres años son cruciales para el desarrollo del lenguaje de un niño. Aprovecha al máximo cada día. |
| Semana 10-<br>mensaje 1 | Sólo un recordatorio de leer por lo menos 15 minutos hoy. |



| Semana 10-<br>mensaje 2 | Al leer, señale las palabras importantes y cómo se pronuncian. |
|---|---|
| Semana 11-<br>mensaje 1 | Lee libros basados en el alfabeto. Esto le ayudará a tu hijo a aprender cada letra. |
| Semana 11-<br>mensaje 2 | Dedica tiempo para enseñarle a tu hijo a deletrear su nombre. Enséñale a escribir otras palabras también. |
| Semana 12-<br>mensaje 1 | Jueguen un juego de adivinanzas con diferentes letras. Por ejemplo, "nombra animales cuyos nombres comiencen con la letra ' A '." |
| Semana 12-<br>mensaje 2 | Lean un libro de imágenes sin palabras y muéstrale a tu hijo cómo interpretar cada imagen. |
| Semana 13-<br>mensaje 1 | Prueba esto: Anota un conjunto de palabras en una página y haz que tu hijo delinee cada letra. Luego de delinear cada palabra, repasa la pronunciación y el significado de esa palabra. |
| Semana 13-<br>mensaje 2 | Intenta leer siempre con emoción. Esto mantendrá a su hijo concentrado e interesado. |
| Semana 14-<br>mensaje 1 | Mira la portada de cada libro que lean juntos y trata de predecir con tu hijo/a de qué tratará la historia. |
| Semana 14-<br>mensaje 2 | Mientras lees, señala la diferencia entre mayúsculas y minúsculas. Explica cuándo se debe usar cada una. |
| Semana 15-<br>mensaje 1 | Háblale en voz alta a tu hijo desde una edad temprana para que él/ella empiece a usar palabras antes. |
| Semana 15-<br>mensaje 2 | Recuerda que la mayoría de las palabras en el vocabulario de un niño provienen de encuentros diarios con el lenguaje. |



| Semana 16-<br>mensaje 1 | Conversa con tu hijo acerca de las cosas de todos los días. Por ejemplo, hablar de cómo el café suele estar caliente y cómo los plátanos son generalmente amarillos. |
|---|---|
| Semana 16-<br>mensaje 2 | Siempre haz preguntas simples como por ejemplo, el color o la forma de un objeto |
| Semana 17-<br>mensaje 1 | Crea una rutina- leale or miren un libro antes de dormir todas las noches! |
| Semana 17-<br>mensaje 2 | El lenguaje viene de muchas fuentes. Trata de maximizar los encuentros con estas fuentes. |
| Semana 18-<br>mensaje 1 | Haz que tu hijo invente una historia. Esto les enseña a los niños a poner sus pensamientos en orden. |
| Semana 18-<br>mensaje 2 | Fomenta las habilidades de escritura tempranas. Ayudale a tu hijo para que aprenda a garabatear, dibujar y escribir una carta. |
| Semana 19-<br>mensaje 1 | Es importante que tu hijo entienda que la escritura es simplemente "hablar por escrito". |
| Semana 19-<br>mensaje 2 | Muéstrale a tu hijo cómo sostener un lápiz. Esta es una habilidad necesaria que se introducirá cuando empiece la escuela. |
| Semana 20-<br>mensaje 1 | Fomenta las habilidades de escritura temprana programando "tiempo para garabatear" para que tu hijo pueda escribir libremente. |
| Semana 20-<br>mensaje 2 | Los niños que conocen las letras del alfabeto antes de ir al jardín de infantes o al kinder, les irá mejor en la escuela. |
| Semana 21-<br>mensaje 1 | Anima a tu hijo a dibujar y garabatear siempre que sea posible. |



| Semana 21-<br>mensaje 2 | Señala cada palabra mientras lees para que tu hijo pueda asociar la palabra hablada con su respectiva palabra escrita. |
|---|---|
| Semana 22-<br>mensaje 1 | Idea de actividad: Compra tiza para aceras y ayudale a tu hijo a crear obras<br>maestras durante los días cálidos. |
| Semana 22-<br>mensaje 2 | Aprender a garabatear y dibujar va de la mano con aprender a leer. Asegúrate de que sea una prioridad en la vida de tu hijo. |
| Semana 23-<br>mensaje 1 | Fomenta el juego creativo para que los niños hablen, inventen y exploren. |
| Semana 23-<br>mensaje 2 | El juego es una parte muy importante del aprendizaje. "Jugar" les ayuda a los<br>niños recordar lo que han aprendido. |
| Semana 24-<br>mensaje 1 | Idea de actividad: arma un rompecabezas con tu hijo. |
| Semana 24-<br>mensaje 2 | Señala las palabras y los signos que ves y describele cada uno a tu hijo. |
| Semana 25-<br>mensaje 1 | Cuando tengas la oportunidad, hazle preguntas sencillas a tu hijo, cómo "¿con qué letra comienza esta palabra?". |
| Semana 25-<br>mensaje 2 | ¡Prueba esto! Ofrécele cajas de cereal vacías, tazas de plástico y muñecas para que tu hijo juegue "la la casita". |
| Semana 26-<br>mensaje 1 | Juega un juego de mesa para niños más pequeños. Tu hijo/a te puede enseñar las letras, colores, formas y colores. |
| Semana 26-<br>mensaje 2 | ¡Felicidades! |

